#### **OFFICIAL TITLE:**

A Phase 2,Randomized, Double-blind, Placebo-Controlled Efficacy, Pharmacokinetics and Safety Study of CA-008 in Subjects Undergoing Total Knee Arthroplasty

#### **NCT NUMBER:**

NCT03731364

#### **DOCUMENT DATE:**

Version 3.2 19 February 2019

### **Clinical Trial Protocol**

Version 3.2 19 February 2019

Version 3.1: 14 January 2019 Version 3.0: 11 December 2018 Version 2.0: 10 October 2018 Version 1.0: 07 September 2018

A Phase 2, Randomized, Double-blind, Placebo-Controlled Efficacy, Pharmacokinetics and Safety Study of CA-008 in Subjects Undergoing Total Knee Arthroplasty

Investigational Product: CA-008 by Injection/Instillation

**IND:** 129114

Concentric Analgesics, Inc.


This protocol is the property of Concentric Analgesics, Inc. (Concentric) and is intended solely for the guidance of the clinical investigation. This protocol may not—in full or part—be passed on, reproduced, published, or distributed to any person or entity who is not bound by written confidentiality agreement, for any purpose, without the prior consent of Concentric.

Version: 19 February 2019 

## SIGNATURE PAGE

Approved by:

**Clinical Operations Director** Concentric Analgesics, Inc.

Authored and Approved by:

Mike A Royal MD JD MBA

Chief Medical Officer

Concentric Analgesics, Inc.

## 1. KEY PERSONNEL CONTACT INFORMATION

| Sponsor | Concentric Analgesics, Inc. (Concentric) |
|---|---|
| Carole Hodge, PhD<br>Clinical Operations Director | Carole@concentricanalgesics.com<br>858-442-9884 |
| Mike A. Royal, MD<br>Chief Medical Officer<br>Sponsor Medical Monitor | Mike@concentricanalgesics.com<br>858-204-1112 |

| CRO | Lotus Clinical Research, LLC (Lotus) | |
|---|---|---|
| Primary<br>Contact | Caitlyn Avila | Project Manager<br>cavila@lotuscr.com<br>530-902-3070 |
| CRO Medical<br>Monitors | Primary: Jon L. Ruckle, MD, CPI | MedicalMonitorCA-PS-<br>203@Lotuscr.com<br>808-349-9812 |
| | Secondary: Royce Morrison, MD | MedicalMonitorCA-PS-<br>203@Lotuscr.com<br>206-799-7386 |


Table of Changes Protocol V 3.2 (19 FEB 2019) vs. V 3.1 (14 JAN 2018)

| Material changes | V 3.1 | V 3.2 |
|---|---|---|
| Synopsis: Rescue Medication during the Inpatient Period p13; §9.2.2 Inpatient Rescue Medicaiton p57 | From the time of PACU discharge through T12h administer IV hydromorphone 0.5 mg q15 min <i>prn</i> for NRS ≥ 4 as reported by subjects. | From the time of PACU discharge through <b>T48h</b> administer IV hydromorphone 0.5 mg q15 min <i>prn</i> for NRS ≥ 4 as reported by subjects. From T12 through T48h the IV hydromorphone may be used as rescue in addition to PO oxycodone for moderate-to-severe pain. After T48, only PO oxycodone may be used as rescue. If a subject still requires IV opioid rescue after T48, then the subject should undergo an early termination due to lack of efficacy. The rationale for the change was poorly controlled pain noted during the recently enrolled Cohort 2 subjects who complained of poor pain control with oral opioids alone. Dr. Leiman and I discussed his request/concern and agreed to the immediate change to be followed by this minimalistic amendment. |

## Table of Changes Protocol V 3.1 (14 JAN 2019) vs. V 3.0 (11 DEC 2018)

| Material changes | V 3.0 | V 3.1 |
|---|---|---|
| Synopsis: Sample Size p11/Dose | Cohorts #2 and #3 anticipated 16 subjects randomized | Elected to return to 100 mL of study treatment with Cohorts |
| Groups p14/Injection of Study | 3:1 to CA-008 vs. placebo using 75 mL of study | #2 and #3 including 18 subjects each with 2:1 randomization. |
| Treatment p15 | treatment | Study treatment administration instructions remain the same |
| §§6.1 p50, 9.1.2 p 58 and 10.1.3 p65 | | as in cohort #1. |
| Synopsis: Anesthesia p13 | Spinal or general anesthesia allowed | Restrict anesthesia to general anesthesia only |
| §10.1.2.2 p65 | Ropivacaine 0.2% for AC block; 50 mL for site infiltration | Increase concentration of ropivacaine to 0.5% from 0.2% for<br>the ac (adductor canal) block and reduce the volume for site<br>infiltration from 50 to 30 mL |
| Synpsis: Intraoperative Analgesia | No IV hydromorphone during surgery | Modified intraoperative and immediate postoperative |
| p15/Postsurgical Care p16/Rescue | IV fentanyl 100 – 300 mcg intraoperatively per | analgesia regimen to remove potential confusion and improve |
| Medication During the Inpatient | anesthesia discretion | pain control. |
| Period p16<br>§9.2.1 p59 | anesanesia discretion | Within 30 min of anesthesia induction give the subject IV |
| §9.2.2 p60 | Minimal PACU stay | hydromorphone 1.5 mg. |


| | Confusion as to PO or IV choice early postoperatively | During the surgery, ensure that each subject has received at least 100 mcg of IV fentanyl with adjustments above this dose per anesthesiologist discretion. |
|---|---|---|
| | | Within 15 min of the end of surgery, give the subject IV hydromorphone 0.5 mg |
| | | Within 15 min of the end of surgery, administer IV ketorolac and IV acetaminophen. |
| Synopsis: Inclusion Criteria p18<br>§8.2.1 p55 | English only | Added Spanish to inclusion criteria (note this will not apply until the IRB approves the Spanish language ICF and related documents) |
| §17.10 Appendix J p 113 | Guidance for Industry: Toxicity Grading Scale for Healthy<br>Adult and Adolescent Volunteers Enrolled in Preventive<br>Vaccine Clinical Trials | Given that patients receiving TKA are not "healthy adult or adolescent volunteers" the CTCAE v5 is a more appropriate guidance. |

## Table of Changes Protocol V 3.0 (10 DEC 2018) vs. V 2.0 (10 OCT 2018)

| Material changes | V 2.0 | V 3.0 |
|---|---|---|
| Synospsis, Study Duration; | Approximately 61 days per subject from screening to the | Approximately 76 days per subject from screening to the day |
| Synopsis, Visit Schedule; Table 1, | day 29 (D29) visit (however this could be longer to follow | 29 (D29) visit (however this could be longer to follow any AE |
| Schedule of Assessments; §7.2, | any AE to resolution or establishment of a new baseline). | to resolution or establishment of a new baseline). |
| Duration of Participation; §9.5, | | Universal were made changes throughout. |
| Prior and Concomitant Therapy; | | |
| §10.1.1, Screening Phase (Day -45 | | |
| to Day -1); §10.1.2.1, Prior to | | |
| Surgery (D-1 to D0); §10.3.4, | | |
| Medication History | | |
| Synopsis, Overall Study Design; | Anticipated a single pilot (exploratory) cohort prior to | Added two additional exploratory cohorts: Cohort #2 CA-008 |
| Dose Groups; Section 6.1; §8.1.1 | the parallel design stage 2. | 10 mg vs. placebo and Cohort #3 CA-008 15 mg vs. placebo |
| Number of Participants; §9.1.2 | | (with each cohort enrolling n=16 randomized 3:1, |
| Study Treatment Description | | respectively) with a volume of 75 mL for each treatment |
| | | group in Cohort #2 and #3. |
| | | Modified text throughout to reflect this change. |
| Synopsis, Injection of Study | Study treatment infiltration 100 mL with instructions as | Decreased study treatment volume to 75 mL (universal |
| Treatment; §10.1.3 Surgery Phase: | follows: | change throughout) with instructions as follows: |


| Administration of Study Medication into the Surgical Site | With the leg in full extension, perform the following (working from top to bottom or using another standardized method per surgeon discretion): 1. Infiltrate 15 mL circumferentially around the distal femur 2. Infiltrate a total of 30 mL divided equally into the medial and lateral gutters ensuring coverage of the periosteal borders 3. Infiltrate 10 mL around the peripatellar region 4. Infiltrate 10 mL divided equally medial and lateral to the tibial tubercle Following closure of the joint capsule, 5. Instill 20 mL "intra-articularly" (lateral approach) and move the joint through full range of motion | Cohorts #2 and #3: Prior to hardware placement, 75 mL of study treatment should be infiltrated/instilled as follows: 1. Infiltrate 15 mL divided equally throughout the posterior capsule With the leg in full extension, perform the following (working from top to bottom or using another standardized method per surgeon discretion): 2. Infiltrate 15 mL circumferentially around the distal femur 3. Infiltrate a total of 10 mL divided equally into the medial and lateral gutters ensuring coverage of the periosteal borders, and infiltrate 10 mL divided equally medial and lateral to the tibial tubercle 4. Infiltrate 5 mL around the peripatellar region Following closure of the joint capsule, 5. Instill 20 mL "intra-articularly" (lateral approach) and move the joint through full range of motion |
|---|---|---|
| Synopsis, Intraoperative and Postoperative Analgesia; §9.2.1 Inpatient Analgesia | Anticipated a single dose of IV ketorolac and IV acetaminophen administered intraoperatively. | Added additional doses of IV ketorolac and IV acetaminophen:<br>Beginning at T6h (±0.5h) administer IV ketorolac 15 mg and IV<br>acetaminophen 1 g with additional doses of each at T12h<br>(±0.5h) and T18h (±0.5h). |
| Synopsis, Inclusion Criteria; §8.2<br>Eligibility Criteria | BMI ≤ 40 kg/m² allowed | BMI threshold reduced to ≤ 36 kg/m² |
| Synopsis, PK Endpoints; Table 1<br>Schedule of Assessments,<br>footnote 15; §10.1.4 Inpatient<br>Phase: Time 0 (Post-Surgery) to<br>Day 4 (Discharge) | 17 samples for PK | Added 3 additional PK samples at T30, T36 and T48h for a total of 20 samples. This was done due to the higher doses anticipated in cohorts 2 and 3 to ensure adequate assessment of the AUC for CA-101 in plasma. Urine collections will continue for each of the additional cohorts. |


| §5.3 Previous Human Experience | At the time of the prior protocol amendment, the results | Added safety results from the Phase 2 bunionectomy study |
|---|---|---|
| | were not available. | (CA-PS-201). The addition of numerous tables required |
| | | renumbering of all subsequent tables. |
| §10.4.3.1 Primary Efficacy | | With the addition of 2 more exploratory cohorts, it was |
| Endpoint | | decided to pool placebos from each cohort for exploratory |
| | | efficacy analyses. |

# Table of Changes Protocol V 2.0 (10 OCT 2018) vs. V 1.0 (07 SEP 2018)

| Material changes | V 1.0 | V 2.0 |
|---|---|---|
| Synopsis, Study Duration<br>Synopsis, Visit Schedule | 76 days (including a 45-day screening period and 31-day follow up) | 61 days (including a 30-day screening period and 31-day follow up): A shorter screening period was requested by the site. |
| Synopsis, Overall Study Design, Study<br>Objectives, Dose Groups<br>Section 6 Study Objectives, Section<br>9.1.2 Study Treatment Description | Study treatment infiltration 75 mL | Increased study treatment volume to 100 mL (universal change throughout) |
| Synopsis, Study Objectives<br>Section 6.1.2, Secondary Objectives,<br>Section 7.1 Overall Study Design and<br>Plan | | Added a 3 <sup>rd</sup> "Secondary Objective" to the Pilot Stage of the study and the Second Stage of the Study: "to evaluate the opioid-sparing effect of CA-008 vs. placebo" |
| Synopsis, Anesthesia Section 10.1.2.2, Anesthesia and Surgery | No AC or IPACK blocks when spinal anesthesia is administered. | Modified anesthesia regimen such that all subjects will have the AC and IPACK blocks regardless of whether a general or spinal anesthesia is administered. This was done to improve analgesia in the first several hours after surgery for all enrolled subjects. Modified the volumes to be used with ropivacaine blocks or surgical site infiltration with the maximum dose not to exceed 200 mg. Added language re: use of tourniquet prior to surgical incision: "A tourniquet will be used in all subjects. After exsanguination, but prior to surgical incision, perform surgical site infiltration with RopiHCl 0.2% 50 mL (100 mg)." Added language: "The dose of fentanyl administered during surgery should be 100 to 300 mcg per anesthesiologist discretion." This was done to standardize opioid administration during surgery. |
| Synopsis, Injection of Study Treatment<br>Section 10.1.3 Surgery Phase:<br>Administration of Study Medication<br>into the Surgical Site | Prior to wound closure, study treatment will be infiltrated/instilled with a total volume of 75 mL. Study treatment will be injected/instilled into the soft tissues, periosteal and osteotomy sites and capsule around surgical sites as follows: | Prior to hardware placement, study treatment should be infiltrated/instilled as follows: 1. Infiltrate 15 mL divided equally throughout the posterior capsule |


| | <ol> <li>Instill 7.5 mL into each osteotomy location with particular attention to the periosteal borders and intramedullary bone (total 15 mL) using either a catheter or needle</li> <li>Instill 10 mL into the posterior capsule using either a catheter or needle prior to closing</li> <li>Infiltrate 5 mL in and around each collateral ligament (total 10 mL)</li> <li>Infiltrate 40 mL into the surrounding soft tissues</li> </ol> | With the leg in full extension, perform the following (working from top to bottom or using another standardized method per surgeon discretion): 2. Infiltrate 15 mL circumferentially around the distal femur 3. Infiltrate a total of 30 mL divided equally into the medial and lateral gutters ensuring coverage of the periosteal borders 4. Infiltrate 10 mL around the peripatellar region 5. Infiltrate 10 mL divided equally medial and lateral to the tibial tubercle Following closure of the joint capsule, 6. Instill 20 mL "intra-articularly" (lateral approach) and move the joint through full range of motion |
|---|---|---|
| Synopsis, Rescue Medication during<br>the Inpatient Period<br>Section 9.2.2, Inpatient Rescue<br>Medication | IV fentanyl 25-50 mcg q2h through T4 | Removed text referring to time after surgery. Provided a graded approach to rescue to allow for more rescue for severe pain. Reduced frequency of fentanyl dosing to 15 min per site request. Added additional IV opioid choices for use per investigator discretion to supplement oral rescue during the first 24h. Removed references to pain at rest triggering rescue. Moved discussion re: opioid rescue in the 12h prior to discharge to the section "Analgesia during the Outpatient Period" AND increased number of tablets in the oxycodone prescription to "9" in case the patient is discharged prior to a long holiday weekend. |
| Synopsis, Inclusion Criteria #1 | | Removed "reasonably healthy" language |
| Section 8.1, Study Population | | |
| Section 8.2.1, Inclusion Criteria #1 Synopsis, Inclusion Criteria #2 | Adult aged 18-75 years to be enrolled. | Per site request, increased age to 80 years for eligibility |
| Section 8.1, Study Population | Addit aged 10-75 years to be emolied. | Ter site request, increased age to objects for enginity |
| Section 8.2.1, Inclusion Criteria #2 | | |
| Synopsis, Exclusion Criteria #6 | | Removed redundant language and collapsed the indented text into |
| Section 8.2.1, Exclusion Criteria #6 | | the main body |
| Synopsis, Monitored Parameters and | | Added rebound pain assessments |
| Parameter Assessment Times | | |
| Synopsis, Safety Parameter | | Removed surgical site assessment and neurosensory testing at 24h |
| Assessment Times, Table 1 | | per site request: surgeons were quite adamant about not removing |


| Section 10.1.4, Inpatient Phase: Time | | dressings until discharge from the unit due to concerns about |
|---|---|---|
| 0 (Post-Surgery) to Day 4 (Discharge) | | infection with manipulation of the dressing. |
| Synopsis, Efficacy Parameter | | Added time range (±15 min) for NRS assessment at the time of rescue |
| Assessment Times, Table 1 | | request. |
| Section 10.1.4, Inpatient Phase: Time | | Removed NRS assessment 4h after rescue administration. |
| 0 (Post-Surgery) to Day 4 (Discharge) | | Made text clarifications to reduce potential for misunderstanding. |
| Synopsis, Key Secondary Efficacy | | Added as 3 <sup>rd</sup> bullet for consistence with protocol body text: Total |
| Endpoints for Pilot Stage | | opioid consumption (in daily oral morphine equivalents) = OC from |
| | | T0 to T96h: OC <sub>0 to 96h</sub> |
| Synopsis, Other Endpoints for Stage 2 | AUC endpoints at rest and with ambulation were merged | Split AUC endpoints at rest and those with ambulation are split into |
| Section 10.4.4.3, Other Endpoints | into one bullet | separate bullets to reduce confusion. |
| | | In Section 4.4, removed redundant boxed text. |
| Synopsis, PK Endpoints | Modified text re: urine collections | Clarified that urine collections are to be done during Stage 2 only. |
| Synopsis, Stopping Rules | Clarified text relating to stopping rule triggers per FDA | Modified text: |
| Section 7.2, Study Stopping Rules | input | 1 or more subjects with any grade 4 "related" TEAE in any of the |
| | | categories shown in the table below |
| | | 2 or more subjects with the same grade 3 "related" TEAE in any |
| | | of the categories shown in the table below |
| Synopsis, Sample Size Justification | | Removed reference to use of an external unblinded biostatistician. |
| Section 9.4, Blinding | | |
| Table 1, Schedule of Assessments | | Made several corrections to clarify timing for specific assessments. |
| | | Modified footnotes to ensure consistency with text in synopsis and |
| | | protocol proper. |
| | | Added knee x-ray to the list of required safety assessments. |
| Section 9.1.2, Study Treatment | | Clarified text describing formulation for CA-008 |
| Description | | |
| Section 10.1, Study Visits | | Added temperature assessments to all mentions of vital signs |
| Section 10.3.7, Digital Photographs of | | Added clarifying text to make it clear that it is optional |
| the Surgical Site | | |
| Section 10.3.13 Rescue Medications | | Augmented the Equianalgesic Conversion Table to accommodate |
| | | additional opioids requested by the site. |
| Section 10.3.17, 12-Lead | | Fixed broken sentences. |
| Electrocardiogram (ECG) | | |


# 2. PROTOCOL SYNOPSIS

| Sponsor: | Concentric Analgesics, Inc. (Concentric) |
|---|---|
| • | One Ferry Building, Suite 255 |
| | San Francisco, CA 94111 |
| CRO: | Lotus Clinical Research (Lotus) |
| | 100 W. California Blvd., Unit 25 |
| | Pasadena CA 91105 |
| <b>Protocol Number:</b> | CA-PS-203 |
| IND# | 129114 |
| Study Title: | A Phase 2, Randomized, Double-blind, Placebo-Controlled Efficacy, Pharmacokinetics and Safety Study of CA-008 in Subjects Undergoing Total Knee Arthroplasty |
| Study Treatment | CA-008, the investigational product (IP), and matching placebo vehicle are collectively referred to as study treatment |
| Planned Study Center(s): | 1 US site |
| Indication: | Acute postsurgical pain |
| Sample Size: | Pilot stage of the study: |
| | • Cohort #1: total N=18 (randomized 1:1 active or placebo) |
| | • Cohort #2: total N=18 (randomized 2:1 active or placebo) |
| | Cohort #3: total N=18 (randomized 2:1 active or placebo) |
| | A second stage of the study is anticipated with a sample size to be determined after an interim analysis of cohort #3 of the pilot stage is conducted. |
| Population: | Adults ages 18 to 80 years, inclusive, who are planning to undergo an elective unilateral total knee arthroplasty (TKA) and otherwise meet eligibility criteria may be considered for enrollment into the study. |
| Study Duration: | Approximately 76 days per subject from screening to the day 29 (D29) visit (however this could be longer to follow any AE to resolution or establishment of a new baseline). |
| Overall Study<br>Design: | This is a Phase 2, single-center, randomized, double-blind, placebo-controlled, parallel design study evaluating, in a pilot stage of the study involving 3 exploratory cohorts, each with a single dose of CA-008 or placebo. |
| | After an interim unblinded analysis of the pilot stage results and review of pilot stage topline results, a protocol amendment will be performed with a second stage using the doses, sample size and number of CA-008 treatment groups vs. placebo to be determined. |


For each subject, the study will be conducted in two parts:

- Inpatient period which continues to 96h (T96h) after completion of study treatment injection (T0).
- Outpatient period which begins on discharge from the inpatient unit through various follow visits to D29±2 (W4) after surgery. Note that additional follow up visits may occur at any time or even after D29/W4 to follow adverse events (AEs) to resolution or establishment of a new baseline.

#### **Study Objectives:**

#### **Pilot Stage (3 Exploratory Cohorts):**

#### **Primary Objective:**

• To evaluate the efficacy of a single intraoperative administration of either CA-008 vs. placebo in subjects undergoing an elective TKA.

#### **Secondary Objectives:**

- To evaluate the safety and tolerability of a single intraoperative administration of CA-008 vs. placebo in subjects undergoing an elective TKA.
- To evaluate the PK profile of a single intraoperative administration of CA-008 in subjects undergoing an elective TKA.
- To evaluate the opioid-sparing effect of CA-008 vs. placebo.

#### **Second Stage (Parallel Design):**

After an interim unblinded analysis of the 3<sup>rd</sup> cohort of the pilot stage of the study:

#### **Primary Objective:**

• To evaluate the efficacy of a single intraoperative administration of CA-008 (the doses and number of active treatment groups to be determined) vs. placebo in subjects undergoing an elective TKA.

#### **Secondary Objectives:**

- To evaluate the safety and tolerability of a single intraoperative administration of CA-008 vs. placebo in subjects undergoing an elective TKA.
- To determine the efficacy of various doses of CA-008 vs. placebo to be administered intraoperatively in subjects undergoing an elective TKA.
- To evaluate the opioid-sparing effect of various doses of CA-008 vs. placebo.
- To evaluate the PK profile of a single intraoperative administration of various doses of CA-008 in subjects undergoing an elective TKA.

#### **Exploratory Objectives:**

Pharmacoeconomic benefits from administration of CA-008 vs. placebo in subjects undergoing an elective TKA.


# **Study Treatment** Study treatment is to be administered intraoperatively as a single administration via **Dosing Schedule:** "surgical site" infiltration/instillation prior to wound closure. "Surgical site" is defined as the area extending approximately 5 cm in all directions (lateral/medial/proximal/distal/deep) from the incision and osteotomy sites and surrounding tissues. Anesthesia: The surgery will be performed under general anesthesia supplemented by an adductor canal (AC) block AND an IPACK infiltration (Interspace between the Popliteal Artery and the Capsule of the posterior Knee between the femoral condyles). Recent literature suggests the AC+IPACK approach is the new "best practice" to supplement anesthesia as part of an enhanced recovery after surgery (ERAS) for TKA (Cullom 2017, Sankineani 2018). Perform the AC+IPACK local anesthetic regional blocks under ultrasound guidance prior to the start of surgery. Using ropivacaine hydrochloride (RopiHCl) o AC block: 20 mL using 0.5% (100 mg) IPACK infiltration: 20 mL using 0.2% (40 mg) A tourniquet will be used in all subjects. After exsanguination, but prior to surgical incision, perform surgical site infiltration with RopiHCl 0.2% 30 mL (60 mg). The total RopiHCl should not exceed 200 mg. See Appendix M (Section 17.12) for guidance on RopiHCl dosing. **Dose Groups:** Pilot Stage (3 Exploratory Cohorts): Cohort #1: total N=18 randomized 1:1 CA-008 5 mg or placebo (100 mL) Cohort #2: total N=18 randomized 2:1 CA-008 10 mg or placebo (100 mL) • Cohort #3: total N=18 randomized 2:1 CA-008 15 mg or placebo (100 mL) Second Stage (100 mL volume): CA-008 (dose groups to be determined) Placebo **Injection of Study** Prior to hardware placement, 100 mL of study treatment should be infiltrated/instilled **Treatment:** as follows: 1. Infiltrate 15 mL divided equally throughout the posterior capsule With the leg in full extension, perform the following (working from top to bottom or using another standardized method per surgeon discretion): 2. Infiltrate 15 mL circumferentially around the distal femur 3. Infiltrate a total of 30 mL divided equally into the medial and lateral gutters ensuring coverage of the periosteal borders 4. Infiltrate 10 mL around the peripatellar region 5. Infiltrate 10 mL divided equally medial and lateral to the tibial tubercle Following closure of the joint capsule,


| | 6. Instill 20 mL "intra-articularly" (lateral approach) and move the joint through full range of motion |
|---|---|
| | Note that T0 is the time that the study treatment injection/instillation is completed. |
| Intraoperative | Within 30 min of anesthesia induction give the subject IV hydromorphone 1.5 mg. |
| Analgesia: | During the surgery, ensure that each subject has received at least 100 mcg of IV fentanyl with adjustments above this dose per anesthesiologist discretion. |
| | Within 15 min of the end of surgery, give the subject IV hydromorphone 0.5 mg |
| | Within 15 min of the end of surgery, administer the following: |
| | <ul> <li>IV ketorolac 30 mg (for example, ketorolac full prescribing information is available at: http://www.sagentpharma.com/wpcproduct/ketorolac-tromethamine-injection-usp/ [Sagent Pharmaceuticals 2018]). Dose adjustments may be made per surgeon/anesthesiologist discretion to accommodate the subject's age and health status.</li> <li>IV acetaminophen 1g (Ofirmev® full prescribing information at http://ofirmev.com/)</li> </ul> |
| | After these have been administered, no additional non-opioid analgesics are to be administered during the inpatient phase (through T96h). |
| Postsurgical Care: | After surgery, subjects will be monitored in the post-anesthesia care unit (PACU) for at least 90 min during which time efficacy asssessments can begin once the subject is awake. During this time, IV fentanyl 25-50 mcg q5 min <i>prn</i> for moderate-to-severe pain (≥ 4) as reported by subjects using the 0 to 10 numerical rating scale of current pain intensity (NRS). After discharge from the PACU, subjects are followed through T96h as an inpatient. Safety and efficacy evaluations will be performed and blood drawn and urine collected for pharmacokinetic (PK) assessments. Subjects will be required to meet standard criteria for discharge to outpatient status. Subjects will continue to be monitored as an outpatient after discharge through D29/W4 for various safety and efficacy assessments, and later if necessary for safety follow up. |
| Rescue Medication during the Inpatient | From the time of PACU discharge through T48h administer IV hydromorphone 0.5 mg q15 min $prn$ for NRS $\geq$ 4 as reported by subjects. |
| Period: | After T12h, administer PO oxycodone 5 mg q2h $prn$ moderate pain (NRS $\geq$ 4 and $\leq$ 6) or 10 mg q2h $prn$ severe pain (NRS $\geq$ 7). From T12 through T48h, IV hydromorphone may be used as rescue in addition to PO oxycodone for moderate-to-severe pain. After T48, only PO oxycodone may be used as rescue. If a subject still requires IV opioid rescue after T48, then the subject should undergo an early termination due to lack of efficacy. |
| | After T24, administer PO oxycodone 5 mg q4h $prn$ moderate pain (NRS $\geq$ 4 and $\leq$ 6) or 10 mg q4h $prn$ severe pain (NRS $\geq$ 7) |


# Subjects will be encouraged to rescue only for moderate-to-severe pain scores (NRS ≥ 4), however rescue may be requested at any time and medication will be provided when requested. Analgesia during the Once discharged from the inpatient unit, all study participants will be instructed to take a combination of over-the-counter (OTC) analgesics at an appropriate dose per medical **Outpatient Period:** judgment to manage any residual or breakthrough postsurgical pain. If a subject is still requiring opioid rescue in the 12h prior to discharge from the inpatient unit (i.e., from T84h on regardless of whether discharge is delayed), then prescribe no more than 9 tablets of oxycodone 5 mg (1 PO tid prn) per investigator discretion for the initial outpatient period. Document the number of tablets prescribed and also document any additional prescriptions required if the subject's pain continues to be an issue requiring additional opioid medication. If needed for pain management, the following oral OTC analgesics will be recommended for subjects to self-administer (note that these medications will not be provided by the Sponsor): A nonsteroidal anti-inflammatory drug (NSAID) (e.g., ibuprofen 200 mg prn up to qid [Advil® or Motrin®] or naproxen 220 mg prn up to tid [Aleve®]) or other NSAID per investigator discretion and Acetaminophen 1000 mg prn up to tid or 650 mg up to qid (3g daily maximum limit) Persistent pain or pain exacerbations during the outpatient period may suggest the need for an unscheduled in-person visit to assess the surgical site. If such a situation occurs, the Investigator should use clinical discretion on adequacy of analgesic treatment, but to capture this event as an adverse event (AE) and document any required treatments. **Inclusion Criteria:** In order to participate, subjects must meet all inclusion criteria: 1. Plan to undergo an elective primary unilateral total knee arthroplasty (TKA or knee replacement), without collateral procedure or additional surgeries. 2. In the medical judgment of the investigator, be an adult aged 18 - 80 years old, inclusive, and American Society of Anesthesiology (ASA) physical Class 1, 2 or 3 at the time of randomization (Section 17.1 Appendix A). 3. If a male, unless he has a same sex partner, be either sterile (surgically or biologically) or commit to an acceptable method of birth control while participating in the study. The site personnel will provide instructions on what is an acceptable method. 4. If a female, must meet all of the following: a. A female of child-bearing potential (FCBP) must have a negative serum pregnancy test at screening and negative urine pregnancy test before surgery; b. No plan to become pregnant or to breast feed during the study; and


- c. Be surgically sterile or at least one year post-menopausal, have a monogamous partner who is surgically sterile, have a same sex partner or (**one** of the following must apply)
  - i. is practicing double-barrier contraception
  - ii. is practicing abstinence (must agree to use double-barrier contraception in the event of sexual activity)
  - iii. is using an insertable, injectable, transdermal or combination oral contraceptive approved by the FDA for at least 2 months prior to screening and commits to the use of an acceptable form of birth control while participating in the study.
- 5. Have a body mass index  $\leq$  36 kg/m<sup>2</sup>.
- 6. Be willing and able to sign the informed consent form (ICF) approved by an Institutional Review Board (IRB).
- 7. Be willing and able to complete study procedures and pain scales and to communicate meaningfully in English or Spanish with study personnel and return for outpatient follow up visits as required.

#### **Exclusion Criteria:**

# If any of the following exclusion criteria apply, subjects may not participate in the study:

- 1. In the opinion of the Investigator,
  - a. have a concurrent painful condition, other than pain in the knee to be replaced, that may require analgesic treatment during the study period or may confound post-surgical pain assessments.
  - b. have active skin disease or other clinically significant abnormality at the anticipated site of surgery that could interfere with the planned surgery.
- 2. Have a known allergy to chili peppers, capsaicin or the components of CA-008, ropivacaine HCl, ketorolac, acetaminophen, fentanyl, hydromorphone, morphine or oxycodone.
- 3. As determined by the investigator (with input from the study's medical monitor if requested by the investigator), have a history or clinical manifestation of significant medical, neuropsychiatric or other condition, including a clinically significant existing arrhythmia, left bundle branch block or abnormal ECG, myocardial infarction or coronary arterial bypass graft surgery within the prior 12 months, significant abnormal clinical laboratory test value, or known bleeding abnormality that could preclude or impair study participation or interfere with study assessments.
- 4. The following are considered disallowed medications:
  - a. Be tolerant to opioids defined as those who have been receiving or have received chronic opioid therapy greater than 15 mg of oral morphine equivalents (Table 9) per day for greater than 3 out of 7 days per week over a one-month period within 6 months of screening.


- b. Within 1 day prior to surgery and throughout the inpatient period, be taking or using any capsaicin-containing products, such as dietary supplements or over-the-counter (OTC) preparations, including topical formulations, and prescription medications.
- c. Within the 7 days prior to surgery, be taking any central nervous system (CNS) active agent as an analgesic adjunct medication, such as anticonvulsants, antidepressants (such as SNRIs, SSRIs, and tricyclic antidepressants), benzodiazepines, sedative-hypnotics, clonidine and other central alpha-2 agents (e.g., tizanidine), ketamine or muscle relaxants. [Note that SNRIs = Serotonin and norepinephrine reuptake inhibitors and SSRI = Selective serotonin reuptake inhibitors.]
  - i. These drugs are permitted if prescribed for non pain indications and the dose has been stable for at least 30 days prior to surgery. Note that the dose must remain stable throughout the study.
  - ii. If the subject is taking centrally- and/or peripherally-acting analgesic medications, such as acetaminophen, NSAIDs, tramadol or opioids, FOR knee-related pain, the subject may participate in the study if 4(a) above is not applicable and the subject is willing to discontinue these medications 3 days prior to surgery. Note that baby aspirin for cardiovascular prophylaxis is allowed during the study.
  - iii. The use of benzodiazepines and the non-benzodiazepines (eszopiclone, ramelteon, zaleplon and zolpidem) are permitted to treat insomnia during the postoperative period.
- d. Within the 7 days prior to the planned surgery and throughout the study, be taking antiarrhythmics except beta-blockers, digoxin, warfarin (see exception below), lithium, or aminoglycosides or other antibiotics for an infection (except for ophthalmic use or for treatment or prophylaxis of postoperative surgical site infections). At the investigator's discretion, agents intended for deep venous thrombosis (DVT) prophylaxis after the surgery is allowed.
- e. Within the 14 days prior to surgery, be taking parenteral or oral corticosteroids (steroid inhaler for allergy or asthma treatment, topical steroid for a non-clinically significant skin condition not involving the area of surgery or ophthalmic steroids are permissible).
- f. Be on an antianginal, antihypertensive agent or diabetic regimen at a dose that has not been stable for at least 30 days or which is not expected to remain stable while participating in the study.
- 5. In the opinion of the Investigator, within the past year have a history of illicit drug use or prescription medicine or alcohol abuse (regularly drinks > 4 units of alcohol per day; where a unit = 8 oz. beer, 3 oz. wine or 1 oz. spirits).


6. Have positive results on the alcohol breath/saliva test indicative of alcohol abuse or urine drug screen indicative of illicit drug use (unless results can be explained by a current prescription or acceptable over-the-counter medication at screening as determined by the investigator) at screening, and/or prior to surgery. Note that for those subjects who test positive for tetrahydrocannabinol (THC), if they are willing to abstain from use or consumption of THC-containing products from 3 days prior to surgery to the day 8 visit, they may be allowed to participate in the study. 7. Willing and able to avoid foods containing capsaicin for 24 hours prior to surgery. 8. Have previously participated in a clinical study with CA-008. 9. Have participated in another clinical trial or used an investigational product within 30 days or five half-lives (whichever is longer) prior to the planned surgery, or is scheduled to receive an investigational product other than CA-008 while participating in the study. Visit Schedule: Screening D-45 to D-1: Subjects undergo screening during this period. All screening assessments (including informed consent form [ICF]) must be completed at least 1 day prior to surgery. Site Unit Admission D0: Day of surgery, subjects will be randomized and baseline evaluations will be performed prior to surgery. **Surgery D0**: TKA procedure is performed; study treatment is injected prior to wound closure with T0 defined as the time of study treatment completion of administration. PK assessments are to be done per protocol-specified time points through T48h. **Post-surgery T0 to T96h**: Subject remains at the surgical and then site facility for study assessments and PK blood draws. Discharge to outpatient status after T96±4h assessments with follow up instructions, particularly on diary completion. Follow Up D8±1 (W1): clinic visit for study assessments Follow Up D15±2 (W2): clinic visit for study assessments Follow Up D29±2 (W4): clinic visit for study assessments and study completion visit, unless follow up for wound healing is needed If needed, Unscheduled visits or Follow Up after D29±2: Clinic visit as needed for any ongoing safety issue occurring between scheduled visits or continuing after the D29 visit Early Termination (ET): For subjects who terminate early, an ET visit will be required if the subject is agreeable. Safety and subject-reported outcome assessments will be performed. If the subject does not wish to participate in these assessments, he/she should be asked to at least return for a wound check. Monitored Treatment-emergent AEs (TEAEs) **Parameters:** Medical history (MHx)


- Physical examination (PE) findings, particularly neurosensory findings at the site of incision and the skin proximal and distal to the incision
- Surgical site assessment for wound healing
- Neurosensory testing near the surgical site
- Clinical laboratory testing (standard chemistry, CBC, coagulation, urinalysis), drug and alcohol testing, pregnancy testing
- X-ray of the knee
- Electrocardiograms (ECGs)
- Blood draws for pharmacokinetics (PK)
- NRS scores at rest and after physical therapy or transfers to/from bed or wheelchair (inpatient) or ambulation for approximately 10 yards (inpatient or outpatient) using a 0 to 10 numeric rating scale for pain intensity
- Presence of rebound pain at the surgical site
- Knee injury and Osteoarthritis Outcome Score (KOOS)
- Total postsurgical opioid consumption converted to an oral morphine equivalent dose (MED)
- Patient global evaluation (PGE) of satisfaction with study treatment
- Investigator global evaluation (IGE) satisfaction with study treatment (performed by any qualified investigator)
- Postsurgical health economic outcome assessments focusing on the use of health services following discharge (phone calls related to postsurgical pain, unscheduled visits and/or treatments related to postsurgical pain and visits to emergency department)

## Safety Parameter Assessment Times:

- Incidence of spontaneous reported TEAEs or SAEs from T0 through D29/W4 or later if necessary:
  - o TEAEs are defined as AEs occurring post T0
  - AEs recorded from the time the informed consent form (ICF) is signed up to D0/T0 will be recorded in medical history.
- PE: full PE at screening (without a breast, genital or rectal examination). Interim targeted PE on D-1 or D0 prior to surgery (to be conducted on D0 if not done on D-1), T96h, and as an outpatient on D8/W1, D15/W2, and D29/W4 (later if necessary).
- Vital signs (heart rate [HR], blood pressure [BP], respiratory rate [RR]) at screening, D0 prior to surgery, post-surgery T1, T2, T4, T6, T12, and T24h, and every 8 hours thereafter until T96h, and as an outpatient on D8/W1, D15/W2, and D29/W4 or later if necessary. Assess temperature on D-1 or D0 prior to surgery. Daily temps can be recorded along with vital signs per site SOPs at 1, 2, 4, 6, 12, 24, and every 8 hours thereafter until discharge from the


- inpatient facility (if awake at the time of assessment between hours of midnight and 6 a.m.).
- Surgical site assessments at T96h (prior to discharge from the unit) and then as an outpatient on D8/W1, D15/W2, and D29/W4 (later if necessary). If there are skin reactions atypical for the type of surgery, e.g., more than expected erythema, drainage, bruising or hematoma, induration, swelling or other skin changes, they should be documented as AEs, graded for severity and followed regularly until resolution or establishment of a new baseline.
- Neurosensory testing near the incision (compared to a similar site on the opposite leg) will be performed at Screening visit, T96h (prior to discharge from the unit) and then as an outpatient on D8/W1, D15/W2, and D29/W4.
  - Numbness at or near the incision need not be considered a neurologic AE since this could occur because of tissue trauma and inflammation from the surgery.
  - Sensory deficits or clinically significant persistent sensory change beyond the area proximal/distal to the incision at time of discharge, such as allodynia or hyperalgesia, must be designated as a neurologic AE. Subjects will be followed until there is a return to baseline or establishment of a new baseline.
- X-ray of the operated knee at D29 and later if any evidence of abnormalities in bone healing until resolution or stabilization
- Query subjects as to whether they have experienced any rebound or worsening pain at the surgical site at D8, 15 and 29.
- ECGs, standard clinical labs at screening and post-surgery as specified in the Schedule of Assessments and outlined below The Investigator is responsible for determining if out of range laboratory values are clinically significant or not. All clinically significant values will be recorded in the eCRF and followed until resolution.
  - o ECG at screening and T24±2 h
  - Hematology/Coagulation at screening and T96±4h: hemoglobin, hematocrit, white blood cell count with differential, red blood cell count, platelet count, activated partial thromboplastin time (aPTT) and prothrombin time (PT) or international normalization ratio (INR).
  - Blood Chemistry at screening and T96±4h to include at least the following: Alanine aminotransferase (ALT; SGPT) and Aspartate aminotransferase (AST; SGOT), total bilirubin (TBili), gammaglutamyl transferase (GGT), albumin, blood urea nitrogen (BUN), creatinine, alkaline phosphatase (ALK), sodium, potassium, calcium, chloride and glucose.
  - Serum and urine pregnancy test for FCBP: βhCG test at screening and urine test usually to be done within 24 hours prior to surgery.
  - O Urinalysis at screening and T96±4h: including macroscopic analysis


and, if indicated, microscopic analysis.

# **Efficacy Parameter Assessment Times:**

- 1. NRS scores will be assessed as follows:
  - During the inpatient stay, NRS at rest beginning with the PACU admission may be assessed once the subject is awake. If the subject is able to provide responses, obtain NRS scores at 0.5, 1, 2, 4, 6, 8, 12, 16, 20, 24, and every 4 hours (if awake at time of assessment) until discharge from the inpatient unit. Time windows: for T0.5 to T2 (±5 min) and from T4 onward (±15 min).
  - Pain scores may be skipped between the hours of midnight and 6 a.m., but the subject may not miss two consecutive assessments.
  - An additional NRS assessment must be obtained prior to rescue medication request (±15 min). The T12, T24, T48, T72 and T96h assessments must be completed even if the subject is asleep at these times.
  - During the inpatient stay, starting on postoperative day 1 (after T24) perform the following each morning at 0800h (±2h) and each evening at 2000h (±2h) document the NRS at rest and after physical therapy or transfers to/from bed or wheelchair (inpatient) or ambulation for approximately 10 yards (inpatient or outpatient). Actual assessment times must be documented. If however these twice daily assessments coincide with timed assessments of NRS at rest, then the time assessment at rest is used in place of the twice daily assessments, but the assessment with ambulation should still be performed. Resting pain scores are performed on the schedule noted above in the first bullet.
  - During the outpatient period (after T96h through W2), instruct the patient to document, if possible, their NRS scores twice daily at 0800h (±4h) and 2000h (±4h) at rest and on ambulation (e.g. with the use of a walker or a cane) for approximately 10 yards. Note that the actual time of these assessments must be documented in the diary whenever possible. Instruct the patient to:
    - Obtain the morning NRS assessment prior to taking any pain medication or 2 (±15min) hours after taking any pain medication
    - Obtain the evening NRS assessment 2 (±15min) hours after taking any pain medication
- 2. Total opioid consumption (OC) and daily opioid (rescue medication) consumption in MEDs will be recorded during the inpatient period.
  - Document subject days in which no rescue medication or analgesic consumption is required (opioid free, OF) during the inpatient and outpatient period.
  - Document daily use of OTC analgesics (and oxycodone if prescribed) during the outpatient period.
  - Document each opioid prescription provided to the subject and the number of and type of tablets provided to the subject.
  - Document the fraction of subjects who rescue at T6, T12, T24, T48, T72 and T96h


| | 3. Knee Injury and Osteoarthritis Outcome Score (KOOS) at Screening, T96h, D8/W1, D15/W2 and D29/W4 |
|---|---|
| | 4. Patient Global Evaluation (PGE) at T96±4h prior to discharge, D8/W1, D15/W2 and D29/W4 clinic visits. |
| | 5. Investigator Global Evaluation (IGE) at T96±4h prior to discharge, D8/W1, D15/W2 and D29/W4 clinic visits. |
| | 6. Healthcare utilization (HCU) costs defined as an overall summary of costs related to prescription medications, additional visits related to post discharge treatments, particularly for pain crises, and other related outpatient or inpatient treatments |
| Primary Efficacy<br>Endpoint for the<br>Pilot Stage: | For each cohort in the pilot stage, time-specific mean pain intensity scores at T96h for CA-008 vs. placebo. |
| Key Secondary | For each cohort in the pilot stage, CA-008 vs. placebo comparison: |
| Efficacy Endpoints for Pilot Stage: | <ul> <li>Weighted sum of pain intensity (SPI) assessments = Area Under the Curve (AUC) of the NRS current pain intensity scores from T0 to 96h at rest (AUC<sub>0 to 96h</sub>).</li> <li>Percentage of subjects who do not require opioids (i.e., opioid free; OF) from</li> </ul> |
| | T0 to T96: OF <sub>0 to 96h</sub> |
| | • Total opioid consumption (in daily oral morphine equivalents) = OC from T0 to T96h: OC <sub>0 to 96h</sub> |
| Primary Efficacy<br>Endpoint for Second<br>Stage: | For each CA-008 dose vs. placebo comparison: AUC <sub>0 to 96h</sub> |
| Key Secondary | For each CA-008 dose vs. placebo comparison: |
| Efficacy Endpoints for Second Stage: | <ul> <li>Percentage of subjects who do not require opioids (i.e., opioid free; OF) from<br/>T0 to T96: OF<sub>0 to 96h</sub></li> </ul> |
| | <ul> <li>Total opioid consumption (in daily oral morphine equivalents) = OC from T0 to T96h: OC<sub>0 to 96h</sub></li> <li>Using NRS at rest: AUC<sub>0 to W1</sub></li> </ul> |
| Other Endneints for | |
| Other Endpoints for Stage 2: | For each CA-008 dose vs. placebo comparison: • Using NRS at rest: AUC 0 to 24h, AUC 0 to 120h, AUC 6 to 96h, AUC24 to 96h, AUC96h to w1, AUC96h to w2 |
| | AUC 0 to 96h (ambulation), AUC 0 to W1 (ambulation), AUC24h to W1(ambulation), AUC96h to W2 |
| | <ul> <li>(ambulation)</li> <li>Time-specific mean NRS scores at T48, T72, T96, T120, T144 and T168h</li> </ul> |
| | • OC <sub>24 to 48h</sub> , OC <sub>24 to 72h</sub> , OC <sub>24 to 96h</sub> |
| | • OF <sub>24 to 96h</sub> , OF <sub>96h to W1</sub> and OF <sub>96h to W2</sub> |
| | KOOS improvement from T96h to D8/W1, D15/W2 and D29/W4 TTER |
| | • TTFR <sub>after T0</sub> and TTFR <sub>after T24h</sub> |


The fraction of subjects who rescue at T6, T12, T24, T48, T72 and T96h Analgesic consumption from T96h to W1 (AC96h to W1) and AC96h to W2 PGE comparing the %age of subjects reporting "poor" + "fair" vs. "good" + "excellent" responses, and the %age reporting each category of response at T96h, D8/W1, D15/W2 and D29/W4 IGE comparing the %age of those reporting "poor" + "fair" vs. "good" + "excellent" responses, and the %age reporting each category at T96h, D8/W1, D15/W2 and D29/W4 Number and %age subjects with an AE of lack of efficacy (LOE) during the inpatient period: LOE<sub>0 to 96h</sub> HCU<sub>96h to W2</sub> and HCU<sub>96h to W4</sub> **PK Endpoints:** The time points for whole blood collection will be at baseline (from checkin and up to 30 min before the start of surgery), and T5min, T10 min, T15min, T30min, T45min, and T1, T1.5, T2, T2.5, T3, T4, T6, T8, T12, T16, T24, T30, T36 and T48h for a total of 20 samples) with T0 = end of study treatment administration. Actual sampling times will be used to calculate plasma-derived PK parameters. The PK will be documented in the PK Analysis Plan document. Additionally, immediately post surgery begin a 24h urine collection to assess urinary CA-101 excretion to be collected in two aliquots: after surgery to T6h and T6h to T24h. **Stopping Rules:** Study enrollment will be paused if subjects experience intolerable "possibly related" TEAEs, as defined below: 1 or more subjects with any grade 4 "related" TEAE in any of the categories shown in the table below 2 or more subjects with the same grade 3 "related" TEAE in any of the categories shown in the table below

Refer to the in-text table below for descriptions of AE grading.


| | | | | | Potentially Life |
|---|---|---|---|---|---|
| | | Mild | Moderate | Severe | Threatening |
| | Category | (Grade 1) | (Grade 2) | (Grade 3) | (Grade 4) |
| | Abnormal Wound Healing: Infection Dehiscence Necrosis | Mild symptoms;<br>clinical or diagnostic<br>observations only;<br>intervention not<br>indicated. No<br>interference with age-<br>appropriate<br>instrumental ADL | Minimal, local or<br>noninvasive<br>intervention<br>indicated; May<br>require local wound<br>care or medical<br>intervention (e.g.,<br>dressings or topical<br>medications) | Severe or medically significant but not immediately lifethreatening; hospitalization or prolongation of existing hospitalization indicated; limiting ADLs. May require IV antibiotics, antifungals, or antivirals or radiologic intervention. | Life-threatening consequences; urgent intervention indicated |
| | ECG/Cardiac<br>issues<br>Vital Signs<br>Labs | Asymptomatic,<br>intervention not<br>indicated | Non-urgent medical intervention indicated | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of existing hospitalization indicated | Life-threatening consequences; urgent intervention indicated |
| | Focused Neurosensory Testing (performed by trained Investigator) | Mild symptoms | Moderate symptoms;<br>limiting instrumental<br>ADL | Severe symptoms requiring medical intervention; limiting self-care ADL | Life-threatening and urgent intervention indicated |
| | Should a stopping rule be triggered, an external independent safety review committee (SRC) will review the data to determine whether or not it is appropriate to continue with enrollment. The SRC Charter details the membership, roles and responsibilities of the SRC. | | | | |
| Sample Size Justification: | Given the uncertainty in estimating a sample size for TKA surgery, the Pilot Stage will be conducted using multiple cohorts to augment the guidance from the results from the Phase 2 bunionectomy study to determine the sample size for Stage 2 parallel design portion of this study. | | | | |
| Study Populations: | <ul> <li>The following three analysis populations are planned for this study:</li> <li>The Safety Population will include all subjects who received any part of a dose of study treatment.</li> <li>The PK Population will include all subjects who receive a full dose of study treatment and have PK assessments through 6h.</li> <li>The intent-to-treat (ITT) population will include all subjects as randomized to study treatment. The modified intent-to-treat (mITT) Population will include all subjects who receive a full dose of study treatment and complete the first 3 pain assessments (through T2h).</li> <li>Study completers (Study Completers) will include all subjects who receive a full dose of study treatment and complete the entire study period through D29±2/W4.</li> </ul> | | | | |
| | randomization | n but prior to rec | eiving study trea | pation (early termina<br>tment will be replace<br>treatment will not be | d. |
| | - | | | e study, will be asked | • |


assessments through T96h if they have not elected to withdraw from all aspects of study participation. Subjects who elect to discontinue participation prior to D8 (W1) will be considered to have terminated as of the date of their election, however they will be asked to return to the site one time, if willing and at their convenience, to ensure that adequate wound healing has occurred. Statistical All safety assessments and baseline characteristics will be summarized using the Safety **Considerations:** Population. Efficacy analyses will be performed using the mITT population. PK analyses will be performed using the PK population. All summaries will be grouped by the actual treatment received. Subjects receiving vehicle placebo will be combined for summaries. Safety and tolerability will be evaluated by examining the occurrence of AEs, including Treatment-Emergent AEs. AEs leading to discontinuation from the study, AEs related to study treatment and AE severity will be summarized by treatment group. Actual and change from baseline in clinical laboratory measures, vital signs, and ECGs will also be assessed and summarized by treatment group. These data will be summarized using descriptive statistics including n, mean, SD, SEM (if appropriate), median, minimum and maximum. Abnormal values will be determined and flagged in the listings. Laboratory shift tables displaying the change (number of subjects) relative to the normal range from baseline to each study visit will also be presented by treatment for each test. The Investigator should exercise medical and scientific judgment in deciding whether an abnormal laboratory finding or other abnormal assessment is clinically significant. While the study is not specifically designed to detect a significant difference in efficacy between CA-008 and placebo, efficacy analyses will be performed as secondary endpoints.


**Table 1. Schedule of Assessments** 

| Assessment | Screening | | | In Pa | tient | | | | ] | Follow-U | p | Unscheduled | Early |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Prior to<br>Surgery | Surgery | Post-<br>Surgery | 24h | 48h | 72h | 96h | | | | Visit <sup>1</sup> | Termination <sup>19</sup> |
| Study Day | -45 to -1 | 0 | 0 | 0 | 1 | 2 | 3 | 4 | 8±1<br>days | 15±2<br>days | 29±2<br>days | | |
| Informed Consent | X | X | | | | | | | | | | | |
| Screening Medical and<br>Surgical History | X | X | | | | | | | | | | | |
| Inclusion/Exclusion Criteria | X | X | | | | | | | | | | | |
| Screens for alcohol/drugs of abuse | X | X | | | | | | | | | | | |
| Enroll/Randomize | | X | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | |
| Subject Pain Assessment<br>Training | X <sup>2</sup> | $X^2$ | | | | | | | | | | | |
| Surgery | | | X | | | | | | | | | | |
| Study treatment Infiltration/instillation | | | X | | | | | | | | | | |
| Pregnancy Test | X <sup>3</sup> (serum) | X <sup>3</sup> (urine) | | | | | | | | | | | |
| Vital Signs | X | X | | $X^4$ | $X^4$ | $X^4$ | $X^4$ | $X^4$ | X | X | X | X | X |
| Temperature | X | X | | $X^4$ | $X^4$ | X <sup>4</sup> | $X^4$ | $X^4$ | X | X | X | X | X |
| Physical Examination | X <sup>5</sup> | X <sup>5</sup> | | | | | | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> | X <sup>5</sup> |
| 12-Lead ECG | X | | | | $X^6$ | | | | | | | | |
| Surgical Site assessment | | | | | | | | $X^7$ | $X^7$ | $X^7$ | $X^7$ | $X^7$ | $X^7$ |
| Neurosensory Exam | X | | | | | | | X8 | X8 | X8 | X <sup>8</sup> | X <sup>8</sup> | X8 |
| Blood draw for laboratory tests | X <sup>9</sup> | | | | | | | X <sup>9</sup> | | | | | |
| Urine sample for urinalysis | $X^9$ | | | | | | | $X^9$ | | | | | |
| Rescue Medication consumption | | | | X | X | X | X | X | X | X | | X | X |
| Concomitant Medication Assessment | X | X | | X | X | X | X | X | X | X | X | X | X |
| Adverse Event Assessment | X | X | X | X | X | X | X | X | X | X | X | X | X |
| NRS pain assessments | | | | $X^{10}$ | $X^{10}$ | $X^{10}$ | $X^{10}$ | $X^{10}$ | $X^{10}$ | $X^{10}$ | | $X^{10}$ | $X^{10}$ |
| Subject home diary record (NRS) | | | | | | | | X <sup>11</sup> | X <sup>11</sup> | X <sup>11</sup> | | X <sup>11</sup> | X <sup>11</sup> |


| Assessment | Screening | | | In Pa | tient | | | | Follow-Up | | | Unscheduled | Early |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Prior to<br>Surgery | Surgery | Post-<br>Surgery | 24h | 48h | 72h | 96h | | | | Visit <sup>1</sup> | Termination <sup>19</sup> |
| Study Day | -45 to -1 | 0 | 0 | 0 | 1 | 2 | 3 | 4 | 8±1<br>days | 15±2<br>days | 29±2<br>days | | |
| Paper Diary (review, distribution and/or collection) | | | | | | | | X <sup>12</sup> | X <sup>12,13</sup> | X <sup>12,13</sup> | | X <sup>12,13</sup> | X <sup>13</sup> |
| Subject home diary (analgesic consumption) | | | | | | | | X | X | X | | X | X |
| Prescription for outpatient opioid rescue if needed | | | | | | | | X <sup>14</sup> | | | | | |
| KOOS Survey | X | | | | | | | X | X | X | X | X | X |
| PGE assessment | | | | | | | | X | X | X | X | X | X |
| IGE assessment | | | | | | | | X | X | X | X | X | X |
| Blood draw for PK analysis | | $X^{16}$ | | X <sup>15, 16</sup> | X <sup>15, 16</sup> | X <sup>15</sup> , | | | | | | | |
| 24h Urine Collection | | | | X <sup>16, 17</sup> | X <sup>16, 17</sup> | | | | | | | | |
| Rebound pain | | | | | | | | | $X^{18}$ | $X^{18}$ | $X^{18}$ | $X^{18}$ | $X^{18}$ |
| Knee x-ray | | | | | 121 22 | | | 4 | | | $X^{20}$ | $X^{20}$ | $X^{20}$ |

Unscheduled visit may occur at any time, however if after Day 29 it should occur if insufficient wound healing is assessed by the Investigator at the Day 29 visit or to follow up any ongoing AE to resolution or establishment of a new baseline. For unscheduled visits prior to Day 15, collect efficacy assessments, including NRS scores and diary logs.

- <sup>2</sup> Pain assessment training with test during screening; rewatch video only prior to surgery.
- Note pregnancy tests are for FCBP; urine pregnancy test is to be performed within 24 hours of scheduled surgery.
- Vital signs and temperature assessed together at 1, 2, 4, 6, 12, 24 and every 8 hours thereafter (if awake at time of assessment between the hours of 00:00 and 06:00) until discharge from the inpatient unit (may not miss two consecutive assessments). There will be a ±5-minute window allowed for the collection of vital signs in the first 4 hours after the end of surgery, after which for vital signs and temperatures there will be a ±15-minute window allowed.
- A complete medical history and physical examination including all major body systems will be performed at Screening. In addition, at the following times, an interim medical history and targeted physical examination will be performed prior to surgery (if not done on D-1), and to capture changes after Surgery, at 96 hours (± 4 hours) after the administration of study medication, but prior to discharge, and Day 8, Day 15 and Day 29 after the administration of study medication or if the subject terminates early, at that time if allowed. Body weight (kg), in indoor clothing, but without shoes, will be measured at Screening and at 96 hours. Height (in cm) will be measured and BMI will be calculated at Screening only.
- <sup>6</sup> Post-Surgery ECG should be performed at 24 hours (±2 hours) after study medication administration.
- Surgical Site assessment: 96 hours (±4 hours after study medication administration but prior to discharge from the inpatient unit) and Day 8, 15 and 29.
- Neurosensory Exam of the area proximal to the surgical incision approximately 3 cm from the incision at Screening visit, 96 hours (±4 hours, but prior to discharge) and Day 8, Day 15 and Day 29 after the administration of study medication or if the subject terminates early, at that time if allowed.
- 9 Clinical Laboratory tests (chemistry, hematology, coagulation and urinalysis) should be performed at screening and prior to discharge from the inpatient unit (Lab collection window for 96h is ±4h hours).
- NRS pain assessments during the inpatient stay, NRS at rest assessments start in the PACU once the subject is awake at 0.5, 1, 2, 4, 6, 8, 12, 16, 20, 24, and every 4 hours (if awake at time of assessment) until discharge from the inpatient unit. Pain scores may be skipped between the hours of midnight and 6 a.m., but the subject may not miss two consecutive assessments. Also assess NRS at the time of rescue request (±15 min). The T12, T24, T48, T72 and T96h assessments must be completed even if the subject is asleep at these times. There will be a ±5-minute window


allowed for the collection of each assessment in the first 2 hours after PACU admission, after which will be a  $\pm 15$ -minute window allowed. During the inpatient period document the NRS at rest and on ambulation (e.g., transitioning from a recumbent position to a sitting or standing position or during transfers to or from a bed to a wheelchair and then to the bathroom) twice daily at 0800h ( $\pm 2h$ ) and 2000h ( $\pm 2h$ ) with the actual time of these assessments documented. These twice daily scores are performed independently of pain scores at rest during the inpatient period. If however these twice daily assessments coincide with timed assessments of NRS at rest, then the time assessment at rest is used in place of the twice daily assessments. During the outpatient period, instruct the subject to document, if possible, their NRS scores twice daily at 0800h ( $\pm 4h$ ) and 2000h ( $\pm 4h$ ) at rest and on ambulation (e.g. with the use of a walker or a cane) for approximately 10 yards after T96 through D15 (not through D29). Note that the actual time of these assessments must be documented in the diary. Instruct the subject to:

- Obtain the morning NRS assessment prior to taking any pain medication or 2 (±15-min) hours after taking any pain medication.
- Obtain the evening NRS assessment 2 (±15-min) hours after taking any pain medication.

If an early termination is elected before Day 15, collect efficacy assessments, including NRS scores and diary logs.

- 11 The subject is expected to document NRS pain scores at rest and on ambulation 2x/day through Day 15 (at the times and qualifications noted above).
- The diary and instructions are provided to the subject prior to discharge (T96h). At each subsequent visit, review Subject Diary instructions with subject and collect their NRS scores and other study-related assessments.
- 13 Collect Subject Diary Data
- 14 If the subject is continuing to require opioids during the 12 hours prior to discharge (any time from T84h onward), then write a prescription for no more than 9 tablets of oxycodone 5 mg tablets for use tid prn per investigator discretion.
- Collect blood samples for PK. The time points for whole blood collection will be at baseline (from Check-in and up to 30 min prior to surgery), and T5min, T10 min, T15min, T30min, T45min, and T1, T1.5, T2, T2.5, T3, T4, T6, T8, T12, T16, T24, T30, T36 and T48h for a total of 20 samples) where T0 = end of study treatment administration. There will be a ±2-minute window allowed for the 5 to 15-minute collections, a ±5-minute window allowed for collections T30 min through T4h, and a ±15-minute window for collections after T4 hours.
- Subjects must abstain from foods containing capsaicin for 24 hours prior to all PK blood draws.
- <sup>17</sup> Collect the subject's urine for 24 hours after surgery in two aliquots: post surgery to T6h and T6h to T24h.
- Assess for presence of rebound pain at the surgical site (yes/no response).
- 19 If the subject terminates early and is willing to come in to complete all safety and efficacy assessments then complete all procedures listed. If unwilling to come in for all such assessments, at least attempt to bring the subject in for a surgical site assessment.
- 20 X-ray of the operated knee on D29 and later if any evidence of abnormal bone healing until resolution or stabilization. Also perform this at early termination if subject gives consent.


## 3. TABLE OF CONTENTS

| 1. K | ey Personnel Contact Information | 3 |
|---|---|---|
| Table o | of changes Protocol V 3.1 (14 JAN 2019) vs. V 3.0 (11 DEC 2018) | 4 |
| Table o | of changes Protocol V 3.0 (10 DEC 2018) vs. V 2.0 (10 OCT 2018) | 5 |
| Table o | of changes Protocol V 2.0 (10 OCT 2018) vs. V 1.0 (07 SEP 2018) | 7 |
| | rotocol Synopsis | |
| | able of Contents | |
| | st of Abbreviations and Definition of Terms | |
| | troduction | |
| 5.1. | Background | |
| 5.1.<br>5.2. | CA-008 Product Introduction. | |
| 5.2.<br>5.3. | Previous Human experience | |
| 5.4. | Study Rationale | |
| 5.4.<br>5.5. | Dose Rationale | |
| | tudy Objectives | |
| | i u | |
| 6.1. | Pilot (Exploratory) Stage of the Study | |
| 6.2. | Second (Parallel Design) Stage of the Study | |
| 7. In | vestigational Plan | |
| 7.1. | Overall Study Design and Plan | |
| 7.2. | Duration of Participation | 49 |
| 7.3. | Study Stopping Rules | 49 |
| 8. Se | election of Study Population | 51 |
| 8.1. | Study Population | 51 |
| 8.2. | Eligibility Criteria | 51 |
| 9. St | tudy Treatments | 55 |
| 9.1. | Study Treatment | 55 |
| 9.2. | Other Interventions | |
| 9.3. | Method of Assigning Subjects to Treatment Groups | 58 |
| 9.4. | Blinding | |
| 9.5. | Prior and Concomitant Therapy | |
| 9.6. | Study Restrictions | |
| 9.7. | Treatment Compliance | 59 |
| 10. | Conduct of the study | 60 |
| 10.1. | · | |
| 10.2. | · | |
| 10.3. | V 1 | |
| 10.4. | • | |
| 11 | ADVEDCE EVENTS | 77 |

| 11.1. | Adverse Events and Serious Adverse Events | 77 |
|---|---|---|
| 12. I | Oata Quality Assurance | 82 |
| 12.1. | Data Collection | |
| 12.2. | Study Auditing and Monitoring | 82 |
| 13. S | Statistical Methods and Determination of Sample Size | <b>Q</b> /1 |
| 13.1. | Statistical and Analytical Plans | |
| 13.1. | Sample Size Justification | |
| 13.3. | Analysis Populations | |
| 13.4. | Planned Analyses | |
| 13.5. | Study Subjects and Demographics | |
| 14 6 | • • | |
| | Site and Investigator Responsibilities | |
| 14.1.<br>14.2. | Regulatory and Ethical Considerations Privacy and Confidentiality | |
| 14.2.<br>14.3. | Study and Site Closure | |
| 14.3.<br>14.4. | Regulatory Documents and Records Retention | |
| 14.4.<br>14.5. | Delegation of Responsibilities and Adequate Resources | |
| 14.6. | Protocol Amendments | |
| 14.7. | Financial Disclosure | |
| | nvestigator Protocol Agreement Page | |
| 16. F | References | 96 |
| 17. A | Appendices | 97 |
| 17.1. | Appendix A: American Society of Anesthesiologists Physical Status Classification S | System |
| (ASA | Class) | |
| 17.2. | Appendix B: 0 to 10 Numerical Rating Scale of Pain Intensity (NRS) | |
| 17.3. | Appendix C: Assessment of Rebound Pain at the Surgical Site (Rebound Pain) | |
| 17.4. | Appendix D: Patient Global Evaluation [of Satisfaction with Study Treatment] (PC | |
| 17.5. | Appendix E: Investigator Global Evaluation of Study Treatment] (IGE) | |
| 17.6. | Appendix F: Surgical Site Assessment | |
| 17.7. | Appendix G: Surgical Wound Adverse Event Grading Guide | |
| 17.8. | Appendix H: Neurosensory Examination Form | |
| 17.9. | Appendix I: Toxicity Grading Scale for Clinical Laboratory Abnormalities | |
| 17.10. | ii v | |
| 17.11. | | |
| 17.12. | 11 9 | |
| 17.13. | Appendix M: Knee Injury and Osteoarthritis Outcome Survey (KOOS) | 113 |
| LIST ( | OF TABLES | |
| Table 1. | | |
| Table 2. | , | |
| Table 3. | Summary of TEAEs by MedDRA SOC/PT (CA-PS-201) | 37 |

| Table 4. | Summary of Related TEAEs by MedDRA SOC/PT | 42 |
|-----------|---------------------------------------------|----|
| Table 5. | Summary of Related TEAEs by Frequency | 44 |
| Table 6. | Summary of Related Local TEAEs by Frequency | 45 |
| Table 7. | Summary of Severe TEAEs by Frequency | |
| Table 8. | Study Stopping Rules | |
| Table 9. | Equianalgesic Conversion Table | |
| Table 10. | Clinical Laboratory Assessments | 72 |


## 4. LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

| Abbreviation | Term |
|---|---|
| AE | Adverse event |
| ALT | Alanine aminotransferase |
| ANCOVA | Analysis of Covariance |
| aPTT | Activated partial thromboplastin time |
| ASA | American Society of Anesthesiologists |
| AST | Aspartate aminotransferase |
| AUC | Area Under the Curve |
| BID | Bis in die (twice daily) |
| BLQ | Below limit of quantitation |
| BP | Blood Pressure |
| CA-008 | Investigational product |
| CA-101 | Cyclic urea |
| CFR | Code of Federal Regulations |
| CK | Creatine kinase |
| CL | Clearance |
| C <sub>max</sub> | Maximum plasma concentration |
| CNS | Central nervous system |
| CRF | Case Report Form (may include electronic data capture systems or paper forms) |
| CRO | Contract research organization |
| CS | Clinically significant |
| CSA | Clinical Study Agreement |
| D# or D-# | Day # (study days after surgery), Day # prior to surgery |
| DBP | Diastolic Blood Pressure |
| DVT | Deep Venous Thrombosis |
| ECG | Electrocardiogram |
| EDC | Electronic data capture |
| ET | Early Termination |
| FCBP | Female of child bearing potential |
| FDA | Food and Drug Administration |
| FIH | First-In-Human |
| FCBP | Female of child-bearing potential |
| G | Gram |
| GCP | Good Clinical Practice |
| GGT | Gamma-glutamyl transferase |
| GLP | Good Laboratory Practice |


| Abbreviation | Term |
|--------------|------------------------------------------------|
| H or HRS | Hours |
| HC1 | Hydrochloride |
| HCU | Health care utilization |
| HED | Human Equivalent Dose |
| HEENT | Head, Eye, Ear, Nose and Throat |
| ICF | Informed consent form |
| ICH | International Conference on Harmonisation |
| IEC | Institutional Ethics Committee |
| IGE | Investigator Global Evaluation |
| INR | International Normalized Ratio |
| IRB | Institutional Review Board |
| ITT | Intent-to-treat |
| LLOQ | Lower limit of quantitation |
| LOE | Lack of efficacy |
| mcg or µ | Microgram |
| MED | Morphine equivalent dose |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Mg | Milligram |
| min | Minutes |
| mL | Milliliter |
| NCS | Not clinically significant |
| NOAEL | No Observed Adverse Effect Level |
| NRS | Numeric Rating Scale of Pain Intensity |
| NSAID | Nonsteroidal anti-inflammatory drug |
| OC | Opioid consumption in morphine equivalent dose |
| OF | Opioid-free days |
| OTC | Over-the-counter |
| PACU | Post-anesthesia care unit |
| PE | Physical examination |
| PGE | Patient Global Evaluation |
| PHN | Postherpetic neuralgia |
| PI | Principal Investigator |
| PK | Pharmacokinetic[s] |
| PO | Per oram (oral) |
| PRN | Pro re nata (as needed) |
| PT | Prothrombin time |


| Abbreviation | Term |
|---|---|
| QID | Quater in die (four times daily) |
| RBC | Red blood cell |
| RopiHCl | Ropivacaine hydrochloride |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SBP | Systolic blood pressure |
| SC | Subcutaneous |
| SD | Standard deviation |
| SE | Standard error |
| SOC | System Organ Class |
| SNRIs | Serotonin-norepinephrine reuptake inhibitors |
| SRC | Safety Review Committee |
| SSRIs | Selective serotonin reuptake inhibitors |
| T# | Time in hours after completion of study medication dosing (T0) |
| t <sub>1/2</sub> | Elimination half-life |
| TEAEs | Treatment emergent adverse event[s] |
| TID | Ter in die (three times daily) |
| TKA | Total knee arthroplasty |
| $T_{\text{max}}$ | Time to maximum plasma concentration |
| TRPV1 | Transient receptor potential vanilloid-1 |
| UDS | Urine drug screen[ing] |
| US | United States |
| V | Volume of distribution |
| W# | Week # visit after surgery |
| WHO | World Health Organization |


#### 5. INTRODUCTION

## 5.1. Background

Concentric Analgesics, Inc. (Concentric) is developing CA-008 to provide long-lasting pain relief of post-surgical pain following a single local administration (for 96h and beyond). CA-008 is a prodrug of trans-capsaicin (trans-8-methyl-N-vanillyl-6-nonenamide), the substance in chili peppers that produces the sensation of spiciness. Capsaicin is a transient receptor potential cation channel, subfamily V (vanilloid), member 1 (TRPV1) agonist. TRPV1 is a ligand-gated, nonselective, cation channel preferentially expressed most densely in C-fiber nociceptors and to a lesser extent on  $A\delta$ -fiber nociceptors (Babbar 2009, Caterina 2001). TRPV1 responds to noxious stimuli including capsaicin, heat, and extracellular acidification, and integrates simultaneous exposures to these stimuli (Suresh 2010, Surh 1995, Tominaga 1998).

Capsaicin exposure to TRPV-1-expressing nociceptor peripheral terminals results in initial excitation of the nociceptor followed by a functional desensitization which continues for some time after removal of capsaicin from the site. Capsaicin, however, is virtually insoluble in aqueous media or local anesthetic solutions which means that capsaicin formulations tend to be quite hydrophobic and viscous making them hard to inject and less likely to permeate surgical site tissues. Anesiva, which had been developing capsaicin for the management of post-surgical pain and osteoarthritis, solubilized capsaicin in polyethylene glycol 300 (Hartrick 2011). The product was instilled into the open surgical site and after waiting for 5 minutes, was removed via surgical suction. This route of administration while simple and perhaps convenient, limited exposure of capsaicin only to the exposed surfaces of cut tissue and bone with little to no ability to penetrate into the affected soft tissues.

To work around the solubility limitations of capsaicin, the highly water soluble capsaicin prodrug CA-008 was developed for local infiltration. It avoids the physicochemical limitations of capsaicin while providing greater target engagement which theoretically would produce superior local analgesia, particularly after surgical trauma. Based upon this mechanism of action, local delivery of a TRPV1 agonist throughout the tissues around the surgical site prior to wound closure to maximize target engagement should result in a meaningful reduction of post-surgical pain over several days to weeks. This improved long-term pain relief has the ability to augment current multimodal analgesia or enhanced recovery programs which may help to avoid the need for supplemental opioid use after surgery.

While no capsaicin products have been approved for injection or instillation into a wound site in the US, several companies have or had clinical development programs for such products. Centrexion Therapeutics has an active development program (CTNX-4975) for intraarticular injection of capsaicin for chronic osteoarthritis and Morton's neuroma (see <a href="http://centrexion.com/our-pipeline/">http://centrexion.com/our-pipeline/</a>). Note that Centrexion is using the Anesiva highly viscous polyethylene glycol formulation for its intraarticular knee joint injections.


### 5.2. CA-008 Product Introduction

The active moiety of CA-008, capsaicin, has certain attractive properties for treatment of post-operative pain from a pharmaceutical perspective. CA-008 is water soluble and easy to inject through a 25 g needle or larger. It readily penetrates surgical site tissues where it releases capsaicin through a non-enzymatic pH-driven process. Local administration of CA-008 at or near the source of pain either topically, by infiltration or by instillation into a surgical site results in low systemic levels of capsaicin.

CA-008 was created to improve delivery of capsaicin without having to account for its poor solubility profile in tissues. CA-008 provides an aqueous formulation that could be simply infiltrated in the wound site to achieve local capsaicin release to produce a maximal effect. The free base form of CA-008 rapidly breaks down at physiological pH to yield capsaicin and a cyclic urea, as shown in the scheme below:

CA-008 was specifically selected for development due to its short half-life (<5 min) at neutral pH. In Tris buffer at pH 7.4 and 37°C, it completely breaks apart to capsaicin and CA-101 as the sole degradants.

The cyclic urea (CA-101) formed has not been previously evaluated for biological activity. While not a known compound in the clinical literature, its safety was evaluated in all nonclinical studies with CA-008 and it was shown to be inactive. The toxicokinetic profiles for CA-008, CA-101, and capsaicin were determined in GLP safety studies and the PK profile for various doses were determined in a Phase 1 ascending dose safety study in patients undergoing bunionectomy.

# 5.3. Previous Human experience

There is substantial clinical support for the potential safety of capsaicin, the active molecule released by CA-008 in vivo. In addition to consumption in hot spicy foods (chili peppers), capsaicin is an approved product for dermal applications for OTC and prescription use (Qutenza; 8% patch for management of neuropathic pain associated with post herpetic neuralgia), is frequently used intradermally in experimental pain models, and has been studied clinically for wound instillation for postsurgical analgesia (Anesiva; Adlea; capsaicin for instillation).

A first-in-human study (Study CA-PS-2017-101) evaluated the safety and tolerability of CA-008 in subjects undergoing a unilateral transpositional first metatarsal osteotomy for correction of hallux valgus deformity, more commonly known as a bunionectomy. This study also evaluated

pharmacokinetic (PK) and preliminary efficacy assessment of CA-008 to inform future studies in our clinical development plan. This study was originally designed to look at 4 different doses of CA-008 (0.5 mg, 1 mg, 2 mg, and 3 mg), however based upon the relatively benign adverse event (AE) profile, the Data Management Committee gave the go-ahead for a 5<sup>th</sup> cohort (4.2 mg) to be added. The safety, efficacy and PK results for the Phase 1 bunionectomy study are shown in the current Investigators' Brochure.

Additionally, a follow-on Phase 2 bunionectomy study (CA-PS-201) was completed with 147 subjects enrolled and randomized to one of 3 active doses: 0.05 mg/mL (0.7 mg), 0.15 mg/mL (2.1 mg) and 0.3 mg/mL (4.2 mg) vs. placebo in a 1:1:1:1 randomization, respectively. The results are still being compiled at the time of this protocol amendment. Based upon topline results, the highest dose of 4.2 mg was statistically significantly superior to placebo for the primary efficacy endpoint of AUC 0-96h (p=0.005) and key secondary efficacy endpoints: AUC 0 to week 1 (p=0.036); mean opioid consumption (reduced by 50%, p<0.002); and percent of subjects who were opioid free from 0 to 96h (26% vs. 5% for placebo; p=0.039). The following Tables 2-7 show the summary of safety for the study based upon summary tables and subject listings. Note that in Table 3, the Summary of TEAEs by MedDRA SOC/PT, there were a number of preferred terms that were somewhat vague, so these are accompanied by footnotes detailing the verbatim terms to provide background context.

Table 2. Summary of Adverse Events (CA-PS-201)

| | | | CA-008 | | |
|---|---|---|---|---|---|
| No. of Subjects<br>TEAEs. | Total<br>(N=147) | 0.7 mg (0.05 mg/mL)<br>N=36<br>n (%) | 2.1 mg (0.15 mg/mL)<br>N=36<br>n (%) | 4.2 mg (0.3 mg/mL)<br>N=37<br>n (%) | (Standard of care alone)<br>N=38<br>n (%) |
| No. of TEAEs | 287 | 69 | 82 | 76 | 60 |
| No. of Subjects with any TEAE <sup>1</sup> | 106<br>(72.1%) | 27 (75.0%) | 28 (77.8%) | 26 (68.4%) | 25 (67.6%) |
| No. of "Related" AEs | 43 | 8 | 11 | 14 | 10 |
| No. of Subjects with any "Related" TEAE | 28<br>(19.1%) | 8<br>7 (19.4%) | 11<br>7 (19.4%) | 14<br>7 (18.4%) | 10<br>7 (18.9%) |
| No. of "Severe" AEs | 7 | 3 | 2 | 2 | 0 |
| No. of Subjects with any "Severe"<br>TEAE | 6 (4.1%) | 2 (5.6%) | 2 (5.6%) | 2 (5.3%) | 0 |
| No. of SAEs | 1 | 0 | 0 | 0 | 1 |
| No. of Subjects with any SAE | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| No. of TEAEs leading to discontinuation | 0 | 0 | 0 | 0 | 0 |
| No. of Subjects with TEAEs leading to discontinuation | 0 | 0 | 0 | 0 | 0 |

Note: TEAE = treatment emergent adverse events; serious TEAEs (SAEs) = serious adverse event

Events with missing severity were imputed as severe. Events with missing relationship were imputed as probably related. Percentages are based on subjects in the Safety Population. For subject counts, if a subject experienced one or more events, they were counted only once.


<sup>&</sup>lt;sup>1</sup> A TEAE is defined as any new AE or an existing AE that worsens in severity during or after study drug administration.

<sup>&</sup>lt;sup>2</sup> Treatment related TEAEs are defined as TEAEs with relationship of "probably" or "possibly" related.

Table 3. Summary of TEAEs by MedDRA SOC/PT (CA-PS-201)

| | | | Placebo | | |
|---|---|---|---|---|---|
| No. of Subjects<br>TEAEs. | Total (N=147) | 0.7 mg (0.05 mg/mL)<br>N=36<br>n (%) | 2.1 mg (0.15 mg/mL)<br>N=36<br>n (%) | 4.2 mg (0.3 mg/mL)<br>N=37<br>n (%) | (Standard of care alone)<br>N=38<br>n (%) |
| No. of TEAEs | 287 | 69 | 82 | 76 | 60 |
| No. of Subjects with any<br>TEAE <sup>1</sup> | 106 (72.1%) | 27 (75.0%) | 28 (77.8%) | 26 (68.4%) | 25 (67.6%) |
| Cardiac disorders | 6 (4.1%) | 1 (2.8%) | 2 (5.6%) | 3 (7.9%) | 0 |
| Angina | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Bradycardia | 2 (1.4%) | 0 | 1 (2.8%) | 1 (2.6%) | 0 |
| Sinus tachycardia | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Tachycardia | 2 (1.4%) | 0 | 0 | 2 (5.3%) | 0 |
| Eye disorders | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Eye hematoma | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Gastrointestinal disorders | 41 (27.9%) | 8 (22.2%) | 10 (27.8%) | 10 (26.3%) | 13 (35.1%) |
| Abdominal pain | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Abdominal pain upper | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Constipation | 10 (6.8%) | 3 (8.3%) | 2 (5.6%) | 1 (2.6%) | 4 (10.8%) |
| Diarrhea | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Dyspepsia | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Flatulence | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Nausea | 29 (19.7%) | 6 (16.7%) | 7 (19.4%) | 7 (18.4%) | 9 (24.3%) |
| Paresthesia oral | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Stomatitis | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Vomiting | 12 (8.2%) | 1 (2.8%) | 4 (11.1%) | 3 (7.9%) | 4 (10.8%) |
| General disorders and administrative site conditions | 20 (13.6%) | 6 (16.7%) | 3 (8.3%) | 5 (13.2%) | 6 (16.2%) |
| Administrative site warmth <sup>2</sup> | 2 (1.4%) | 1 (2.8%) | 0 | 1 (2.6%) | 0 |
| Application site pain <sup>3</sup> | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Application site rash <sup>4</sup> | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Chills | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Feeling hot <sup>5</sup> | 6 (4.1%) | 1 (2.8%) | 2 (5.6%) | 1 (2.6%) | 2 (5.4%) |
| Impaired healing | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |


| Infusion site edema <sup>6</sup> | 6 (4.1%) | 3 (8.3%) | 0 | 1 (2.6%) | 2 (5.4%) |
|---|---|---|---|---|---|
| | | 1 (2.8%) | _ | 0 | ( / |
| Infusion site pain <sup>7</sup> | 3 (2.0%) | (, | 1 (2.8%) | | 1 (2.7%) |
| Edema peripheral <sup>8</sup> | 2 (1.4%) | 0 | 0 | 2 (5.3%) | 0 |
| Pain <sup>9</sup> | 4 (2.7%) | 1 (2.8%) | 1 (2.8%) | 1 (2.6%) | 1 (2.7%) |
| Infections and infestations | 9 (6.1%) | 0 | 5 (13.9%) | 3 (7.9%) | 1 (2.7%) |
| Cellulitis | 3 (2.0%) | 0 | 1 (2.8%) | 1 (2.6%) | 1 (2.7%) |
| Pharyngitis | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Post procedural cellulitis | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Post procedural infection | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Post procedural wound infection | 3 (2.0%) | 0 | 1 (2.8%) | 1 (2.6%) | 1 (2.7%) |
| Tooth infection | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Injury, poisoning and procedural complications | 18 (12.2%) | 3 (8.3%) | 5 (13.9%) | 3 (7.9%) | 7 (18.9%) |
| Foot fracture | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Incision site erythema <sup>10</sup> | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Incision site hematoma <sup>11</sup> | 2 (1.4%) | 1 (2.8%) | 1 (2.8%) | 0 | 0 |
| Scar <sup>12</sup> | 1 (0.7%) | 11 (2.8%) | 0 | 0 | 0 |
| Wound <sup>13</sup> | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Wound dehiscence <sup>14</sup> | 15 (10.2%) | 2 (5.6%) | 5 (13.9%) | 3 (7.9%) | 5 (13.5%) |
| Investigations | 7 (4.8%) | 2 (5.6%) | 2 (5.6%) | 3 (7.9%) | 0 |
| Alanine aminotransferase<br>increased <sup>15</sup> | 3 (2.0%) | 0 | 0 | 3 (7.9%) | 0 |
| Aspartate aminotransferase<br>increased 15 | 3 (2.0%) | 0 | 0 | 3 (7.9%) | 0 |
| Blood glucose increased | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Blood pressure increased | 2 (1.4%) | 2 (5.6%) | 0 | 0 | 0 |
| Body temperature increased | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Gamma-glutamyltransferase<br>increased | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Metabolism and nutrition disorders | 3 (2.0%) | 0 | 1 (2.8%) | 2 (5.3%) | 0 |
| Decreased appetite | 3 (2.0%) | 0 | 1 (2.8%) | 2 (5.3%) | 0 |
| Musculoskeletal and connective tissue disorder | 17 (11.6%) | 7 (19.4%) | 5 (13.9%) | 4 (10.5%) | 1 (2.7%) |


| Arthralgia | 2 (1.4%) | 1 (2.8%) | 1 (2.8%) | 0 | 0 |
|---|---|---|---|---|---|
| Back pain | 4 (2.7%) | 2 (5.6%) | 0 | 2 (5.3%) | 0 |
| Joint stiffness | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Limb discomfort16 | 2 (1.4%) | 2 (5.6%) | 0 | 0 | 0 |
| Muscle spasms <sup>17</sup> | 3 (2.0%) | 0 | 3 (8.3%) | 0 | 0 |
| Muscle twitching <sup>18</sup> | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Musculoskeletal pain <sup>19</sup> | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Musculoskeletal stiffness <sup>20</sup> | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Neck pain | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Pain in extremity <sup>21</sup> | 4 (2.7%) | 1 (2.8%) | 0 | 2 (5.3%) | 1 (2.7%) |
| Nervous system disorders | 53 (36.1%) | 17 (47.2%) | 14 (38.9%) | 14 (36.8%) | 8 (21.6%) |
| Burning sensation | 4 (2.7%) | 2 (5.6%) | 0 | 2 (5.3%) | 0 |
| Dizziness | 12 (8.2%) | 4 (11.1%) | 5 (13.9%) | 1 (2.6%) | 2 (5.4%) |
| Headache | 28 (19.0%) | 7 (19.4%) | 8 (22.2%) | 7 (18.4%) | 6 (16.2%) |
| Hyperesthesia | 2 (1.4%) | 1 (2.8%) | 0 | 1 (2.6%) | 0 |
| Hypoesthesia | 2 (1.4%) | 0 | 1 (2.8%) | 1 (2.6%) | 0 |
| Paresthesia | 3 (2.0%) | 1 (2.8%) | 0 | 1 (2.6%) | 1 (2.7%) |
| Presyncope | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Somnolence | 6 (4.1%) | 2 (5.6%) | 0 | 2 (5.3%) | 2 (5.4%) |
| Syncope | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Psychiatric disorders | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Depressed mood | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Renal and urinary disorders | 4 (2.7%) | 0 | 4 (11.1%) | 0 | 0 |
| Polyuria | 4 (2.7%) | 0 | 4 (11.1%) | 0 | 0 |
| Urge incontinence | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Reproductive system and breast disorders | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Vaginal hemorrhage | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Respiratory, thoracic and mediastinal disorders | 6 (4.1%) | 3 (8.3%) | 0 | 3 (7.9%) | 0 |
| Dysphonia | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Hypoxia | 4 (2.7%) | 2 (5.6%) | 0 | 2 (5.3%) | 0 |
| Rhinorrhea | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Skin and subcutaneous | 13 (8.8%) | 2 (5.6%) | 4 (11.1%) | 1 (2.6%) | 6 (16.2%) |


| tissue disorders | | | | | |
|---|---|---|---|---|---|
| Dermatitis | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Dry skin | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Hyperhidrosis <sup>22</sup> | 4 (2.7%) | 2 (5.6%) | 0 | 0 | 2 (5.4%) |
| Petechiae | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Pruritus <sup>23</sup> | 3 (2.0%) | 0 | 1 (2.8%) | 0 | 2 (5.4%) |
| Rash <sup>24</sup> | 2 (1.4%) | 0 | 0 | 0 | 2 (5.4%) |
| Rash erythematous <sup>25</sup> | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Skin maceration | 3 (2.0%) | 0 | 1 (2.8%) | 0 | 2 (5.4%) |
| Surgical and medical procedures | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Wound drainage | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Vascular disorders | 9 (6.1%) | 2 (5.6%) | 3 (8.3%) | 4 (10.5%) | 0 |
| Deep vein thrombosis | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Diastolic hypotension | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Hot flush <sup>26</sup> | 2 (1.4%) | 0 | 0 | 2 (5.3%) | 0 |
| Hypertension | 2 (1.4%) | 0 | 0 | 2 (5.3%) | 0 |
| Hypotension | 2 (1.4%) | 0 | 2 (5.6%) | 0 | 0 |
| Thrombophlebitis | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |

Abbreviations: Related = possibly or probably related; TEAE = treatment emergent adverse event, SOC = System Organ Class, PT = Preferred Term.

- A TEAE is defined as any new AE or an existing AE that worsens in severity during or after study drug administration. At each level of summarization (SOC or PT), subjects who experienced more than one TEAE were only counted once. All adverse events were coded using MedDRA, Version 21.0. Percentages are based on the number of subjects in the Safety Population. Many of the preferred terms chosen by investigators were vague and, in these cases, the verbatim terms are noted below for these.
- "Administration site warmth": Two cases with the verbatim terms "warm feeling on surgical foot" and "warmth top of surgical foot".
- "Application site pain": One case with the verbatim term "burning sensation at L foot surgical site"
- "Application site rash": One case with the verbatim term "rash on both arms from tape"
- "Feeling hot": Six cases with the following verbatim terms:
  - a. "feeling hot" from 32h to 33h post study treatment
  - b. "generalized warm feeling all over body" from days 5-11 post study treatment
  - "warm sensation lower torso" from 17.6h to 96.6h post study treatment
  - d. "warmth at neck area" from 0.9h to 1.2h post study treatment

  - e. "feeling hot" from 18.7h-24.4h post study treatment f. "feeling hot" from 51.9h-54.4h post study treatment
- "Infusion site edema": Six cases with the following verbatim terms:
  - a. "edema at left hand IV site
  - b. "edema left arm proximal to AC IV site"
  - c. "edema distal to left hand IV site"
  - d. "edema at left forearm IV site"
  - e. "edema on right hand at IV site"
- f. "edema left wrist at IV site"
- 7. "Infusion site pain": Three cases with the following verbatim terms:
  - a. "soreness at left hand IV site"

- b. "stinging sensation at IV site upon attempting to flush"
- c. "pain left wrist at IV site"
- \*Edema peripheral": Two cases with the verbatim terms "right forearm edema proximal to IV site" and "moderate edema right foot"
- "Pain": Four cases with the following verbatim terms:
  - a. "stinging sensation on the dorsal aspect of the left foot" (the operated foot: one event on day 11 and one on day 13)
  - b. "intermittent generalized body aches"
  - c. "increased pain in right foot after putting pressure on toes"
  - d. "worsening of post operative pain"
- 10. "Incision site erythema": one case with the verbatim term "erythema dorsum right foot over 3-4 metatarsal retention incision" noted on days 10-14
  - "Incision site hematoma": two cases with the verbatim terms "superficial hematoma at surgical site" noted on days 10-17 post study treatment, and "superficial hematoma at incision" on days 9-16 post study treatment.
- 12. "Scar": One case with the verbatim term "full thickness fibrotic tissue proximal to the surgical site". The PI at this site noted that the individual who was performing surgical site assessments did not characterize findings as "typical" for the surgery and therefore not an AE or "atypical" and thus an AE.
- 13. "Wound": One case with the verbatim term "full thickness open wound at incision" noted on day 29 post study treatment and treated with wound debridement and resolved by day 58.
- "Wound dehiscence": Each site was instructed to capture "atypical" findings at the surgical site as an AE with "atypical" being a finding different than what is normally seen with this type of surgery. All wound dehiscence cases were identified at site 102. The PI at this site noted that the individual who was performing surgical site assessments did not characterize findings as typical for the surgery (therefore not an AE) or atypical and thus designated as an AE, but instead captured all findings as an AE. Once the PI realized this, the individual was removed from study assessments. Unfortunately, this occurred after database lock and could not be adjusted. The PI noted that in retrospect the cases were mild in severity and most were likely typical for the type of surgery (examples 1-2 mm of wound puckering, a stitch showing or similar minor issues).
- 18. "ALT or AST increased": As can be seen, these 3 cases of each were captured in the CA-008 4.2 mg group. At site 102, 2 of the transaminase elevations were captured as related AEs. Subject 102-060 had "mild" increases in ALT 147 (4.6 X ULN) and AST 88 (2.2 X ULN) at the T96h assessment. They resolved without treatment and returned to normal by day 16. Subject 102-068 had "severe" increase in ALT 170 (5.3 X ULN) and "moderate" increase in AST 140 (3.5 X ULN). They resolved without treatment and returned to normal by day 15. While these were the only 2 related AEs captured for transaminases, Subject 102-053 had mild and unlikely related elevations ALT/AST were 51 (1.6X ULN)/41 (1.03X ULN) at T96h and an Alk Phos elevation 142 (1.2X ULN). Additionally, there were 3 cases in the CA-008 0.7 mg group, 2 in the 2.1 mg group, 2 other cases in the 4.2 mg group, and 3 cases in the placebo group (one of which was a 9X increase from baseline value), respectively, that were normal at baseline and because elevated at T96h, but not captured as TEAEs. Additionally, there were 2, 3 and 2 cases, respectively, in the CA-008 0.7, 2.1 and 4.2 mg groups, where the transaminases were elevated at screening, but became normal at T96h.
- 16. "Limb discomfort": Two cases with the verbatim terms "pressure on plantar aspect of left foot" and "discomfort on dorsal aspect of left foot" (the operated foot in each case).
- 17. "Muscle spasm": Three cases with the following verbatim terms:
  - a. "bilateral leg cramps"
  - b. "muscle spams in neck and upper back"
  - c. "muscle spams in left side of hip"
  - d. "cramping in left calf"
- 18. "Muscle twitching": One case with the verbatim term "left shoulder twitching"
- 19. "Musculoskeletal pain": One case with the verbatim term "pain, right buttocks"
- 20. "Musculoskeletal stiffness": One case with the verbatim term "stiff neck"
- 21. "Pain in extremity": Four cases with the following verbatim terms:
  - "pain on top of left foot"
  - b. "left foot pain"
  - c. "right heel pain'
  - d. "severe pain in right surgical foot".
- 22. "Hyperhidrosis": Four cases with the following verbatim terms:
  - a. "diaphoresis" from 19.7h to 19.8h post study treatment
    - b. "diaphoresis" from 12.7h to 87.7h post study treatment
    - c. "intermittent diaphoresis" from 7.2h to 33.3h post study treatment
    - d. "intermittent diaphoresis" from 51.9h to 54.4h post study treatment
- 23. "Pruritus": Three cases with the following verbatim terms:
  - "pruritus dorsal aspect of left foot" from 78.3h to 96.3h post study treatment
  - b. "right foot pruritis [sic]" from 39.9h to 40.9h post study treatment
  - c. "pruritis [sic] on left hand from 20.3h to 90.3h post study treatment
- 24. "Rash": Two cases with the verbatim terms "rash (back)" and "rash of left hand"
- 25. "Rash erythematous": One case with the following verbatim term: "erythematic rash on foot"
- 26. "Hot flush": One case with the verbatim term "hot flash" from 19.1h to 23.9h post study treatment

Source: Post-text Table TBD (Subject Listing TBD)

Table 4. Summary of Related TEAEs by MedDRA SOC/PT

| | | | CA-008 | | Placebo |
|---|---|---|---|---|---|
| No. of Subjects | Total (N=147) | 0.7 mg (0.05 mg/mL) | 2.1 mg (0.15 mg/mL) | 4.2 mg (0.3 mg/mL) | (Standard of care alone) |
| TEAEs | 10tai (11–147) | N=36 | N=36 | N=37 | N=38 |
| | | N (%) | N (%) | N (%) | N (%) |
| No. of Subjects with any related TEAE <sup>1</sup> | 28 (19.0%) | 7 (19.4%) | 7 (19.4%) | 7 (18.4%) | 7 (18.9%) |
| Gastrointestinal disorders | 3 (2.0%) | 0 | 1 (2.8%) | 0 | 2 (5.4%) |
| Nausea | 2 (1.4%) | 0 | 1 (2.8%) | 0 | 1 (2.7%) |
| Paresthesia oral | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Vomiting | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| General disorders and administrative site conditions | 3 (2.0%) | 2 (5.6%) | 0 | 0 | 1 (2.7%) |
| Administrative site warmth <sup>2</sup> | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Impaired healing | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Pain <sup>3</sup> | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Infections and infestations | 2 (1.4%) | 0 | 1 (2.8%) | 1 (2.6%) | 0 |
| Cellulitis | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Post procedural cellulitis | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Injury, poisoning and procedural complications | 5 (3.4%) | 1 (2.8%) | 0 | 0 | 4 (10.8%) |
| Incision site erythema <sup>4</sup> | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Scar <sup>5</sup> | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Wound dehiscence <sup>6</sup> | 3 (2.0%) | 0 | 0 | 0 | 3 (8.1%) |
| Investigations | 2 (1.4%) | 0 | 0 | 2 (5.3%) | 0 |
| Alanine aminotransferase increased <sup>7</sup> | 2 (1.4%) | 0 | 0 | 2 (5.3%) | 0 |
| Aspartate aminotransferase increased <sup>7</sup> | 2 (1.4%) | 0 | 0 | 2 (5.3%) | 0 |


| Musculoskeletal and connective tissue disorder | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
|---|---|---|---|---|---|
| Limb discomfort8 | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Nervous system disorders | 11 (7.5%) | 3 (8.3%) | 2 (5.6%) | 5 (13.2%) | 1 (2.7%) |
| Burning sensation | 4 (2.7%) | 2 (5.6%) | 0 | 2 (5.3%) | 0 |
| Headache | 4 (2.7%) | 1 (2.8%) | 1 (2.8%) | 2 (5.3%) | 0 |
| Hypoesthesia | 2 (1.4%) | 0 | 1 (2.8%) | 1 (2.6%) | 0 |
| Paresthesia | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Renal and urinary disorders | 3 (2.0%) | 0 | 3 (8.3%) | 0 | 0 |
| Polyuria | 3 (2.0%) | 0 | 3 (8.3%) | 0 | 0 |
| Urge incontinence | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Respiratory, thoracic and mediastinal disorders | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Rhinorrhea | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Skin and subcutaneous tissue disorders | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Pruritus <sup>9</sup> | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Skin maceration | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Vascular disorders | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Hot flush <sup>10</sup> | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |

Abbreviations: Related = possibly or probably related; TEAE = treatment emergent adverse event, SOC = System Organ Class, PT = Preferred Term.

- 1. A TEAE is defined as any new AE or an existing AE that worsens in severity during or after study drug administration. At each level of summarization (SOC or PT), subjects who experienced more than one TEAE were only counted once. All adverse events were coded using MedDRA, Version 21.0. Percentages are based on the number of subjects in the Safety Population.
- 2. "Administration site warmth": One case with the verbatim term "warm feeling on surgical foot" which lasted 3.5h 15.9h post study treatment
- 3. "Pain": One case with the verbatim term "worsening of post operative pain" required medication and physical therapy
- 4. "Incision site erythema": One case with the verbatim term "erythema dorsum right foot over 3-4 metatarsal retention incision" noted on days 10-14
- s. "Scar": One case with the verbatim term "full thickness fibrotic tissue proximal to the surgical site". The PI at this site noted that the individual who was performing surgical site assessments did not characterize findings as "typical" for the surgery and therefore not an AE or "atypical" and thus an AE.
- 6. "Wound dehiscence": Each site was instructed to capture "atypical" findings at the surgical site as an AE with "atypical" being a finding different than what is normally seen with this type of surgery. All wound dehiscence cases were identified at site 102. The PI at this site noted that the individual who was performing surgical site assessments did not characterize findings as typical for the surgery (therefore not an AE) or atypical and thus designated as an AE, but instead captured all findings as an AE. Once the PI realized this, the individual was removed from study assessments. Unfortunately, this occurred after database lock and could not be adjusted. The PI noted that in retrospect the cases were mild in severity and most were likely typical for the type of surgery (examples 1-2 mm of wound puckering, a stitch showing or similar minor issues).
- "ALT or AST increased": As can be seen, these 3 cases of each were captured in the CA-008 4.2 mg group. At site 102, 2 of the transaminase elevations were captured as related AEs. Subject 102-060 had "mild" increases in ALT 147 (4.6 X ULN) and AST 88 (2.2 X ULN) at the T96h assessment. They resolved without treatment and returned to normal by day 16. Subject 102-068 had "severe" increase in ALT 170 (5.3 X ULN) and "moderate" increase in AST 140 (3.5 X ULN). They resolved without treatment and returned to normal by day 15. While these were the only 2 related AEs captured for transaminases, Subject102-053 had mild and unlikely related elevations ALT/AST were 51 (1.6X ULN)/41 (1.03X ULN) at T96h and an Alk Phos elevation 142 (1.2X ULN). Additionally, there were 3 cases in the CA-008 0.7 mg group, 2 other cases in the 4.2 mg group, and 3 cases in the placebo group (one of which was a 9X increase from baseline value), respectively, that were normal at baseline and because elevated at T96h, but not captured as TEAEs. Additionally, there were 2, 3 and 2 cases, respectively, in the CA-008 0.7, 2.1 and 4.2 mg groups, where the transaminases were elevated at screening, but became normal at T96h.
- 8. "Limb discomfort": while it was the preferred term chosen, the verbatim description was "discomfort on dorsal aspect of left foot" (the operated foot).
- 9. "Pruritus": One case with the following verbatim term: "right foot pruritis [sic]" from 39.9h to 40.9h post study treatment
- 10. "Hot flush": One case with the verbatim term "hot flash" from 19.1h to 23.9h post study treatment

Table 5. Summary of Related TEAEs by Frequency

| | T-4-1 | | Placebo | | |
|---|---|---|---|---|---|
| No. of Subjects | Total<br>(N=147) | 0.7 mg (0.05 mg/mL)<br>N (%) | 2.1 mg (0.15 mg/mL)<br>N (%) | 4.2 mg (0.3 mg/mL)<br>N (%) | (Standard of care alone)<br>N (%) |
| No. of TEAEs | 287 | 69 | 82 | 76 | 60 |
| No. of Subjects with any TEAE <sup>1</sup> | 106<br>(72.1%) | 27 (75.0%) | 28 (77.8%) | 26 (68.4%) | 25 (67.6%) |
| No. of "Related" AEs | 43 | 8 | 11 | 14 | 10 |
| No. of Subjects with any<br>"Related" TEAE | 28 (19.1%) | 7 (19.4%) | 7 (19.4%) | 7 (18.4%) | 7 (18.9%) |
| Burning sensation | 4 (2.7%) | 2 (5.6%) | 0 | 2 (5.3%) | 0 |
| Headache | 4 (2.7%) | 1 (2.8%) | 1 (2.8%) | 2 (5.3%) | 0 |
| Polyuria | 3 (2.0%) | 0 | 3 (8.3%) | 0 | 0 |
| Wound dehiscence | 3 (2.0%) | 0 | 0 | 0 | 3 (8.1%) |
| Alanine transaminase increase | 2 (1.4%) | 0 | 0 | 2 (5.3%) | 0 |
| Aspartate transaminase increase | 2 (1.4%) | 0 | 0 | 2 (5.3%) | 0 |
| Hypoesthesia | 2 (1.4%) | 0 | 1 (2.8%) | 1 (2.6%) | 0 |
| Nausea | 2 (1.4%) | 0 | 1 (2.8%) | 0 | 1 (2.7%) |
| Administration site warmth | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Cellulitis | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Hot flush | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Impaired healing | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Incision site erythema | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Limb discomfort | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Pain | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Paresthesia | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Paresthesia oral | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Pruritus | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Rhinorrhea | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Scar | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Skin maceration | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Urge incontinence | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Vomiting | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |


Abbreviations: Related = possibly or probably related; TEAE = treatment emergent adverse event, SOC = System Organ Class, PT = Preferred Term.

<sup>1</sup>A TEAE is defined as any new AE or an existing AE that worsens in severity during or after study drug administration. At each level of summarization (SOC or PT), subjects who experienced more than one TEAE were only counted once. All adverse events were coded using MedDRA, Version 21.0. Percentages are based on the number of subjects in the Safety Population.

**Table 6. Summary of Related Local TEAEs by Frequency** 

| | Tetal | | | Placebo | |
|---|---|---|---|---|---|
| No. of Subjects | Total<br>(N=147) | 0.7 mg (0.05 mg/mL)<br>N (%) | 2.1 mg (0.15 mg/mL)<br>N (%) | 4.2 mg (0.3 mg/mL)<br>N (%) | (Standard of care alone)<br>N (%) |
| No. of TEAEs | 287 | 69 | 82 | 76 | 60 |
| No. of Subjects with any TEAE <sup>1</sup> | 106<br>(72.1%) | 27 (75.0%) | 28 (77.8%) | 26 (68.4%) | 25 (67.6%) |
| No. of "Related" AEs | 43 | 8 | 11 | 14 | 10 |
| No. of Subjects with any<br>"Related" TEAE | 28 (19.1%) | 7 (19.4%) | 7 (19.4%) | 7 (18.4%) | 7 (18.9%) |
| Burning sensation | 4 (2.7%) | 2 (5.6%) | 0 | 2 (5.3%) | 0 |
| Wound dehiscence | 3 (2.0%) | 0 | 0 | 0 | 3 (8.1%) |
| Hypoesthesia | 2 (1.4%) | 0 | 1 (2.8%) | 1 (2.6%) | 0 |
| Administration site warmth | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Cellulitis | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Impaired healing | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Incision site erythema | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Limb discomfort | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Pain | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Paresthesia | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |
| Scar | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Skin maceration | 1 (0.7%) | 0 | 0 | 0 | 1 (2.7%) |


Abbreviations: Related = possibly or probably related; TEAE = treatment emergent adverse event, SOC = System Organ Class, PT = Preferred Term.

A TEAE is defined as any new AE or an existing AE that worsens in severity during or after study drug administration. At each level of summarization (SOC or PT), subjects who experienced more than one TEAE were only counted once. All adverse events were coded using MedDRA, Version 21.0. Percentages are based on the number of subjects in the Safety Population.

| | Total | | Placebo | | |
|---|---|---|---|---|---|
| No. of Subjects | Total<br>(N=147) | 0.7 mg (0.05 mg/mL)<br>N (%) | 2.1 mg (0.15 mg/mL)<br>N (%) | 4.2 mg (0.3 mg/mL)<br>N (%) | (Standard of care alone)<br>N (%) |
| No. of TEAEs | 287 | 69 | 82 | 76 | 60 |
| No. of Subjects with any TEAE <sup>1</sup> | 106<br>(72.1%) | 27 (75.0%) | 28 (77.8%) | 26 (68.4%) | 25 (67.6%) |
| Burning sensation | 2 (1.4%) | 1 (2.8%) | 0 | 1 (2.6%) | 0 |
| Alanine aminotransferase increased | 1 (0.7%) | 0 | 0 | 1 (2.6%) | 0 |
| Deep vein thrombosis | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |
| Dizziness | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Hyperhidrosis | 1 (0.7%) | 1 (2.8%) | 0 | 0 | 0 |
| Sinus tachveardia | 1 (0.7%) | 0 | 1 (2.8%) | 0 | 0 |

Table 7. Summary of Severe TEAEs by Frequency

Abbreviations: Related = possibly or probably related; TEAE = treatment emergent adverse event, SOC = System Organ Class, PT = Preferred Term.

# 5.4. Study Rationale

CA-008 is being investigated as a potential therapy for treatment of pain following surgery.

#### 5.5. Dose Rationale

#### **5.5.1.** Selection of Doses

The safety of CA-008 was established in relevant animal models and supported by two studies after bunionectomy (CA-PS-2017-101 and CA-PS-201) and knowledge from prior human studies with an injectable formulation of capsaicin. Taken together, the characterization of the pharmacology, pharmacokinetics, and toxicology profiles are considered sufficient to support the intended use of CA-008 in this study.

### 5.5.2. Selection and Timing of Dose

CA-008 is a pH labile prodrug of capsaicin that rapidly releases capsaicin after administration into tissue. Decision for single administration at the time of surgery is based on capsaicin's mechanism of action. Capsaicin exposure results in initial excitation followed by a functional desensitization of TRPV-1-expressing nociceptors which continues for some time after removal capsaicin from the site. Administration while the patient is under anesthesia for the procedure supplemented by a regional local anesthetic block or local anesthetic infiltration of the surgical site should sufficiently address any transient pain that results from TRPV1 agonism. Administration of CA-008 during the wound closure process is ideal for delivering therapy to the surgical site, thus optimizing target engagement. During closure, the surgical tissue is exposed and visible which allows for complete and adequate delivery of CA-008 (and capsaicin) to the potential areas where noxious pain is generated.


<sup>&</sup>lt;sup>1</sup>A TEAE is defined as any new AE or an existing AE that worsens in severity during or after study drug administration. At each level of summarization (SOC or PT), subjects who experienced more than one TEAE were only counted once. All adverse events were coded using MedDRA, Version 21.0. Percentages are based on the number of subjects in the Safety Population.

#### 6. STUDY OBJECTIVES

# 6.1. Pilot (Exploratory) Stage of the Study

### 6.1.1. Primary Objectives

• To evaluate the efficacy of a single intraoperative administration of CA-008 vs. placebo (100 mL volume) in subjects undergoing an elective TKA.

Note that in the pilot stage cohort #1 evaluates 5 mg CA-008 vs. placebo (100 mL volume). For cohort #2, CA-008 10 mg will be evaluated vs. placebo (100 mL volume) and in cohort #3, CA-008 15 mg will be evaluated vs. placebo (100 mL volume).

#### 6.1.2. Secondary Objectives

- To evaluate the safety and tolerability of a single intraoperative administration of CA-008 vs. placebo in subjects undergoing an elective TKA.
- To evaluate the PK profile of a single intraoperative administration of CA-008 in subjects undergoing an elective TKA.
- To evaluate the opioid-sparing effect of CA-008 vs. placebo in subjects undergoing an elective TKA.

# **6.2.** Second (Parallel Design) Stage of the Study

### 6.2.1. Primary Objectives

• After an interim unblinded analysis of the pilot stage of the study, to evaluate the efficacy of a single intraoperative administration of CA-008 vs. placebo in subjects undergoing an elective TKA

Note that for the second (parallel design) stage, an amendment will be performed after receiving the cohort #3 results from the pilot stage. This amendment will designate the number and doses of active treatment groups, and volume to be used for active and placebo groups.

#### 6.2.2. Secondary Objectives

- To evaluate the safety and tolerability of a single intraoperative administration of CA-008 vs. placebo in subjects undergoing an elective TKA.
- To determine the efficacy of various doses of CA-008 vs. placebo administered intraoperatively in subjects undergoing an elective TKA.
- To evaluate the PK profile of a single intraoperative administration of CA-008 in subjects undergoing an elective TKA


# **6.2.3.** Exploratory Objective

 Pharmacoeconomic benefits from administration of CA-008 vs. placebo in subjects undergoing an elective TKA.


#### 7. INVESTIGATIONAL PLAN

# 7.1. Overall Study Design and Plan

This is a Phase 2, multi-center, randomized, double-blind, placebo-controlled, two stage study (exploratory pilot stage followed by a parallel design stage) evaluating a single dose of CA-008 vs. placebo injected/instilled during an elective TKA.

The choice between the two doses of CA-008 for cohort #1 of the pilot stage of the study was based upon the topline results from the Phase 2 bunionectomy study. Additionally, two more pilot stage cohorts will be added.

After an interim unblinded analysis of the pilot stage results (cohorts #1 through #3), a second stage will be performed with dose and volume levels, sample size and number of CA-008 treatment groups vs. placebo to be determined.

For each subject, the postoperative assessments will be conducted in two parts:

- Inpatient period which starts with completion of study treatment injection (T0) and continues through 96h (T96h).
- Outpatient period which begins on discharge from the inpatient unit through various follow-up visits to day 29 (D29±2) (W4) after surgery or later if necessary for ongoing safety assessments. Note that additional follow up visits could occur after D29/W4 to follow adverse events (AEs) to resolution or establishment of a new baseline.

# 7.2. Duration of Participation

Each subject is expected to be in the study up to 76 days (screening through end-of-study visit).

# 7.3. Study Stopping Rules

Study enrollment will be paused if subjects experience intolerable possibly related TEAEs (shown in Table 8) as defined:

- 1 or more subjects with any grade 4 "related" TEAE in any of the categories
- 2 or more subjects with the same grade 3 "related" TEAE in any of the categories

Refer to Table 8 below for descriptions/definitions of AE severity grading.

An external independent Safety Review Committee (SRC) will be consulted should a stopping rule be triggered to determine whether it is appropriate to continue with dosing in the study. This committee will be independent of the Sponsor or CRO and will in no way be involved with study conduct. The SRC Charter details the membership, roles and responsibilities of the SRC.


**Table 8.** Study Stopping Rules

| Category | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Abnormal<br>Wound Healing:<br>Infection<br>Dehiscence<br>Necrosis | Mild symptoms;<br>clinical or diagnostic<br>observations only;<br>intervention not<br>indicated. No<br>interference with age-<br>appropriate<br>instrumental ADL | Minimal, local or<br>noninvasive<br>intervention<br>indicated; May<br>require local wound<br>care or medical<br>intervention (e.g.,<br>dressings or topical<br>medications) | Severe or medically significant but not immediately lifethreatening; hospitalization or prolongation of existing hospitalization indicated; limiting ADLs. May require IV antibiotics, antifungals, or antivirals or radiologic intervention. | Life-threatening consequences; urgent intervention indicated |
| ECG/Cardiac<br>issues<br>Vital Signs<br>Labs | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Severe or medically significant but not immediately lifethreatening; hospitalization or prolongation of existing hospitalization indicated | Life-threatening<br>consequences;<br>urgent intervention<br>indicated |
| Focused Neurosensory Testing (performed by trained Investigator) | Mild symptoms | Moderate symptoms;<br>limiting instrumental<br>ADL | Severe symptoms requiring medical intervention; limiting self-care ADL | Life-threatening and<br>urgent<br>intervention<br>indicated |


#### 8. SELECTION OF STUDY POPULATION

## 8.1. Study Population

The study population consists of adults, aged 18-80 years old inclusive, who are undergoing elective TKA.

#### 8.1.1. Number of Participants

Pilot (exploratory) Stage:

- Cohort #1: N=18 randomized 1:1, CA-008 vs. placebo
- Cohort #2: N=18 randomized 2:1, CA-008 vs. placebo, respectively
- Cohort #3: N=18 randomized 2:1, CA-008 vs. placebo, respectively

A second (parallel design) stage of the study is anticipated with a much larger sample size to be determined after an interim analysis of the pilot stage cohort #3 is conducted.

# 8.2. Eligibility Criteria

#### 8.2.1. Inclusion Criteria

Subjects must meet all of the following criteria to be considered eligible to participate in the study:

- 1. Plan to undergo an elective primary unilateral total knee arthroplasty (TKA or knee replacement), without collateral procedure or additional surgeries.
- 2. In the medical judgment of the investigator, be an adult aged 18 80 years old, inclusive, and American Society of Anesthesiology (ASA) physical Class 1, 2 or 3 at the time of randomization (Section 17.1 Appendix A).
- 3. If a male, unless he has a same sex partner, be either sterile (surgically **or** biologically) or commit to an acceptable method of birth control while participating in the study. The site personnel will provide instructions on what is an acceptable method.
- 4. If a female, must meet all of the following:
  - a. A female of child-bearing potential (FCBP) must have a negative serum pregnancy test at screening and negative urine pregnancy test before surgery;
  - b. No plan to become pregnant or to breast feed during the study; and
  - c. Be surgically sterile or at least one year post-menopausal, have a monogamous partner who is surgically sterile, have a same sex partner or (**one** of the following must apply)
    - i. is practicing double-barrier contraception
    - ii. is practicing abstinence (must agree to use double-barrier contraception in the event of sexual activity)
    - iii. is using an insertable, injectable, transdermal or combination oral


contraceptive approved by the FDA for at least 2 months prior to screening and commits to the use of an acceptable form of birth control while participating in the study.

- 5. Have a body mass index  $\leq$  36 kg/m<sup>2</sup>.
- 6. Be willing and able to sign the informed consent form (ICF) approved by an Institutional Review Board (IRB).
- 7. Be willing and able to complete study procedures and pain scales and to communicate meaningfully in English or Spanish with study personnel and return for outpatient follow up visits as required.

#### 8.2.2. Exclusion Criteria

Subjects will not be eligible to participate in this study if any one of the following exclusion criteria is met:

- 1. In the opinion of the Investigator,
  - a. have a concurrent painful condition, other than pain in the knee to be replaced, that may require analgesic treatment during the study period or may confound post-surgical pain assessments.
  - b. have active skin disease or other clinically significant abnormality at the anticipated site of surgery that could interfere with the planned surgery.
- 2. Have a known allergy to chili peppers, capsaicin or the components of CA-008, ropivacaine HCl, ketorolac, acetaminophen, fentanyl, hydromorphone, morphine or oxycodone.
- 3. As determined by the investigator (with input from the study's medical monitor if requested by the investigator), have a history or clinical manifestation of significant medical, neuropsychiatric or other condition, including a clinically significant existing arrhythmia, left bundle branch block or abnormal ECG, myocardial infarction or coronary arterial bypass graft surgery within the prior 12 months, significant abnormal clinical laboratory test value, or known bleeding abnormality that could preclude or impair study participation or interfere with study assessments.
- 4. The following are considered disallowed medications:
  - a. Be tolerant to opioids defined as those who have been receiving or have received chronic opioid therapy greater than 15 mg of oral morphine equivalents (Table 9) per day for greater than 3 out of 7 days per week over a one-month period within 6 months of screening.
  - b. Within 1 day prior to surgery and throughout the inpatient period, be taking or using any capsaicin-containing products, such as dietary supplements or over-the-counter (OTC) preparations, including topical formulations, and prescription medications.
  - c. Within the 7 days prior to surgery, be taking any central nervous system (CNS) active agent as an analgesic adjunct medication, such as anticonvulsants,


antidepressants (such as SNRIs, SSRIs, and tricyclic antidepressants), benzodiazepines, sedative-hypnotics, clonidine and other central alpha-2 agents (e.g., tizanidine), ketamine or muscle relaxants. [Note that SNRIs = Serotonin and norepinephrine reuptake inhibitors and SSRI = Selective serotonin reuptake inhibitors.]

- i. These drugs are permitted if prescribed for non pain indications and the dose has been stable for at least 30 days prior to surgery. Note that the dose must remain stable throughout the study.
- ii. If the subject is taking centrally- and/or peripherally-acting analgesic medications, such as acetaminophen, NSAIDs, tramadol or opioids, FOR knee-related pain, the subject may participate in the study if 4(a) above is not applicable and the subject is willing to discontinue these medications 3 days prior to surgery. Note that baby aspirin for cardiovascular prophylaxis is allowed during the study.
- iii. The use of benzodiazepines and the non-benzodiazepines (eszopiclone, ramelteon, zaleplon and zolpidem) are permitted to treat insomnia during the postoperative period.
- d. Within the 7 days prior to the planned surgery and throughout the study, be taking antiarrhythmics except beta-blockers, digoxin, warfarin (see exception below), lithium, or aminoglycosides or other antibiotics for an infection (except for ophthalmic use or for treatment or prophylaxis of postoperative surgical site infections). At the investigator's discretion, agents intended for deep venous thrombosis (DVT) prophylaxis after the surgery is allowed.
- e. Within the 14 days prior to surgery, be taking parenteral or oral corticosteroids (steroid inhaler for allergy or asthma treatment, topical steroid for a non-clinically significant skin condition not involving the area of surgery or ophthalmic steroids are permissible).
- f. Be on an antianginal, antihypertensive agent or diabetic regimen at a dose that has not been stable for at least 30 days or which is not expected to remain stable while participating in the study.
- 5. In the opinion of the Investigator, within the past year have a history of illicit drug use or prescription medicine or alcohol abuse (regularly drinks > 4 units of alcohol per day; where a unit = 8 oz. beer, 3 oz. wine or 1 oz. spirits).
- 6. Have positive results on the alcohol breath test indicative of alcohol abuse or urine drug screen indicative of illicit drug use (unless results can be explained by a current prescription or acceptable over-the-counter medication at screening as determined by the investigator) at screening, and/or prior to surgery. Note that for those subjects who test positive for


- tetrahydrocannabinol (THC), if they are willing to abstain from use or consumption of THC-containing products from 3 days prior to surgery to the day 8 visit, they may be allowed to participate in the study.
- 7. Willing and able to avoid foods containing capsaicin for 24 hours prior to surgery and PK blood draws.
- 8. Have previously participated in a clinical study with CA-008.
- 9. Have participated in another clinical trial or used an investigational product within 30 days or five half-lives (whichever is longer) prior to the planned surgery, or is scheduled to receive an investigational product other than CA-008 while participating in the study.


### 9. STUDY TREATMENTS

## 9.1. Study Treatment

Complete details of study drug packaging, storage, dispensation, preparation and tracking are provided in the pharmacy manual.

#### 9.1.1. CA-008 HCl Description

CA-008, provided as the hydrochloride salt is a white solid, highly soluble in water. It degrades rapidly to capsaicin at neutral pH but is stable for several days at room temperature in aqueous solution at pH~3. Capsaicin is known to be irritating to mucous membranes when aerosolized and is a skin irritant.

## 9.1.2. Study Treatment Description

The active drug product will be provided as CA-008 frozen concentrate solution for injection in a 1.0 mL vial with doses calculated as the freebase.

The placebo comparator is identical in appearance.

The proposed doses of CA-008 to be evaluated in the Pilot Stage of the study are:

- Cohort #1: CA-008 5 mg vs. placebo in 100 mL of vehicle
- Cohort #2: CA-008 10 mg vs. placebo in 100 mL of vehicle
- Cohort #3: CA-008 15 mg vs. placebo in 100 mL of vehicle

An unblinded pharmacist or designee may use unblinded vials identified as to contents. However, at the time of reconstitution, the anesthesia and surgical team and study site personnel will be blinded as to study treatment. At time of use, the concentrate will be completely reconstituted and used for treatment (see the Pharmacy Manual). These details will be reflected in the Unblinding Plan and the Pharmacy Manual.

#### 9.1.3. Study Treatment Storage

Study treatments will be shipped to sites and stored at -20°C (-15°C to -30°C) until the day of surgery. All study treatment should be stored in a secured area and in accordance with the product labeling and all applicable laws, regulations, and local/institutional requirements. A description of storage conditions for all investigational products will be provided in the Pharmacy Manual.

#### 9.1.4. Study Treatment Accountability

All study treatment will be transported, received, stored, and handled strictly in accordance with the container or product label, the instructions provided to the research site, and applicable regulations. Detailed drug accountability records must be maintained, including the dates


shipments are received, the quantity of material received, the dates dispensed and the running inventory. The unused quantities will be returned to the Sponsor's drug supply vendor at the end of the trial. All unused supplies will be checked against the drug accountability records during the study and/or at the end of the study. The Investigator or designee must maintain an inventory record of all dispensed rescue medications to subjects. Additional details are provided in the Pharmacy Manual.

Only eligible subjects participating in the study will receive the study treatment. Only authorized research site staff may supply, prepare or administer the study treatments. Once dispensed, study treatment may not be relabeled or reassigned for use by other subjects.

### 9.1.5. Control of Study Treatment and Rescue Medication

Mishandling, potential theft, significant loss of clinical supplies, including study treatments, systemic analgesia medications and rescue medications at the site, or other suspected diversion must be reported to the Sponsor or designee within 24 hours of first knowledge of the issue. If diversion is confirmed or suspected (e.g., excessive use of rescue medications), the study staff will be required to complete a clinical supply documentation form, including information related to situations in which a subject sold drug or gave drug to a friend or relative, there is a discrepancy in drug accountability and suspected diversion, or a subject had drug stolen, or if there was diversion or theft by site staff or others.

#### 9.2. Other Interventions

#### 9.2.1. Inpatient Analgesia

Within 30 min of anesthesia induction give the subject IV hydromorphone 1.5 mg.

During the surgery, ensure that each subject has received at least 100 mcg of IV fentanyl with adjustments above this dose per anesthesiologist discretion.

Within 15 min of the end of surgery, give the subject IV hydromorphone 0.5 mg

Within 15 min of the end of surgery, administer the following:

- IV ketorolac 30 mg (for example, ketorolac full prescribing information is available at: http://www.sagentpharma.com/wpcproduct/ketorolac-tromethamine-injection-usp/ [Sagent Pharmaceuticals 2018]). Dose adjustments may be made per surgeon/anesthesiologist discretion to accommodate the subject's age and health status.
- IV acetaminophen 1 g (Ofirmev®, Mallinckrodt Pharmaceuticals 2018) full prescribing information at http://ofirmev.com/.


After these non-opioids have been administered, no additional non-opioid analysis are to be administered during the inpatient phase of the study.

## 9.2.2. Inpatient Rescue Medications

After surgery, subjects will be monitored in the post-anesthesia care unit (PACU) for at least 90 min during which time efficacy asssessments can begin once the subject is awake. During this time, IV fentanyl 25-50 mcg q5 min prn for moderate-to-severe pain ( $\geq$  4) as reported by subjects using the 0 to 10 numerical rating scale of current pain intensity (NRS). After discharge from the PACU, subjects are followed through T96h as an inpatient.

From the time of discharge from the PACU through T48h administer IV hydromorphone 0.5 mg q15 min prn for NRS  $\geq$  4 as reported by subjects.

After T12h, administer PO oxycodone 5 mg q2h prn moderate pain (NRS  $\geq$  4 and  $\leq$  6) or 10 mg q2h prn severe pain (NRS  $\geq$  7). From T12 through T48h, IV hydromorphone may be used as rescue in addition to PO oxycodone for moderate-to-severe pain. After T48, only PO oxycodone may be used as rescue. If a subject still requires IV opioid rescue after T48, then the subject should undergo an early termination due to lack of efficacy.

Subjects will be encouraged to rescue only for moderate pain scores (NRS  $\geq$  4), however rescue may be requested at any time and medication will be provided when requested.

## 9.2.3. Outpatient Analgesic Medications

Once discharged from the inpatient unit, all study participants will be instructed to take a combination of over-the-counter (OTC) analgesics at an appropriate dose per medical judgment to manage any residual or breakthrough postsurgical pain.

Outpatient period: after T96h discharge through D29/W4, if needed for pain management, the following oral OTC analgesics will be recommended for subjects to self-administer (note that these medications will not be provided by the sponsor):

- A nonsteroidal anti-inflammatory drug (NSAID) (e.g., ibuprofen 200 mg prn up to qid [Advil® or Motrin®] or naproxen 220 mg prn up to tid [Aleve®]) or other NSAID per investigator discretion and
- Acetaminophen 1000 mg prn up to tid or 650 mg up to qid (3g daily maximum limit)

If a subject is still requiring opioid rescue in the 12h prior to discharge from the inpatient unit (i.e., from T84h on regardless of whether discharge is delayed), then prescribe no more than 9 tablets of oxycodone 5 mg (1 PO tid prn) per investigator discretion for the initial outpatient period. If refills are necessary, an unscheduled visit may be important to understand why there is continued pain, as persistent pain or pain exacerbations during this period may suggest the need to assess the surgical site. If such a situation occurs, the Investigator should use clinical discretion on adequacy of analgesic treatment but capture this event as an AE and document any required treatments.


# 9.3. Method of Assigning Subjects to Treatment Groups

Randomization will be used to avoid bias in the assignment of subjects to treatments, to increase the likelihood that known and unknown subject attributes (e.g., demographics, baseline characteristics) are evenly balanced across treatment groups, and to enhance the validity of statistical comparisons across treatment groups.

Subjects who have provided written informed consent will be assigned a unique number in the screening process. This number will be used to identify the subject throughout the study.

In the Pilot Stage, subjects in each cohort will be randomized to either the active medication or placebo. Subsequently, the number of active treatment groups and sample size will be determined after the interim unblinded analysis of topline data from cohort #3 of the Pilot Stage.

Once any subject number or randomization number is assigned, it cannot be reassigned to any other subject. This study will use manual randomization.

Subjects may be rescreened if the screening window is exceeded due to scheduling issues.

## 9.4. Blinding

To reduce the potential for bias in the study, treatment group assignments will be double-blinded during the study. The subject, investigational site personnel, Sponsor, and Sponsor designees directly involved in the conduct and/or monitoring of this study will not be aware of the treatment group assignments. Note that the placebo is identical in appearance to CA-008 once reconstituted.

Under normal circumstances, the blind will not be broken until all participants have completed treatment. In case of emergency, and only if the information is required by the Investigator to ensure subject's safety in managing a medical condition, the treatment may be unblinded at the site by using a code break module. The code break module will be provided by the Sponsor or designee. If possible, the Investigator should contact the Sponsor prior to unblinding and after any actions have been taken. Whenever a treatment sequence is prematurely unblinded, the reason, date and time of the unblinding, and the individual who broke the blind must be documented. Individual code breaks will result in withdrawal of the participant from the study.

It is assumed that the need to unblind a study subject's treatment assignment will occur in the setting of an SAE, and therefore, all procedures for the reporting of a SAE must be followed.

# 9.5. Prior and Concomitant Therapy

All non-study medications, including prescription, over-the-counter, or herbal therapies, used by the subject will be documented for the 45 days prior to screening and throughout the study. The


Investigator will determine if the prior/concomitant medication(s) affect the subject's eligibility to participate or continue to participate in the study.

On a case-by-case basis, the Investigator is permitted to allow the use of some concomitant medications, for example, to treat an AE, if the Investigator determines that the medication will not affect the subject's safety or study integrity. Wherever possible, the Investigator should obtain approval from the Medical Monitor prior to administering the medication.

## 9.6. Study Restrictions

In addition to the criteria described in Sections 8.2, 9.2, 9.5, and 10.1.2 the subject must agree to abide by the following study restrictions:

Abstain from the following during the inpatient portion of the study:

- consuming any alcohol
- smoking or vaping (nicotine-containing or other substances)
- illicit drug use or non-medical use of therapeutic drugs not allowed by the protocol
- any foods containing capsaicin for 24 hours prior to PK blood draws

Abstain from the following during the outpatient portion of the study:

- Subjects will be asked to abstain from consuming more than 1 (women) or 2 drinks (men) per day of alcohol
- Subjects will be asked to abstain from illicit drug use or non-medical use of therapeutic drugs
- Subjects will be asked to abstain from taking prohibited medications

# 9.7. Treatment Compliance

Because all study medication is being administered by study personnel, no compliance procedures are necessary. Diversion will be monitored and recorded through rescue medication accountability. Any suspected or confirmed diversion will be documented and reported.


#### 10. CONDUCT OF THE STUDY

All study assessments will be performed at the visits and timepoints outlined in the Schedule of Assessments (Table 1); the following sections outline the detailed timing and procedures associated with the visits and assessments.

# 10.1. Study Visits

### **10.1.1.** Screening Phase (Day -45 to Day -1):

Subjects will be screened for participation at the study within 45 days of surgery/study drug administration. The following assessments will be completed:

- Informed Consent
- Inclusion / Exclusion evaluation
- Demographics
- Medical and surgical history
- Prior/current medications
- Complete Physical Exam (PE), including height and weight
- Vital signs including temperature (Section 17.10 Appendix J)
- Baseline neurosensory exam
- Clinical laboratory tests (chemistry/coagulation, hematology, and urinalysis) (Section 17.9 Appendix I)
- Urine Drug Screening (UDS)
- Alcohol breath/saliva test
- Serum Pregnancy test (FCBP), if applicable
- 12-Lead Electrocardiograms (ECG)
- KOOS Survey
- Subject pain assessment training
- Adverse Event (AE) assessment (record any current conditions as medical history)

### 10.1.2. Surgery Phase: Day 1- Prior to surgery (baseline) up to the end of surgery

#### **10.1.2.1. Prior to Surgery (D-1 to D0)**

Subjects who meet the selection criteria at the Screening Visit and are eligible to participate in the study will be required to return to the study center for surgery within 45 days of screening. The following assessments will be performed:

- Confirm informed consent
- Review of Inclusion / Exclusion


- Review of medical and surgical history since screening
- Review of prior and current concomitant medications
- Interim targeted PE with inspection of the planned area of surgery (if not done at Screening visit)
- Urine Pregnancy test (FCBP) if applicable
- UDS
- Alcohol breath/saliva test
- Blood draws and urine collections for PK analyses
- Vital signs and temperature
- Subject pain training review (watch video)
- Randomize to treatment after confirmation of continued eligibility

#### 10.1.2.2. Anesthesia and Surgery

The surgery will be performed under general anesthesia with either supplemented by an adductor canal (AC) block AND an IPACK infiltration (Interspace between the Popliteal Artery and the Capsule of the posterior Knee between the femoral condyles). Recent literature suggests the AC+IPACK approach is the new "best practice" to supplement anesthesia as part of an enhanced recovery after surgery (ERAS) for TKA (Cullom 2017, Sankineani 2018).

Perform the AC+IPACK local anesthetic regional blocks under ultrasound guidance prior to the start of surgery. The dose of IV fentanyl administered during surgery should be 100 to 300 mcg with adjustments per anesthesiologist discretion.

- Using ropivacaine hydrochloride (RopiHCl)
  - o AC block: 20 mL of 0.5% (100 mg)
  - o IPACK infiltration: 20 mL of 0.2% (60 mg)

A tourniquet will be used in all subjects. After exsanguination, but prior to surgical incision, perform surgical site infiltration with RopiHCl 0.2% 30 mL (100 mg).

The total RopiHCl should not exceed 200 mg. See Appendix M (Section 17.12) for guidance on RopiHCl dosing.

#### 10.1.3. Surgery Phase: Administration of Study Medication Into the Surgical Site

Study treatment is to be administered intraoperatively as a single administration via "surgical site" infiltration. The "surgical site" is defined as the area extending approximately 5 cm in all directions (lateral/medial/proximal/distal/deep) from the incision and osteotomy sites and surrounding tissues which may be affected by infiltration of the study treatment.

Note that T0 is the time that the study treatment injection/instillation is completed.

#### **Pilot Stage:**


Prior to hardware placement, 100 mL of study treatment should be infiltrated/instilled as follows:

1. Infiltrate 15 mL divided equally throughout the posterior capsule

With the leg in full extension, perform the following (working from top to bottom or using another standardized method per surgeon discretion):

- 2. Infiltrate 15 mL circumferentially around the distal femur
- 3. Infiltrate a total of 30 mL divided equally into the medial and lateral gutters ensuring coverage of the periosteal borders
- 4. Infiltrate 10 mL around the peripatellar region
- 5. Infiltrate 10 mL divided equally medial and lateral to the tibial tubercle

Following closure of the joint capsule,

6. Instill 20 mL "intra-articularly" (lateral approach) and move the joint through full range of motion

#### **Second Stage:**

Instructions for study treatment infiltration/instillation will be designated in the protocol amendment to follow the Pilot Stage.

#### 10.1.4. Inpatient Phase: Time 0 (Post-Surgery) to Day 4 (Discharge)

Following surgery, subjects will be transferred to the appropriate recovery unit where they will undergo an assessment of safety and efficacy over the next 96 hours. The schedule of assessments are as follows:

- Subjects with inadequately controlled pain may request rescue at any time; however, subjects will be encouraged to receive rescue medication only with an NRS ≥ 4.
- Pain intensity (assessed with NRS):
  - Ouring the inpatient stay, beginning with the PACU admission and after the subject is awake: assess the NRS at rest at 0.5, 1, 2, 4, 6, 8, 12, 16, 20, and 24 hours, and every 4 hours (if awake at time of assessment) until discharge from the inpatient unit. Time windows: for T0.5 to T2 (±5 min) and from T4 onward (±15 min).
  - O Pain scores may be skipped between the hours of midnight and 6 a.m., but the subject may not miss two consecutive assessments. The T12, T24, T48, T72 and T96h assessments must be completed even if the subject is asleep at these times.
  - o Pain intensity (NRS) will be completed at the time of rescue medication request ( $\pm 15$  minutes).
  - O During the inpatient stay, starting on postoperative day 1 (after T24): each morning on ambulation at 0800h (±2h) and each evening at 2000h (±2h) document the NRS after physical therapy or with partial or full weightbearing for transfers to/from bed or frank ambulation of approximately 10 yards. Actual assessment times must be documented. These assessments are in addition to the time-specific NRS assessments at rest. If


however, these twice daily assessments coincide with timed assessments of NRS at rest, then the time assessment at rest is used in place of the twice daily assessments.

- Vital signs (heart rate [HR], blood pressure [BP], respiratory rate [RR]) and temperature are assessed together post-surgery at T1, T2, T4, T6, T12, and T24h, and every 8 hours thereafter until T96h. Assessments between the hours of 00:00 and 06:00 may be skipped if the subject is sleeping; however, two consecutive assessments may not be skipped. The allowable window is ±5 minutes for the first 4 hours post-surgery, and ±15 minutes for all other times.
- Targeted Physical exam: 96 (±4) hours after the administration of study medication (prior to discharge from the unit).
- ECG: 24 ( $\pm$ 2) hours after the administration of study medication.
- Surgical site assessment: 96 (±4) hours after the administration of study medication. If the investigator determines there are atypical wound healing or visible abnormal findings, a digital picture of the wound site should be performed.
- Neurosensory testing of the surgical area: 96 (±4) hours after the administration of study medication.
- KOOS Survey: T96h (±4h) prior to discharge from the unit
- Clinical laboratory tests: T96h (±4h) prior to discharge from the unit.
- Blood draw for PK analysis: The time points for whole blood collection will be at check-in/baseline (up to 30 min prior to surgery), and T5min, T10 min, T15min, T30min, T45min, and T1, T1.5, T2, T2.5, T3, T4, T6, T8, T12, T16, T24, T30, T36 and T48h for a total of 20 samples).
- 24h urine collection in two aliquots: end of surgery to T6h and T6h to T24h.
- Subject completes Patient Global Evaluation (PGE) assessment and KOOS survey at T96h (±4) prior to discharge
- Investigator completes Investigator Global Evaluation (IGE) assessment at T96 (±4) prior to discharge. Note that the IGE may be performed by any investigator or sub-investigator.
- Record rescue medication consumption and concomitant medications throughout the inpatient period.
- Record AEs throughout the inpatient period (Section 17.11 Appendix K may be useful to the investigator for assessing systemic [general] AEs)

After completing the assessments through T96h, the diary for at-home use will be reviewed and subjects will be discharged from the study center with diary to record pain assessments and pain medication at home. Subjects will be provided routine standard of care for pain management after discharge from the study center. Subjects will be instructed to return to the study center on Day 8  $[\pm 1 \text{ day}]$  for follow-up assessments.


### 10.1.5. Outpatient Phase: Days 4 (after discharge) through 8:

In their diary, subjects will assess their pain intensity at rest and after ambulation (of approximately 10 yards) once in the morning (08:00  $\pm$ 4 hours), and once in the evening (20:00  $\pm$ 4 hours) using the NRS (two separate scores "at rest" and after "ambulation". Subjects will also record any medication they take to treat their pain.

Subjects will return to the study center on Day 8 [ $\pm 1$  day] for the following assessments:

- Subject home diary review (pain intensity and pain medication)
- Pain Intensity assessment (NRS)
- KOOS Survey on Day 8±1
- Vital signs including temperature
- Targeted PE
- Surgical Site assessment (If the investigator determines there are atypical wound healing or visible abnormal findings, a digital picture of the wound site should be performed if the subject has consented to such a photo)
- Neurosensory testing of the surgical area
- Query the subject as to any rebound pain
- Concomitant Medication Use/Concomitant Treatments
- AE Assessment
- PGE
- IGE

#### 10.1.6. Outpatient Phase: Days 9 through 15:

In their diary, subjects will assess their pain intensity at rest and after ambulation (of approximately 10 yards) once in the morning (08:00  $\pm$ 4 hours), and once in the evening (20:00  $\pm$ 4 hours) using the NRS (two separate scores "at rest" and after "ambulation". Subjects will also record any medication they take to treat their pain.

Subjects will return to the study center on Day 15 [±2 days] for the following assessments:

- Subject home diary review (pain intensity and pain medication)
- Pain Intensity assessment (NRS)
- KOOS Survey
- Vital signs including temperature
- Targeted PE
- Surgical Site assessment (If the investigator determines there are atypical wound healing or visible abnormal findings, a digital picture of the wound site should be performed if the subject has consented to such a photo)
- Neurosensory testing of the surgical area


- Query the subject as to any rebound pain
- Concomitant Medication Use/Concomitant Treatments
- AE Assessment
- PGE
- IGE

#### 10.1.7. Outpatient Phase: Day 29

Subjects will return to the study center on Day 29 [±2 days], or at the time of discontinuation, for the following assessments:

- Subject home diary review (pain intensity and pain medication)
- KOOS Survey
- Vital signs
- Targeted PE
- Surgical Site assessment (If the investigator determines there are atypical wound healing or visible abnormal findings, a digital picture of the wound site should be performed if the subject has consented to such a photo)
- Neurosensory testing of the surgical area
- Knee x-ray of the operated site
- Concomitant Medication Use/Concomitant Treatments
- Query the subject as to any rebound pain
- AE Assessment
- PGE
- IGE

### 10.1.8. Outpatient Phase: Early Termination

Subjects who elect to ET and are willing to perform study completion assessments will return to the study center at a convenient time after discontinuation, for the following assessments:

- Subject home diary review (pain intensity and pain medication)
- Pain Intensity assessment (NRS)
- KOOS Survey
- Vital signs including temperature
- Targeted PE
- Surgical Site assessment (If the investigator determines there are atypical wound healing or visible abnormal findings, a digital picture of the wound site should be performed if the subject has consented to such a photo)
- Neurosensory testing of the surgical area
- Knee x-ray of the operated site


- Concomitant Medication Use/Concomitant Treatments
- Query the subject as to any rebound pain
- AE Assessment
- PGE
- IGE

If the subject has elected an early termination and is unwilling to come in to have the assessments performed, at least try to have them return to their surgeon for a wound assessment and x-ray.

#### 10.1.9. Outpatient Phase: Unscheduled Visit

Note that unscheduled visits will be at the discretion of the Investigator but should include the following if performed prior to D15 visit:

- Subject home diary review (pain intensity and pain medication)
- Pain Intensity assessment (NRS)
- KOOS Survey
- Vital signs including temperature
- Surgical Site assessment (If the investigator determines there are atypical wound healing or visible abnormal findings, a digital picture of the wound site should be performed)
- Targeted Physical Exam
- Neurosensory testing of the surgical area
- Concomitant Medication Use/Concomitant Treatments
- Query the subject as to any rebound pain
- AE Assessment

If after D15 visit, subjects will return for the following assessments:

- Surgical Site assessment (If the investigator determines there are atypical wound healing or visible abnormal findings, a digital picture of the wound site should be performed)
- Neurosensory testing of the surgical area
- KOOS Survey
- Concomitant Medication Use/Concomitant Treatments
- Query the subject as to any rebound pain
- AE assessment

If after D29 visit, the investigator has clinical discretion on when subjects should return for follow up and what is performed at the visit. The following are the minimum assessments:

- Surgical Site assessment (If the investigator determines there are atypical wound healing or visible abnormal findings, a digital picture of the wound site should be performed)
- Neurosensory testing of the surgical area
- KOOS Survey


- Knee x-ray of the operated site to ensure proper healing. Follow subject until resolution or stabilization.
- Concomitant Medication Use/Concomitant Treatments
- Query the subject as to any rebound pain
- AE Assessment

# 10.2. Subject Completion and Withdrawal

### 10.2.1. Subject Completion

A subject is considered to have completed the study once all end-of-study assessments are completed at D29 (or later if necessary), or at the last visit upon early termination of the study.

### 10.2.2. Subject Withdrawal

A subject is free to withdraw his/her consent and discontinue participation in the study at any time for any reason. A subject's participation must therefore be terminated immediately upon his/her request, and the reason(s) for discontinuation appropriately documented.

A subject may be discontinued from the study for any of the following reasons:

- Safety reasons, including AEs or significant concomitant illness, injury, or urgent surgeries/procedures that would, in the judgment of the Investigator, affect assessments of clinical status to a significant extent, require discontinuation of study drug, or both
- At the request of the Sponsor, regulatory agency, or Institutional Review Board (IRB)
- Subject is lost to follow-up
- Subject treatment allocation is unblinded (i.e., individual code break; Section 9.4)
- Death of subject

A subject may also be discontinued from the study, at the discretion of the Investigator and/or Sponsor, for any of the following reasons:

- Subject refuses or is unable to adhere to the study protocol
- Major protocol violation
- Pregnancy
- Use of unacceptable concomitant medication(s)
- It is not considered in the best interest of the subject to continue
- Administrative reasons (e.g., termination of enrollment or study)

The Investigator must maintain a record of all subjects who discontinue from the study prior to completion; the reason(s) for study discontinuation will be documented. If a subject chooses to withdraw from the study, the Investigator should make a reasonable attempt to obtain and record


the reason(s) for withdrawal in as much detail as possible, although the subject is not obligated to provide such a reason.

Subjects who elect to discontinue participation prior to D8 (W1) will be considered to have terminated as of the date of their election, however they will be asked to return to the site or their surgeon, if willing and at their convenience, to ensure adequate wound healing. If a subject should refuse to complete early termination/Follow-up procedures or continued data collection, this information will be recorded.

# 10.3. Study Procedures and Assessments

#### 10.3.1. Informed Consent

The nature of the study and its risks and benefits will be explained to the subject by the Investigator or designated study personnel. The subject must voluntarily provide written informed consent on an ethics-approved informed consent form (ICF), prior to performing any study-related procedures. The subject's source records must document that the consent process has been completed and that written informed consent has been obtained from the subject prior to the initiation of any study-specific procedures. Documentation that the subject was given adequate time to ask the Investigator (or designee) questions about their participation in the study and that a signed and dated copy of the ICF was provided to the subject should also be included in the medical records or clinical chart.

## 10.3.2. Demographics

The following demographics will be recorded: age (birthdate), sex, race, and ethnicity.

#### 10.3.3. Medical and Surgical History

The complete medical and surgical history will include histories of acute, chronic, or infectious disease; surgical or oncologic histories; and any reported conditions affecting major body systems. All findings on medical history will be evaluated by the Investigator for clinical significance.

#### **10.3.4. Medication History**

All medications (prescription and non-prescription, herbal medications/natural health products, or investigational drugs) taken by the subjects during the 45 days prior to Screening will be recorded in the source documentation as medication history.

#### 10.3.5. Contraceptive Requirements

Female subjects of childbearing potential must be using and willing to continue using medically acceptable contraception during the study unless they have a same sex partner. Examples of medically acceptable forms of contraception include true abstinence, hormonal contraceptives (combined oral pill, patch or vaginal ring, intrauterine device or system, progestin implant or


injection), bilateral tubal ligation, or double-barrier methods (i.e., male condom in addition to a diaphragm or a contraceptive sponge).

Female subjects of non-childbearing potential are not required to use contraception or undergo pregnancy tests; however, they must be surgically sterile (e.g., hysterectomy and/or bilateral oophorectomy or salpingo-oophorectomy, as determined by subject medical history) or congenitally sterile or must be post-menopausal. Post-menopausal is defined as being amenorrheic for at least one year without another cause.

Male subjects, unless in a relationship with a same sex partner or a female partner who is of non-childbearing potential (see above), must either be sterile (surgically **or** biologically) or commit to using double-barrier methods (i.e., male condom in addition to a diaphragm or a contraceptive sponge) during the study.

## 10.3.6. Subject Pain Assessment Training

Subjects will undergo study participation education on pain assessments and written testing procedures according to the Schedule of Study Procedures.

### 10.3.7. Digital Photographs of the Surgical Site

During the informed consent process, subjects will be asked if they are willing to allow digital photographs to be taken of the surgical site. This is optional, and their response will in no way affect their inclusion in the study. Their response will be included on the ICF.

#### 10.3.8. Numerical Rating Scale for Pain Intensity (NRS)

The NRS is an 11-point scale with anchors 0 (no pain) and 10 (worst possible pain) (Section 17.2 Appendix B).

Subjects will report or record the intensity of their current pain at designated times during the study after administration of study treatment. Subjects should be at rest for at least 5-10 minutes prior to completing NRS resting assessment and have sat or stood up from a recumbent position within the 5-10 minutes prior to completing NRS assessment after this change in position.

#### 10.3.9. Rebound Pain at the Surgical Site

Subjects will be queried at each outpatient follow up visit as to whether they have noted any worsening pain (rebound pain) at the surgical site since the prior visit report (Section 17.3 Appendix C).

#### 10.3.10. Knee Injury and Osteoarthritis Outcome Score (KOOS)

Subjects will complete the KOOS survey at designated times during the study after administration of study treatment (Section 17.13 Appendix M). The KOOS survey was developed in the 1990s as an instrument to assess the patient's opinion about their knee and


associated problems (see <a href="http://www.koos.nu/">http://www.koos.nu/</a>). Note that for purposes of this study, responses in the KOOS will not be considered or captured as spontaneous AEs.

### 10.3.11. Patient Global Evaluation (PGE)

Each subject will be asked to report their satisfaction with the study treatment for pain using a 4-point categorical scale. Each subject will be asked the following question:

"How would you rate the study treatment that you have received for pain? Poor (0), Fair (1), Good (2), or Excellent (3)" (see Section 17.4 Appendix D).

### 10.3.12. Investigator Global Evaluation (IGE)

The investigator will report their satisfaction with the subject's study treatment for pain using a 4-point scale at designated times during the study after administration of study treatment. A study investigator will be asked the following question:

"How would you rate the study treatment that the patient received for pain? Poor (0), Fair (1), Good (2), or Excellent (3)" (see Section 17.5 Appendix EAppendix E).

#### 10.3.13. Rescue Medications

The details of rescue medication (doses and times) will be recorded beginning from the end of surgery through 14 days after the end of surgery (D15 visit) or to Early Termination Visit if applicable. Subjects will be instructed on the proper use and timing of rescue medication.

Use Table 9 to calculate the oral morphine equivalent dose (MED) of various opioids.

**Table 9. Equianalgesic Conversion Table** 

| Conversion Factor to IV morphine | Conversion Factor to PO morphine |
|----------------------------------|----------------------------------|
| 100 | |
| 6 | |
| 1 | 6* |
| | 1 |
| | 1 |
| | 1.5 |
| | 0.1 |
| | IV morphine |

For any IV opioid, we will use a 2-step process to calculate its oral (PO) morphine equivalent dose (MED).


- 1. Convert its IV dose to IV morphine MED by multiplying by the conversion factor for IV equivalence.
- 2. Once the IV morphine MED is calculated, convert to the PO morphine MED using the conversion factor for PO equivalence.

For any PO opioid, use the conversion factor to calculate the PO MED.

\*Note that for non-tolerant patients, we are using the 6:1 conversion for IV to PO morphine.

#### 10.3.14. Clinical Laboratory Assessments

All protocol-specified laboratory tests on blood and urine samples will be collected, processed, shipped and analyzed according to instructions from a selected central laboratory. The lab will generate laboratory reports and forward them to the clinical site in a timely manner. It is the responsibility of the Investigator to review and sign all lab reports expeditiously, to document appropriate safety monitoring of study subjects. The Investigator should sign and date each lab report concurrent with her or his review and should indicate the clinical significance of each abnormal/flagged value by noting "NCS" (not clinically significant) or "CS" (clinically significant), for example. Notations indicating that a value is clinically significant should also include a brief description of the underlying disease or condition that is associated with the value, e.g., "CS/mild anemia." In general, and as determined by the investigator, abnormal, clinically significant laboratory values are expected to be associated with an item recorded in medical history or with an AE.

Additional laboratory samples may be taken at the discretion of the Investigator if the results of any tests fall outside reference ranges or clinical symptoms necessitate testing to ensure safety. Specific hematology, coagulation, biochemistry, and urinallysis assessments are listed in Table 10.

**Table 10. Clinical Laboratory Assessments** 

| Hematology | Chemistry | Urinalysis |
|---|---|---|
| Hematocrit | Sodium | Color |
| Hemoglobin | Potassium | Turbidity |
| Red blood cell (RBC) count | Calcium | рН |
| Total and differential (absolute) | Chloride | Specific gravity |
| white blood cell count | Glucose | Ketones |
| Platelet count | Creatinine | Protein |
| Coagulation | BUN | Glucose |
| | Albumin | Bilirubin |
| Activated partial | Tot Bili | Occult blood / Nitrite |
| thromboplastin time (aPTT) | ALT | Urobilinogen |
| Prothrombin time (PT) / International normalized ratio | AST | Leukocyte esterase |
| (INR) | GGT | Microscopic examination of |
| | Alkaline phosphatase | sediment, only if urinalysis dipstick results are abnormal |

The clinical laboratory tests will be completed per the Schedule of Assessments. In addition to the clinical laboratory tests, a serum pregnancy test will be performed at the Screening Visit and a urine pregnancy test will be performed prior to surgery for women of childbearing potential. ALT or AST > 3x ULN / Tot. Bili > 2 X ULN / Alk Phos. >2X ULN will be considered an adverse event, as well as any other changes deemed clinically significant by the Investigator.

#### 10.3.15. Urine Drug Screen and Alcohol Test

Urine drug screen and alcohol breath/saliva tests will be completed at screening and preprocedure. All subjects will be tested for drugs-of-abuse (e.g., amphetamines, barbiturates, benzodiazepines, cocaine, opiates, phencyclidine, tetrahydrocannabinol, methadone, methamphetamine, tricyclic anti-depressants, oxycodone and others).

The drug and alcohol screens will be performed in-house at the Clinical Unit. If any of these tests are positive, the subject will not be allowed further participation in the trial. However, a positive test may be repeated at the discretion of the investigator.

### **10.3.16.** Vital Signs

Vital signs will consist of BP, HR, and RR and temperature following a rest period. Vital signs will be assessed per the Schedule Assessments.


#### 10.3.17. 12-Lead Electrocardiogram (ECG)

12-Lead ECGs will be performed per the Schedule of Assessments after the subject has been resting in a recumbent/supine position for at least 5 minutes. The ECG variables will include ventricular heart rate and the PR, QRS, QT and QTcF intervals. ECGs will be signed and dated by a medically-qualified individual to confirm review of the ECG and verify whether any abnormalities are clinically significant. In general, abnormal, clinically significant ECGs are expected to be associated with an item recorded in medical history (e.g., at Screening) or with an AE (if it occurred post study treatment). Note that for QTc, clinically significant changes in ECG (using QTCf, should be <450 msec for male subjects / < 470 msec for female subjects. Clinically significant changes in ECG are: an increase of QTcF of 30msec or greater, as well as any other changes deemed by the Investigator as significant will be considered an AE.

#### 10.3.18. Physical Examination

A complete PE including all major body systems (HEENT, neurologic, cardiovascular, respiratory, gastrointestinal, dermatologic and musculoskeletal systems) will be performed at Screening. A focused interim or targeted PE will be performed pre-surgery and after surgery during the inpatient and outpatient periods (see Table 1).

Body weight (kg), in indoor clothing, but without shoes, will be measured at Screening and 96 hours. Height in centimeters (cm) will be measured, and BMI will be calculated at Screening only. BMI shall be calculated as kg/m<sup>2</sup>. The site should use NIH website BMI calculator (available at: http://www.nhlbi.nih.gov/health/educational/lose\_wt/BMI/bmi-m.htm).

#### 10.3.19. Surgical Site Assessment

The surgical site should be assessed per the Schedule of Assessments to determine if any site related AEs have occurred. The investigator will evaluate their satisfaction with the healing of the wound during this Surgical Site assessment using an 11-point scale (0-10) where a score of 0 is "Completely unsatisfied," and a score of 10 is "Completely satisfied." (Section 17.6 Appendix F). Assessments will also be performed at each of the Follow-up visits or at the time of early discontinuation. When assessed on Day 29, if the Investigator observes insufficient wound or bone healing or to ensure an ongoing AE has resolved, the subject will be scheduled for a follow-up visit.

If there are skin reactions atypical for the type of surgery, e.g., more than expected erythema, drainage, bruising or hematoma, induration, swelling or other skin changes, they should be documented as AEs, graded for severity and followed regularly until resolution or establishment of a new baseline (the grading guide for atypical wound findings may be useful to the investigator: Section 17.7 Appendix G).


#### 10.3.20. Neurosensory Testing

Neurosensory testing of the skin surrounding the incision will be conducted per the Schedule of Events. This evaluation will include the details described in Section 17.8 Appendix H. Numbness or other sensory changes at or near the incision need not be considered a neurologic AE since these could occur because of tissue trauma and inflammation from surgery.

Sensory deficits or clinically significant persistent sensory change beyond the area proximal to the incision at time of discharge, such as allodynia or hyperalgesia, must be designated as a neurologic AE. Subjects will be followed until there is full return to baseline for the neurosensory assessment or until there is a determination that it has reached a resolution or establishment of a new baseline

#### 10.3.21. Assessment of Adverse Events

All AEs and SAEs will be documented and followed from the time the subject has signed the ICF until Day 29 or later as necessary. All SAEs and non-serious AEs will be documented and followed from the time of administration of study treatment until Day 29 or until resolution or establishment of a new baseline. AEs that occur between Screening and the surgery should be considered medical history, and be added to the subject's medical record, unless related to a study procedure. Serious AEs and AEs that have been designated as possibly related to study drug will be followed until resolution or stabilization. Further details on AEs, including definitions, elicitation, and reporting are provided in Section 11.

#### 10.3.22. Pharmacokinetic Assessments and Samples

Details for the collection and processing of blood samples for measurement of PK (CA-008, Capsaicin, and CA-101) and urine collections are outlined in the Lab Manual.

## 10.4. Safety, PK and Efficacy Endpoints

#### 10.4.1. Safety Endpoints

Safety endpoints include the following:

- Incidence of spontaneously reported TEAEs or SAEs
- Clinical laboratory test results
- Vital sign measurements
- ECG results
- PE findings
- Surgical Site wound assessment findings
- Neurosensory testing results


- Knee x-ray
- Presence of rebound pain
- Concomitant Medication Use/Concomitant Treatments

#### 10.4.2. Pharmacokinetic Endpoints

Full details of pharmacokinetic endpoints will be described in a separate PK Analysis Plan. The time points for whole blood collection are outlined in the Schedule of Assessments. Actual sampling times will be used to calculate plasma-derived PK parameters.

#### 10.4.3. Pilot Stage Efficacy Endpoints

#### 10.4.3.1. Primary Efficacy Endpoint

Time-specific mean pain intensity scores at T96h for CA-008 vs. placebo.

Note that pooled placebo for cohorts #2 and #3 will be used for the primary and key secondary efficacy assessments during the exploratory pilot stage.

#### 10.4.3.2. Key Secondary Efficacy Endpoints

For the CA-008 vs. placebo comparison:

- Weighted sum of pain intensity (SPI) assessments = Area Under the Curve (AUC) of the NRS current pain intensity scores from T0 to 96h at rest (AUC<sub>0 to 96h</sub>).
- Percentage of subjects who do not require opioids (i.e., opioid free; OF) from T0 to T96:
   OF<sub>0 to 96h</sub>
- Total opioid consumption (in daily oral morphine equivalents) = OC from T0 to T96h: OC<sub>0</sub> to 96h

#### 10.4.4. Stage 2 Efficacy Endpoints

All analyses will compare each CA-008 dose group vs. the placebo group.

#### 10.4.4.1. Primary Efficacy Endpoint

Weighted sum of pain intensity (SPI) assessments = Area Under the Curve (AUC) of the NRS current pain intensity scores from T0 to 96h at rest (AUC<sub>0 to 96h</sub>).

#### 10.4.4.2. Key Secondary Efficacy Endpoints

- Percentage of subjects who do not require opioids (i.e., opioid free; OF) from T0 to T96:
   OF<sub>0 to 96h</sub>
- Total opioid consumption (in daily oral morphine equivalents) = OC from T0 to T96h: OC<sub>0 to 96h</sub>
- Using NRS at rest: AUC<sub>0 to W1</sub>


#### 10.4.4.3. Other Endpoints

- Using NRS at rest: AUC 0 to 24h, AUC 0 to 120h, AUC 6 to 96h, AUC24 to 96h, AUC96h to W1, AUC96h to W2
- $\bullet \quad AUC \ 0 \ to \ 96h \ (ambulation), \ AUC \ 0 \ to \ W1 \ (ambulation), \ AUC \ 24h \ to \ W1 (ambulation), \ AUC \ 96h \ to \ W2 \ (ambulation)$
- Time-specific mean NRS scores at T48, T72, T96, T120, T144 and T168h
- OC<sub>24 to 48h</sub>, OC<sub>24 to 72h</sub>, OC<sub>24 to 96h</sub>
- OF<sub>24 to 96h</sub>, OF<sub>96h to W1</sub> and OF<sub>96h to W2</sub>
- KOOS improvement from T96h to D8/W1, D15/W2 and D29/W4
- TTFR<sub>after T0</sub> and TTFR<sub>after T24h</sub>
- The fraction of subjects who rescue at T6, T12, T24, T48, T72 and T96h
- Analgesic consumption from T96h to W1 (AC<sub>96h to W1</sub>) and AC<sub>96h to W2</sub>
- PGE comparing the %age of subjects reporting "poor" + "fair" vs. "good" + "excellent" responses, and the %age reporting each category of response at T96h, D8/W1, D15/W2 and D29/W4
- IGE comparing the %age of those reporting "poor" + "fair" vs. "good" + "excellent" responses, and the %age reporting each category at T96h, D8/W1, D15/W2 and D29/W4
- Number and %age subjects with an AE of lack of efficacy (LOE) during the inpatient period: LOE<sub>0 to 96h</sub>
- HCU<sub>96h to W2</sub> and HCU<sub>96h to W4</sub>


#### 11. ADVERSE EVENTS

#### 11.1. Adverse Events and Serious Adverse Events

The following definitions, developed in accordance with the United States (US) Code of Federal Regulations (CFR) and the International Conference on Harmonization (ICH) Clinical Safety Data Management Guidance for Industry, E2A, will be used to identify AEs in this study.

An AE is any untoward medical occurrence in a subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., including an abnormal laboratory finding), symptom, or increase in severity of a preexisting abnormality, temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product.

Since this is a study using a surgical pain model, findings that are "typical" for the surgery should not be captured as an AE. Atypical or worse than typical findings should be captured as AEs.

A "suspected adverse reaction" means any AE for which there is a reasonable possibility that the drug caused the event. "Reasonable possibility" means there is evidence to suggest a causal relationship between the drug and the adverse event.

#### 11.1.1. Relationship to Study Treatment

A qualified investigator must make the determination of relationship to the investigational product for each AE. The Investigator should decide whether, in his or her medical judgment, there is a reasonable possibility that the event may have been caused by the study treatment.

| Causality<br>Category | Description |
|---|---|
| Unlikely related | A clinical event, including laboratory test abnormality, with a temporal relationship to study treatment administration which makes a causal relationship improbable or if other drugs, chemicals or underlying disease provide more plausible explanations. While temporal sequence may be an important factor in determining causality: i.e., whether the observed reaction or event began after the study treatment, it may well be that the surgery, anesthesia, a concurrent medical condition or concomitant medications administered during or after surgery were more likely than not to be responsible for the AE. The investigator should use clinical judgment to evaluate the evidence and determine whether there is a reasonable possibility that study |


| | treatment actually caused the AE or whether based upon the evidence it |
|---|---|
| | is more likely that something else is responsible. If the former, choose |
| | "possibly related" and if the latter, "unlikely related." |
| | For the purpose of this protocol, the term "unlikely related" will be |
| | considered an AE not related to study treatment. |
| | A clinical event, including laboratory test abnormality, with a temporal |
| | relationship to study treatment administration, which also may be |
| | explained by concurrent disease or other drugs or chemicals. In such |
| | cases, if the investigator using clinical judgment is unable to rule out a |
| Possibly related | reasonable possibility that study treatment was partly responsible, then |
| | choose "possibly related." |
| | For the purpose of this protocol, an event that has possible relationship |
| | to study treatment will be defined as a "Suspected Adverse Drug |
| | Reaction". |
| | A clinical event, including laboratory test abnormality, with a temporal |
| | relationship to study treatment administration, in which the investigator |
| Drobobly related | has determined that the event is unlikely to be attributed to other |
| Probably related | factors. |
| | For the purpose of this protocol, an event that has probable relationship |
| | to study treatment will be defined as an "Adverse Drug Reaction". |

#### 11.1.2. Adverse Event Reporting

All AEs must be entered on the AE CRF, regardless of causality or severity. AEs include new AEs, worsening baseline conditions, clinically significant laboratory findings, disease-related signs and symptoms that were not present at baseline, and any events or findings that the Investigator feels are clinically significant.

Disease-related signs and symptoms that are present at baseline should not be recorded as AEs unless they worsen in severity or increase in frequency.

Information collected concerning AEs will include the following:

- Name of the event
- Onset date
- Resolution date
- Severity (i.e., mild, moderate, severe or potentially life-threatening)
- Relationship to study treatment
- Action and outcome
- Seriousness of event


All SAEs will be documented and followed from the time the subject has signed the ICF until D29±2 after the completion of surgery. All SAEs and non-serious AEs will be documented and followed from the time of administration of study treatment until Day 29 or later if necessary. AEs that occur between Screening and the administration of study medication should be considered medical history and added to the subject's medical record, unless the AE is due to a study-related procedure (such as phlebotomy), in which case it will be recorded as a non-treatment emergent AE. Serious AEs and AEs that have been designated as possibly related to study treatment will be followed until resolution or stabilization.

#### 11.1.3. Serious Adverse Event (SAE)

An SAE or reaction is any adverse drug experience occurring at any dose that results in any of the following outcomes:

- Death
- Is life-threatening (at the time of the event)
- Requires subject hospitalization or prolongation of existing hospitalization,
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly/birth defect (in an offspring)
- An Important medical event that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, the event may jeopardize the subject and/or may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

All AEs requiring hospitalization or prolongation of a pre-existing hospitalization should be reported as SAEs unless they occur  $\geq$  14 days after the Day 29 visit, or 21 days after an early termination AND are not considered to be study treatment-related by the Investigator.

Hospitalizations meeting the following criteria will not be reported as an SAE but must be recorded on the appropriate CRF: study specified hospitalization, short-term administrative hospitalization for procedures, tests or treatments of conditions that would not otherwise constitute an SAE, elective hospitalizations.

#### 11.1.3.1. Serious Adverse Event Reporting

Serious AEs must be reported to the Sponsor or designee within 24 hours of knowledge of the event. All SAEs that occur while a subject is receiving study treatment and within 14 days following the study completion visit (or 21 days following an ET if applicable) are reportable within 24 hours. During this follow-up period beyond study completion or after an ET, only those SAEs considered to be possibly related to study treatment should be reported within 24 hours.


The procedure for reporting an SAE is as follows:

- All SAEs must be reported immediately (within 24 hours of discovery) by email to the CRO Medical Monitor or designee. Calls related to SAEs should first be directed to the CRO Medical Monitor or designee.
  - o CRO Medical Monitor: Jon Ruckle, MD
  - o 24/7 Emergency contact: 808-349-9812 / (253) 448-8690
  - o SAE Reporting email: MedicalMonitorCA-PS-203@Lotuscr.com
- The Sponsor's Medical Monitor is available for questions about safety-related issues or to request waivers to modify postoperative patient care: Mike A. Royal, MD JD MBA; 858-204-1112 or mike@concentricanalgesics.com.
- The initial report should include all information known at the time of the report (additional information can be reported as discovered). Do not delay the initial reporting to obtain resolution or follow-up information.
- The site will enter into the electronic database (or fax, if the database cannot be accessed for any reason) an SAE report, or similar form, that includes the following information, as available:
  - Subject ID
  - o Basic demographic information (age, gender, weight)
  - Outcomes attributed to the event (death, life-threatening hospitalization [new or prolonged], disability, congenital anomaly, required medical intervention to prevent permanent impairment/damage, etc.)
  - Onset date and severity of the event
  - Brief description of the event including frequency and severity of symptoms leading to diagnosis
  - List of relevant test results and laboratory data
  - Any other relevant history
  - Whether the study treatment was discontinued
  - o Investigator's assessment of causality

The CRO Medical Monitor or another representative of the Sponsor may contact the Investigator to request additional information regarding the event or to confirm information. All SAEs will be entered on the AE CRF. The same nomenclature should be used on both the SAE report and the AE CRF. The Investigator is responsible for the complete and timely reporting of all SAEs to the Sponsor (or designee), reporting pertinent follow-up information on the SAE, and notifying the appropriate IRB of the occurrence of and details surrounding the event. In the event there is a question as to whether the AE is serious, the event should be reported.


## 11.2. Severity Grading for AEs

Grading the severity of AEs is per investigator discretion (the guidance reflected in Sections 17.9, 17.10 and 17.11; Appendices I, J and K may be helpful). Additionally, the following general guideline may be helpful:

- Grade 1 (mild) = asymptomatic or mild symptoms requiring no treatment, only clinical or diagnostic observation
- Grade 2 (moderate) = event or symptoms limit age-appropriate activities of daily living (ADLs) more than is expected from the surgery itself, requiring minimal treatment or local noninvasive intervention indicated.
- Grade 3 (severe) = medically-significant but not immediately life-threatening, significantly limiting of self-care ADLs, requiring of medical treatment and may require hospitalization or prolongation of hospitalization.

## 11.3. Pregnancy

If a female subject becomes pregnant at any time during the study, the Investigator must notify the CRO Medical Monitor or designee within 48 hours of learning about the pregnancy. The Investigator will be required to follow the subject through the pregnancy term, and report to the CRO Medical Monitor or designee the course of the pregnancy, including perinatal or neonatal outcome. Information on the status of the mother and the child will be forwarded to the CRO Medical Monitor or designee. Any premature termination of the pregnancy will also be reported on this form. Although pregnancy occurring in a clinical study is not considered to be an SAE, any pregnancy complication or elective termination of a pregnancy for medical reasons will be recorded as an AE and will be followed as such. A spontaneous abortion is considered to be an SAE.


## 12. DATA QUALITY ASSURANCE

This study will be conducted under Good Clinical Practice (GCP) and all applicable regulatory requirements. To ensure compliance, the Sponsor or designee may conduct a quality assurance audit, as outlined in Section 12.2.

Actions to ensure the accuracy and reliability of data include the selection of qualified investigators and appropriate study centers; the review of protocol procedures with the Investigator and study personnel prior to study start; the design of suitable source documents with appropriate instructions for use (where applicable); the internal audit of source data according to GCP and internal procedures to ensure their accuracy, completeness, and verifiability; as well as the periodic site monitoring by the Sponsor. The Sponsor or designee will review source documents for accuracy and completeness during on-site monitoring visits and after their return to the Sponsor; any discrepancies will be resolved with the Investigator, as appropriate.

Significant and/or repeated non-compliance will be investigated, and remedial action instituted when appropriate. Failure to comply with remedial actions may result in investigational site termination and regulatory authority notification.

#### 12.1. Data Collection

Source documents include, but are not limited to, original documents, data and records such as hospital/medical records (including electronic health records), clinic charts, lab results, participant diaries, data recorded in automated instruments, microfilm or magnetic media, and pharmacy records, etc. This study will use electronic data capture (EDC). At a minimum, all data required by the protocol should have supporting source documentation for entries in the EDC system.

All CRFs will be completed by the site staff prior to review by the Sponsor's monitor or designated representative. The Sponsor's monitor or designated representative will review all source records on-site and compare them to the data collected on the CRF. All entries, corrections, and alterations will be made by the Investigator or other authorized study personnel. All data entries will be verified for accuracy and correctness by independent monitors. The electronic data capture system maintains a full audit trail.

## 12.2. Study Auditing and Monitoring

Monitoring of the study site (including, but not limited to, reviewing CRFs for accuracy and completeness) will be performed by the Sponsor's designated monitor(s). The extent, nature, and frequency of on-site visits will be based on such considerations as the study objectives and/or


endpoints, the purpose of the study, study design complexity, and enrollment rate. By signing the protocol, the Investigator agrees that, within local regulatory restrictions and institutional and ethical considerations, authorized representatives of the Sponsor, a regulatory authority, and/or an IRB may visit the site to perform audits or inspections, including the drug storage area, study drug stocks, drug accountability records, participant charts and source documents, and other records related to study conduct. The purpose of the Sponsor audit or inspection is to systematically and independently examine all study-related activities and documents to determine whether the study-related activities were conducted, and data recorded, analyzed, and accurately reported according to the protocol, the site's standard operating procedures, GCP guidelines of the ICH, and any applicable regulatory requirements. The Investigator should contact the Sponsor immediately if contacted by a regulatory agency regarding an inspection.


## 13. STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

## 13.1. Statistical and Analytical Plans

The sections of the Statistical Considerations describe the statistical methods to be used to analyze the efficacy and safety. These methods may be revised and updated due to reasons such as regulatory requirements or need for further clarifications. The final analysis will be documented in a formal Statistical Analysis Plan (SAP) that must be finalized before database lock. The SAP will include details on how variables will be derived, how missing data will be handled, and how data will be presented as well as the details on statistical methods to be used for safety and efficacy analyses. The final clinical study report will discuss deviations from the SAP, if any.

## 13.2. Sample Size Justification

Given the uncertainty in estimating a sample size for TKA surgery, the results from the Phase 2 bunionectomy study and the Pilot Stage (cohorts #1 through #3) topline data from the current study will be used to determine active treatment doses and sample size for Stage 2 of this study. To this end, an interim unblinded analysis will be performed after the last subject has completed the D8/W1 visit (details may be found in the SAP). Topline results will be generated and used for the subsequent protocol amendment plan wherein several CA-008 dose groups are planned compared to placebo in a prospective, randomized, parallel design for Stage 2 of the study.

## 13.3. Analysis Populations

The following analysis populations are planned for this study:

- The Safety Population will include all subjects who received any part of a dose of study treatment
- The PK Population will include all subjects who receive a full dose of study treatment and complete all PK assessments.
- The intent-to-treat (ITT) population will include all subjects as randomized to study treatment.

Membership in analysis populations will be determined before unblinding.

Subjects who elect to discontinue study participation (early termination or ET) after randomization but prior to receiving study treatment will be replaced.

Subjects who elect to ET after receiving study treatment will not be replaced, however those who ET during the inpatient phase of the study, will be asked to continue with assessments through


T96h if they have not elected to withdraw from all aspects of study participation.

## 13.4. Planned Analyses

Unless otherwise indicated, all testing of statistical significance will be 2-sided, and a difference resulting in a P value of less than or equal to 0.05 will be considered statistically significant. Furthermore, the baseline will be the last assessment before the dosing of study medication.

All inferential assessments will be 2-sided tests performed at the 0.05 alpha level unadjusted for multiple comparisons. A hierarchical alpha testing strategy will be utilized to control for the overall experiment-wise alpha. First the primary analysis will be performed at the 0.05 alpha level. If the primary analysis is statistically significant, then a limited number of key secondary analyses will be analyzed in a pre-specified order and analyses will be considered as statistically significant only if the preceding test is statistically significant. The order of the secondary analyses will be specified in the SAP and signed off prior to unblinding.

Summary statistics will be provided for the variables described in the following sections. For continuous variables, these statistics will typically include the number of subjects, mean, standard deviation (SD), median, minimum, and maximum. For categorical variables, these statistics will typically include the number and percentage of subjects in each category.

## 13.5. Study Subjects and Demographics

#### 13.5.1. Disposition and Withdrawals

The numbers of subjects randomized, completing, and withdrawing, along with reasons for withdrawal, will be tabulated overall and by treatment group. The number of subjects in each analysis population will be reported.

#### 13.5.2. Protocol Deviations

Major protocol deviations will be classified and documented before database lock and will be discussed in the CSR. All protocol deviations, both minor and major, will be presented in a data listing.

## 13.5.3. Demographics and Other Baseline Characteristics

Demographic and baseline characteristics (including age, sex, race, weight, and height) will be summarized for each treatment group and for the overall population by descriptive statistics. Medical history and clinical laboratory tests will be listed.

Prior and concomitant medications will be summarized by treatment group, by the number and percentage of subjects taking each medication, classified using World Health Organization Drug Dictionary Anatomical Therapeutic Chemical classes and preferred terms.


#### **13.5.4.** Exposure

Since this is a single dose study, study drug administration will be summarized in terms of total exposure by cohort and treatment group.

#### 13.5.5. General Considerations

All continuous study assessments will be summarized by treatment and time point (as applicable) using the descriptive statistics n, mean, SD, median, and range (minimum, and maximum). Categorical assessments will be summarized by treatment and time point (as applicable) using frequency counts and rates of occurrence (%). Changes from baseline for continuous outcomes will be presented as their corresponding continuous measures for post-baseline visits. All study data will be listed by treatment group, subject and time point.

No preliminary rounding will be performed; rounding will only occur after the analysis. Means and medians will be presented with one more decimal place than the precision of the data. Standard deviations will be presented with two more decimal places than the precision of the data. Percentages will be presented with one decimal place. A percentage of 0% or 100% will be reported as 0% or 100%, respectively. Minimums and maximums will be presented with the same precision as the original data.

All analyses will be performed using the SAS System® version 9.3 or higher. The domain (Study data tabulation Model [SDTM]) and analysis (Analysis Data Model [ADaM]) data sets will be taken as input to the SAS programs that generate the report-ready tables, figures and listings. The submission ready SDTM and ADaM data sets will be provided to the sponsor along with display deliveries. The specifications for the domain data sets and analysis data sets will be provided in a separate document.

The following conventions will be used throughout the study analysis:

- Time T0 is the time of completion of study treatment administration.
- Day of surgery is defined as D0
- Assessment visit times are defined by time T0/D0.
- Baseline value is defined as the last valid measurement prior to beginning study treatment administration.
- Change from baseline is defined as post-baseline value minus baseline value.
- Duration of an AE will be computed in days for AEs lasting longer than 24 hours, and as hours for AEs lasting less than 24 hours. Duration in hours will be calculated as the stop date/time of the event minus the start date/time. Duration in days will be calculated by using stop date minus the start date +1 if AE occur on or after taking study medication. If AE occur prior to the study medication, then the duration will be calculated by using stop date minus the start date. If reported as ongoing at the time of database lock, the duration will be calculated using the date of the last visit or the last date of any AE for the subject in the


database, whichever is later. Missing dates will be imputed as described in the Study's Statistical Analysis Plan (SAP).

- The number of days in the study is computed as: [Date of study completion or withdrawal minus the date of study drug administration (Day 1)] + 1.
- If duplicate values are obtained at a given visit (e.g., repeated vital sign measurements), the last value will be used unless it is noted that the measurement was in error for that value. Values that compromise interpretation will not be used in summaries (e.g., values that were obtained post-dose will not be summarized as pre-dose values).

#### 13.5.6. Analysis of Efficacy Measures

All efficacy endpoints (e.g., NRS scores), will be summarized over time by treatment using descriptive statistics including confidence intervals as appropriate.

AUC calculations will be done using the standard trapezoidal rule

AUC = 
$$\sum_{i=0}^{x} \left( \frac{NRS_i + NRS_{i+1}}{2} \right) * (T_{i+1} - T_i)$$

Where:  $NRS_i = NRS$  at time i, and  $(T_{i+1} - T_i)$  is the Time difference in minutes between time i and time i+1. A similar calculation and handling of missing data will be performed for the NRS scores with position changes.

Missing NRS will be handled as discussed in the Study's SAP.

The AUC analyses will be presented in a summary table with standard summary statistics for each dose cohort and placebo as well as active vs. placebo mean differences, standard errors, confidence intervals and comparison p-values as appropriate. Comparisons of individual dose cohorts for dose response may also be presented for certain secondary AUC endpoints.

The AUC analyses will be presented in a summary table with standard summary statistics for each treatment group mean differences standard errors, confidence intervals and comparison p-values as appropriate.

Mean NRS scores over time (in-clinic and diary) will be graphed over time by treatment group. NRS over time by each subject may also be displayed graphically as warranted. The individual NRS and the computed AUC variables will be listed for all individual subjects.

In this study, subjects are permitted to take rescue medication for analgesia. It is expected subjects randomized to placebo arm will take rescue medication more often. During both inpatient and outpatient portions of the studies, the subjects will be instructed to record NRS immediately prior to taking rescue medication.

For subjects who take rescue, the pre-rescue pain score will be used to impute scheduled assessments for 4 hours. Intermittent missing pain scores (due to subject sleeping, etc.) will not


be imputed, and AUC will be calculated based on non-missing values. For subjects who drop out of the study prior to Day 15 due to Lack of Efficacy or Adverse Events, scheduled assessments may be imputed using worst prior pain score carried forward. All other subjects who drop out will have their last pain score carried forward.

Sensitivity analysis of the primary efficacy variable using different methods of imputation for rescue medication may also be performed.

Additional sensitivity analysis with different missing value imputation methods for subjects who drop out of the study may also be performed.

All imputation methods for pain intensity will be documented in the SAP.

#### 13.5.7. Handling of Dropouts or Missing Data

All efforts will be made to minimize missing data. These efforts will include the following:

- Subjects are required to consent continuous data collection even after subjects discontinue the study medication;
- Continue data collection after subjects taking rescue medication;
- Establish robust efficacy data collection procedures.

With the procedures above, it is expected that the missing would be minimal. Missing at random is expected to be a reasonable assumption and the primary analyses are expected to be sufficient for this dose escalation study. Additional sensitivity analyses will be performed to support robust conclusions, if warranted and details are presented in a detailed SAP prior to database lock.

For subjects who take rescue medication a windowed last pain score carried forward (wLOCF) will be used. The pre-rescue pain score will be used to impute scheduled assessments for 30 minutes following the rescue use when IV fentanyl is used, 2 hours when IV hydromorphone is used, and 4 hours when PO oxycodone is used. Intermittent missing pain scores (due to subject sleeping, etc.) will not be imputed, and AUC will be calculated based on non-missing values. For subjects who drop out of the study prior to Day 15, scheduled assessments will first be imputed using the worst prior pain score carried forward (WOCF). As sensitivity analyses, the AUC will also be calculated where assessments after drop out will be imputed using LOCF, using the last scheduled non missing pain score prior to drop out, and the median scores for the remainder of the group continuing in the study, without imputation using actual data.

For secondary continuous efficacy endpoints, similar methods as the primary analysis will be used. For categorical endpoints, when assessments are imputed for data after a subject discontinues from the study, a WOCF method will be used.

Sensitivity analysis of the primary efficacy variable using different methods of imputation for rescue medication may also be performed. Additional sensitivity analysis with different missing


value imputation methods for subjects who drop out of the study may also be performed. All imputation methods for pain intensity will be documented in the SAP.

#### 13.5.8. Analysis of Safety

Safety analyses will be conducted using data from the Safety Population (as defined in Section 13.2).

Safety will be assessed through treatment-emergent AEs (TEAEs); hematologic, biochemical, and urinalysis laboratory parameters; vital signs measurements; ECGs; physical exam, surgical site and neurosensory assessments.

No formal statistical comparisons will be performed for safety endpoints.

#### 13.5.8.1. Adverse Events

Adverse events will be coded by system organ class (SOC) and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA) reporting system. Treatment-emergent AEs are defined as any of the following:

- Non-serious AEs with onset on the date of treatment with the study drug through Day 29 or Early Termination, whichever occurs first;
- Serious AEs with onset on the date of treatment with the study drug through 30 days after Day 29 or Early Termination, whichever occurs first;
- AEs that start before the start of treatment but increase in severity or relationship at the time of or following the start of treatment through Day 29 or Early Termination, whichever occurs first.

The number and percentage of subjects with TEAEs will be displayed for each treatment group by SOC and preferred term. Additionally, TEAEs will be tabulated for each treatment group by severity and by relationship to the study drug. A listing of SAEs will be provided if applicable.

#### 13.5.9. Clinical Laboratory Evaluations

For continuous laboratory parameters, descriptive statistics will be presented for the value at each assessment time and for the changes from baseline by treatment group.

Additionally, clinical laboratory parameters will be categorized as low, normal, or high according to laboratory range specifications and the number and percentage of subjects in each category will be presented in shift tables.

Laboratory values that are outside the normal range will also be flagged in the data listings, along with corresponding normal ranges.


#### 13.5.10. Vital Signs and ECG

Descriptive summaries (mean, SD, median, minimum, and maximum) of actual values and changes from Baseline will be calculated for vital signs and ECG. Detailed description of the analysis will be included in the Study SAP.

The incidence of abnormal ECG findings will be summarized for each visit.

#### 13.5.11. Physical Examination Findings

Physical and Surgical Site examination data will be presented in the listings. Abnormal or clinically significant physical exam and surgical site findings will be recorded as AEs.


#### 14. SITE AND INVESTIGATOR RESPONSIBILITIES

Additional details may be outlined in the Clinical Study Agreement between the sponsor and the investigational site.

#### 14.1. Regulatory and Ethical Considerations

#### 14.1.1. Ethical Conduct of the Study

The Investigator will conduct the study in accordance with GCP and all applicable regulations, including, where applicable, the Declaration of Helsinki. The study will also be carried out in keeping with applicable national and local laws and regulations. This may include an inspection by the Sponsor's representatives and/or regulatory authority's representatives at any time.

## 14.1.2. Ethics Approval

The investigational site's IRB must meet all relevant regulatory requirements. The study protocol and ICF will be reviewed by the IRB prior to enrolling participants into the study; written approval from the committee must be received by the sponsor before drug will be released to the Investigator. The Investigator is responsible for submitting all protocol or ICF changes and SAE reports to the IRB according to local procedures. At a minimum, all SAEs requiring an investigational new drug safety report must be immediately reported.

In accordance with applicable local regulatory requirements, the Investigator may be obligated to provide periodic safety updates on the conduct of the study at his or her research site and notification of study closure to the IRB. Such periodic safety updates and notifications are the responsibility of the Investigator and not of the Sponsor. The Sponsor will be provided with copies of all notifications sent to the IRB.

All relevant correspondence from the IRB will be forwarded by the respective study site to the Sponsor in a timely fashion.

#### 14.1.3. Subject Informed Consent

The Investigator (or authorized designee) will ensure that the participant (or the participant's legal representative) is given full and adequate oral and written information about the nature, purpose, potential and possible risks and benefits of the study. Each prospective subject will receive an IRB-approved ICF that summarizes the pertinent study information and will be given ample time to read the form and ask questions about the study. All information is to be provided in a language understandable to the participant and must not include any language that waives the participant's legal rights. Prospective participants must also be informed of their right to withdraw consent without prejudice at any time during the study. If the participant chooses to participate, he/she must sign the ICF before any study-related procedures are performed.


Significant changes to the protocol or product safety information may require a revision of the ICF, which must be reviewed and signed by all applicable study participants.

The time that informed consent is obtained must be documented. The Investigator must maintain the original, signed ICF in the participant's source documents. A copy of the signed ICF must be given to the study participant.

## 14.2. Privacy and Confidentiality

The Investigator is responsible for complying with applicable privacy regulations, per his or her jurisdiction. Only information identified in this protocol will be collected. The information collected will only be used for the purposes identified in this protocol.

To ensure anonymity and to limit disclosure, participants will be assigned a unique identifier at their first assessment. This identifier will be cross-referenced in the participant's chart. The identifier will not contain any potentially identifiable information. An identifier log will be maintained, linking each participant's name to the corresponding identifier. This log will be stored at the research site in a secure location.

The knowledge gained through this study is the property of the Sponsor. The Sponsor, representatives and affiliated companies of the Sponsor, the IRB, and regulatory agencies (such as the United States FDA) may inspect medical records related to the study to check the validity and accuracy of the data gathered in this study. Participant medical records (with participant's initials and/or date of birth) may be copied. Confidentiality of participant records will be maintained except where release of information is required by law.

The results of this study will be reported in such a manner that participants will not be identifiable in any way. Published reports or presentations will refer to grouped data or coded individual data and not to any identifiable individuals. Study reports sent to the Sponsor or drug regulatory agencies will not include participant names.

By signing the ICF, the participant consents to the collection, access, use, and disclosure of his or her information as described in the ICF document. If a participant withdraws consent, some of the subject's information may still be collected, used, and disclosed by those involved in this study, per applicable laws.

By signing this protocol, the Investigator affirms that he or she will maintain in confidence information furnished to him or her by the Sponsor and will divulge such information to his or her respective IRB or IEC under an appropriate understanding of confidentiality with such board. All data will be considered the sole property of the Sponsor. Please refer to the Clinical Study Agreement for details.


## 14.3. Study and Site Closure

Upon completion of the study, all study data will be provided to the Sponsor following review of site study records for completeness, and data clarifications and resolutions. Accounting, reconciliation, and final disposition of used and unused study drugs, treatment codes, and emergency code break envelopes will be performed, as applicable.

In addition, the Sponsor reserves the right to temporarily suspend or prematurely discontinue this study at any time and for any reason. If such action is taken, the Sponsor will discuss this with the Investigator (including the reasons for taking such action) at that time. The Sponsor will promptly inform any other investigators and/or institutions conducting the study, if the study is suspended or terminated for safety reasons and will inform the regulatory authorities of the suspension or termination of the study and the reason(s) for the action. If required by applicable regulations, the Investigator will inform the IRB promptly and provide the study participants with the reason for the suspension or termination. If the study is prematurely discontinued, all study data will be returned to the Sponsor.

## 14.4. Regulatory Documents and Records Retention

The Investigator is responsible for creating and/or maintaining all study documentation required by 21 CFR 50, 54, 56 and 312, ICH E6 section 8, as well as any other documentation defined in the protocol or Clinical Study Agreement. The Investigator must provide key documents to the Sponsor prior to the start of the study. A complete list of required regulatory documents will be supplied by the Sponsor or its representative.

Federal and local regulations require that the Investigator retain a copy of all regulatory documents and records that support the data for this study for whichever of the following is the longest period of time:

- A period of 2 years following the final date of approval by the FDA or other regulatory agency of the study drug for the purposes that were the subject of the investigation; or
- A period of 5 years following the date on which the results of the investigation were submitted to the FDA or other regulatory agency in support of, or as part of, an application for a research or marketing permit for the study drug for the purposes that were the subject of the investigation.

The Sponsor will notify investigators once one of the above 2 timeframes has been satisfied.

If the investigation does not result in the submission of the data in support of, or as part of, an application for a research or marketing permit, records must be retained for a period of 2 years following notification by the Sponsor that the entire clinical investigation (not merely the Investigator's portion) is completed, terminated, or discontinued or 2 years following withdrawal


of the Investigational New Drug application/Clinical Trial Authorization or request for marketing approval (New Drug Application/Marketing Authorization Application).

If the Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Study records should not be destroyed without consultation with the Sponsor.

## 14.5. Delegation of Responsibilities and Adequate Resources

The Investigator should have adequate time to conduct the study properly and should have an adequate number of qualified staff to assist with the conduct of the study.

The term "Investigator" used throughout this protocol refers to the principal investigator and/or qualified sub-investigators. However, the Investigator may delegate responsibilities to other investigational site personnel. The Investigator shall delegate tasks only to individuals qualified by education, training and experience to perform the delegated tasks. The Investigator shall have direct oversight of all delegated activities and shall document delegation of responsibilities. The Investigator is responsible for ensuring all delegated staff has been properly trained on the protocol and their assigned study responsibilities. A delegation log identifying all delegated duties and the individual to whom they have been delegated will be maintained at the investigational site.

#### 14.6. Protocol Amendments

Approval of a protocol amendment by the Investigator's IRB must be obtained before implementation of the protocol amendment, unless a change is necessary to eliminate an apparent immediate hazard to the participant or when the change involves logistical or administrative aspects of the study. The protocol amendment must be signed and dated by both the Sponsor and the Investigator. The Sponsor or designee will submit protocol amendments to the appropriate regulatory authorities, if required.

#### 14.7. Financial Disclosure

Clinical investigators are required to provide financial disclosure information for the submission of certification or disclosure statements required under 21 CFR § 54. As defined in 21 CFR § 54.2, a clinical investigator is a listed or identified investigator or sub-investigator who is directly involved in the treatment or evaluation of research participants. The term also includes the spouse and each dependent child of the investigator. In addition, investigators must promptly update financial disclosure information if any relevant changes occur during the course of the investigation and for 1 year following completion of the study


## 15. INVESTIGATOR PROTOCOL AGREEMENT PAGE

A Phase 2, Randomized, Double-blind, Placebo-Controlled Efficacy, Pharmacokinetics and Safety Study of CA-008 in Subjects Undergoing Total Knee Arthroplasty

| Version: 3.2 | | |
|---|---|---|
| Date: 19 February 2019 | | |
| I have read this protocol and I agree to conduct t<br>protocol and with all applicable government<br>Conference on Harmonisation/Good Clinical Pract | regulations and | |
| Principal Investigator's Name (please print or type) | | |
| Principal Investigator's Signature | | (DD-MMM- |

YYYY)


#### 16. REFERENCES

- 1. Babbar S, Marier JF, Mouksassi MS et al. Pharmacokinetic analysis of capsaicin after topical administration of a high-concentration capsaicin patch to patients with peripheral neuropathic pain. *Ther Drug Monit* 2009; 31:502-10.
- 2. Caterina MJ, Julius D. The vanilloid receptor: a molecular gateway to the pain pathway. *Annu Rev Neurosci* 2001 24:487-517.
- 3. Cullom C, Weed JT. Anesthetic and analgesic management for outpatient knee arthroplasty. *Curr Pain Headache Rep*
- 4. Dudley-Cash AI, Brennan TJ. The effect of low concentration capsaicin infiltration on acute pain from incision. *Soc Neuroscience* 2012, New Orleans.
- 5. Hartrick CT, Pestano C, Carlson N, Hartrick S. Capsaicin instillation for postoperative pain following total knee arthroplasty: a preliminary report of a randomized, double-blind, parallel-group, placebo-controlled, multicentre trial. *Clin Drug Investig* 2011 Dec 1;31(12):877-82.
- 6. Sankineani SR, Reddy ARC, Eachempati KK et al. Comparison of adductor canal block and IPACK block (interspace between the popliteal artery and the capsule of the posterior knee) with adductor canal block alone after total knee arthroplasty: a prospective control trial on pain and knee function in immediate postoperative period. *Eur J Orthop Surg Traumatol* 2018; doi: 10.1007/s00590-018-2218-7 [Epub ahead of print]
- 7. Suresh D, Srinivasan K. Tissue distribution & elimination of capsaicin, piperine & curcumin following oral intake in rats. *Indian J Med Res* 2010; 131:682-91.
- 8. Surh YJ, Lee RC, Park KK et al. Chemoprotective effects of capsaicin and diallyl sulfide against mutagenesis or tumorigenesis by vinyl carbamate and N-nitrosodimethylamine. *Carcinogenesis* 1995: 16:2467-71.
- 9. Tominaga, M., Caterina, M.J., Malmberg, A.B., Rosen, T.A., Gilbert, H., Skinner, K., Raumann, B.E., Basbaum, A.I., Julius, D., 1998. The cloned capsaicin receptor integrates multiple pain-producing stimuli. *Neuron* 21, 531–543.


#### 17. APPENDICES

## 17.1. Appendix A: American Society of Anesthesiologists Physical Status Classification System (ASA Class)

| | Definition | Examples, including, but not limited to: |
|---|---|---|
| ASA I | A normal healthy patient | Healthy, non-smoking, no or minimal alcohol use |
| ASA II | A patient with mild systemic disease | Mild diseases only without substantive functional limitations. Examples include (but not limited to): current smoker, social alcohol drinker, pregnancy, obesity (30 < BMI < 40), well-controlled DM/HTN, mild lung disease |
| ASA III | A patient with severe systemic disease | Substantive functional limitations; One or more moderate to severe diseases. Examples include (but not limited to): poorly controlled DM or HTN, COPD, morbid obesity (BMI ≥40), active hepatitis, alcohol dependence or abuse, implanted pacemaker, moderate reduction of ejection fraction, ESRD undergoing regularly scheduled dialysis, premature infant PCA < 60 weeks, history (>3 months) of MI, CVA, TIA, or CAD/stents. |
| ASA IV | A patient with severe systemic disease that is a constant threat to life | Examples include (but not limited to): recent ( < 3 months) MI, CVA, TIA, or CAD/stents, ongoing cardiac ischemia or severe valve dysfunction, severe reduction of ejection fraction, sepsis, DIC, ARD or ESRD not undergoing regularly scheduled dialysis |
| ASA V | A moribund patient who is not expected to survive without the operation | Examples include (but not limited to): ruptured abdominal/thoracic aneurysm, massive trauma, intracranial bleed with mass effect, ischemic bowel in the face of significant cardiac pathology or multiple organ/system dysfunction |
| ASA VI | A declared brain-dead patient whose organs are being removed for donor purposes | |

<sup>\*</sup>The addition of "E" denotes Emergency surgery: (An emergency is defined as existing when delay in treatment of the patient would lead to a significant increase in the threat to life or body part)

Available at: https://www.asahq.org/resources/clinical-information/asa-physical-status-classification-system


## 17.2. Appendix B: 0 to 10 Numerical Rating Scale of Pain Intensity (NRS)

| | Pain Intensity - Numerical Rating Scale (NRS) | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | On a scale of 0-10, please rate your pain by marking the appropriate box that best describes your pain NOW. | | | | | | | | | | |
| | □0 | □1 | □2 | □3 | □4 | □5 | □6 | □7 | □8 | □9 | □10 |
| | No Pain | | | | | | | | | | Worst pain<br>imaginable |
| 5 | Subject Initials: | | | | | | | | | | |

# 17.3. Appendix C: Assessment of Rebound Pain at the Surgical Site (Rebound Pain)

| Rebound Pain | |
|---|---|
| Ask the subject the following question: "Have you noticed any increase in pain at the surgical s (rebound pain) since your last visit?" | |
| □ yes □ | no |
| Subject Initials: | |

Rebound pain may also be characterized as worsening pain at the surgical site.


# 17.4. Appendix D: Patient Global Evaluation [of Satisfaction with Study Treatment] (PGE)

| Patient Global Evaluation (PGE) |
|---|
| <i>Instructions to Subject:</i> Please respond to the question below. When completed, please initial at the bottom of the page. |
| How would you rate your satisfaction with the study treatment that you received during surgery for postop pain? |
| (Mark one box) |
| □ Excellent (3) |
| □ Good (2) |
| □ Fair (1) □ Page (0) |
| □ Poor (0) Subject Initials: |


# 17.5. Appendix E: Investigator Global Evaluation of Study Treatment] (IGE)

| Investigator Global Evaluation (IGE) |
|---|
| <i>Instructions to Investigator</i> : Please respond to the question below. When completed, please initial at the bottom of the page. |
| How would you rate the study treatment that this patient received during surgery for pain? |
| (Mark one box) |
| □ Excellent (3) |
| □ Good (2) |
| ☐ Fair (1) |
| □ Poor (0) |
| Investigator Initials: |


## 17.6. Appendix F: Surgical Site Assessment

The investigator should grade the level of satisfaction with wound healing using this 0-10 scale with 0=completely unsatisfied and 10=completely satisfied.

| Post-Operative Surgical Site Assessment | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| <i>Instructions to Investigator</i> : Please respond to the question below. When completed, please initial at the bottom of the page. | | | | | | | | | | |
| On a scale of 0 to 10, please rate your clinical satisfaction with the wound healing. | | | | | | | | | | |
| □0 | □1 | □2 | □3 | □4 | □5 | □6 | □7 | □8 | □9 | □10 |
| Completely <u>unsatisfied</u> Completely <u>satisfied</u> | | | | | | | | | | |
| Investiga | tor Initia | als: | | | | | | | | |

In the assessment of satisfaction with wound healing, it should be performed with what is typically observed for surgeries of this type in the investigator's clinical opinion. The surgical wound adverse event grading scale which follows may be helpful is there is an atypical or abnormal finding.


## 17.7. Appendix G: Surgical Wound Adverse Event Grading Guide

The investigator may find the following table to be a useful guide for grading specific AEs using this 4-point categorical scale for common wound complications. The investigator should use clinical discretion in determining whether the particular parameter is atypical or unusual compared to what is expected as a typical healing process.

| PARAMETER | GRADE | DESCRIPTION |
|---|---|---|
| | 0 | NONE |
| | 1 | VERY SLIGHT (BARELY PERCEPTIBLE) |
| ERYTHEMA | 2 | SLIGHT (WELL DEFINED) |
| ERTTIENT | 3 | MODERATE |
| | 4 | SEVERE (BEET REDNESS) TO SLIGHT ESCHAR FORMATION (INJURIES IN DEPTH) |
| | 0 | NONE |
| | 1 | SEROUS |
| DRAINAGE | 2 | SEROSANGUINOUS |
| | 3 | BLOODY |
| | 4 | PURULENT |
| | 0 | NONE |
| | 1 | VERY SLIGHT (BARELY PERCEPTIBLE) |
| EDEMA | 2 | SLIGHT (EDGES WELL DEFINED) |
| <b>LDL</b> IVILL | 3 | MODERATE (RAISED APPROXIMATELY 1 MM) |
| | 4 | SEVERE (RAISED > 1 MM AND BEYOND AREA OF EXPOSURE) |
| | 0 | NONE |
| | 1 | MINIMAL |
| INDURATION | 2 | MILD (SPONGY TISSUE) |
| | 3 | MODERATE (FIRM, WARM) |
| | 4 | SEVERE (HARD, RED, HOT, CREPITUS) |
| | 0 | NONE |
| | 1 | MINIMAL |
| HEMATOMA | 2 | MILD |
| | 3 | MODERATE |
| | 4 | SEVERE |


## 17.8. Appendix H: Neurosensory Examination Form

| Subject Number | | Subject I | nitials | Date:// 2 0<br>(DD-MMM-20YY) | | Protoco | ol Number | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | (00-101101101-2011) | | | CA- | PS-203 |
| A STATE OF THE STA | uctions to the Investigo<br>uestions below. Please er | | | | | | | | te) and answer |
| Time | of Assessment: | н | : M | M | - 1 | Not Done, Reas | son: | Investigator Initi | ials: |
| Neur | osensory Examination o | f the TKA s | ite using the | e opposite | knee as a cont | rol site | | | |
| 1. | Was the Neurosensory Exan | n completed | ? | ☐ Yes | . □ No | | | Control site: | |
| | | Ceph | nalad to w | ound | Cauc | lad to wou | ınd | Opposite | knee |
| 2. Visual Exam of the Surgical site: | | □ Normal | ☐ Abnormal, | describe: | □ Normal | ☐ Abnormal, | describe: | If abnormal in co<br>to the control sit<br>whether it is red<br>absent and for b<br>stimulation, add | te, note<br>uced or<br>rush |
| 3. | Light touch | □ Normal □ Reduced □ Absent □ Normal □ Reduced □ Abser | | ☐ Absent | whether there is | | | | |
| 4. Von Frey stimulation | | □ Normal | ☐ Reduced | ☐ Absent | □Normal | ☐ Reduced | ☐ Absent | Note that allody<br>from a normally | • |
| 5. | Brush stimulation | □ Normal | ☐ Reduced | ☐ Absent | □ Normal | ☐ Reduced | ☐ Absent | stimulus. | · |
| | | in (Allodynia) | | □P | ain (Allodynia) | | | | |

Neurosensory testing should be performed in an area approximately 3 to 5 cm above and below the surgical incision site in all 4 quadrants of the leg compared to the control site. The instructions below may assist the investigator or designee in performing neurosensory testing.

- Monofilament (von Frey) Testing: For this examination, the filament should initially be prestressed (4-6 perpendicular applications to the dorsum of the examiner's first finger). The filament is then applied perpendicularly at the location to be assessed and briefly, (<1 second) with even pressure. When the filament bends, the force of 10 grams has been applied. The subject, whose eyes are closed, is asked to respond yes if he / she feels the filament. Eight correct responses out of 10 applications is considered normal: one to seven correct responses indicate reduced sensation and no correct responses translates into absent sensation.
- **Testing for Allodynia:** performed at the location to be assessed using a foam brush. Note that allodynia testing is best assessed by using the foam brush, and while it may be elicited using von Frey filament testing, document presence of allodynia only with brush stimulation. For **allodynia assessment** the foam brush will be lightly stroked 3 times across the skin in the location to be assessed. Subject will be asked to compare sensation to the control site just distal to the costal margin. If the sensation is described as painful or very unpleasant then allodynia will be reported as present. If sensation is slightly


unpleasant or mildly irritating compared to the control area then hyperaesthesia will be reported as present. If subject reports the stimulus as the same as the control area then sensation will be reported as normal. If sensation is less than the control area then sensation will be reported as reduced, and if sensation is not felt as all then it will be reported as absent.


## 17.9. Appendix I: Toxicity Grading Scale for Clinical Laboratory Abnormalities

The following tables are excerpted from the Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. The grading system can be "useful in defining a particular study's stopping rules (e.g., a certain number of adverse events, as defined in the table, may call for stopping the study.)"

The Guidance may be found in its entirety at: https://www.fda.gov/downloads/BiologicsBloodVaccines/ucm091977.

For clinical laboratory values not covered in this Guidance, the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (November 27, 2017) may be useful as a reference. CTCAE v5.0 and prior versions are available at

https://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm.


#### B. Tables for Laboratory Abnormalities

The laboratory values provided in the tables below serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.

| Serum * | Mild (Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4)** |
|---|---|---|---|---|
| Sodium – Hyponatremia mEq/L | 132 – 134 | 130-131 | 125 – 129 | < 125 |
| Sodium – Hypernatremia mEq/L | 144 – 145 | 146 - 147 | 148-150 | > 150 |
| Potassium – Hyperkalemia mEq/L | 5.1 - 5.2 | 5.3 - 5.4 | 5.5 - 5.6 | > 5.6 |
| Potassium – Hypokalemia mEq/L | 3.5 – 3.6 | 3.3 – 3.4 | 3.1 - 3.2 | < 3.1 |
| Glucose - Hypoglycemia mg/dL | 65 – 69 | 55 – 64 | 45 – 54 | < 45 |
| Glucose – Hyperglycemia | | | | Insulin |
| Fasting - mg/dL | 100 - 110 | 111 - 125 | >125 | requirements or |
| Random – mg/dL | 110 – 125 | 126-200 | >200 | hyperosmolar<br>coma |
| Blood Urea Nitrogen<br>BUN mg/dL | 23 – 26 | 27 – 31 | > 31 | Requires<br>dialysis |
| Creatinine - mg/dL | 1.5 – 1.7 | 1.8 – 2.0 | 2.1 – 2.5 | > 2.5 or requires<br>dialysis |
| Calcium - hypocalcemia mg/dL | 8.0 - 8.4 | 7.5 – 7.9 | 7.0 - 7.4 | < 7.0 |
| Calcium - hypercalcemia mg/dL | 10.5 - 11.0 | 11.1 - 11.5 | 11.6-12.0 | > 12.0 |
| Magnesium - hypomagnesemia mg/dL | 1.3 – 1.5 | 1.1 – 1.2 | 0.9 - 1.0 | < 0.9 |
| Phosphorous – hypophosphatemia<br>mg/dL | 2.3 – 2.5 | 2.0 – 2.2 | 1.6-1.9 | < 1.6 |
| CPK - mg/dL | 1.25 – 1.5 x<br>ULN*** | 1.6 – 3.0 x ULN | 3.1 –10 x ULN | > 10 x ULN |
| Albumin - Hypoalbuminemia g/dL | 2.8 - 3.1 | 2.5 - 2.7 | < 2.5 | _ |
| Total Protein - Hypoproteinemia g/dL | 5.5 - 6.0 | 5.0 - 5.4 | < 5.0 | _ |
| Alkaline phosphate –<br>increase by factor | 1.1 – 2.0 x ULN | 2.1 – 3.0 x ULN | 3.1 – 10 x ULN | > 10 x ULN |
| Liver Function Tests –ALT, AST<br>increase by factor | 1.1 – 2.5 x ULN | 2.6 - 5.0 x ULN | 5.1 – 10 x ULN | > 10 x ULN |
| Bilirubin - when accompanied | 1.1 - 1.25 x ULN | 1.26 - 1.5 x ULN | 1.51 - 1.75 x ULN | > 1.75 x ULN |
| by any increase in Liver Function Test<br>increase by factor | | | | |
| Bilirubin – when Liver Function Test<br>is normal; increase by factor | 1.1 – 1.5 x ULN | 1.6 – 2.0 x ULN | 2.0 – 3.0 x ULN | > 3.0 x ULN |
| Cholesterol | 201 - 210 | 211-225 | > 226 | _ |
| Pancreatic enzymes - amylase, lipase | 1.1-1.5 x ULN | 1.6-2.0 x ULN | 2.1 - 5.0 x ULN | > 5.0 x ULN |

<sup>\*</sup> The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.


<sup>\*\*</sup> The clinical signs or symptoms associated with laboratory abnormalities might result in characterization of the laboratory abnormalities as Potentially Life Threatening (Grade 4). For example, a low sodium value that falls within a grade 3 parameter (125-129 mE/L) should be recorded as a grade 4 hyponatremia event if the subject had a new seizure associated with the low sodium value.

<sup>\*\*\*</sup>ULN" is the upper limit of the normal range.
| Hematology * | Mild (Grade 1) | Moderate<br>(Grade 2) | Severe (Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Hemoglobin (Female) - gm/dL | 11.0 - 12.0 | 9.5 - 10.9 | 8.0 - 9.4 | < 8.0 |
| Hemoglobin (Female) | Any decrease - 1.5 | 1.6-2.0 | 2.1 - 5.0 | > 5.0 |
| change from baseline value - gm/dL | | | | |
| Hemoglobin (Male) - gm/dL | 12.5 - 13.5 | 10.5 - 12.4 | 8.5 - 10.4 | < 8.5 |
| Hemoglobin (Male) | Any decrease - 1.5 | 1.6-2.0 | 2.1-5.0 | > 5.0 |
| change from baseline value - gm/dL | | | | |
| WBC Increase - cell/mm <sup>3</sup> | 10,800 - 15,000 | 15,001 - 20,000 | 20,001 - 25,000 | > 25,000 |
| WBC Decrease - cell/mm <sup>3</sup> | 2,500 - 3,500 | 1,500 - 2,499 | 1,000 - 1,499 | < 1,000 |
| Lymphocytes Decrease - cell/mm <sup>3</sup> | 750 - 1,000 | 500 - 749 | 250 - 499 | < 250 |
| Neutrophils Decrease - cell/mm <sup>3</sup> | 1,500 - 2,000 | 1,000 - 1,499 | 500 - 999 | < 500 |
| Eosinophils - cell/mm <sup>3</sup> | 650 - 1500 | 1501 - 5000 | > 5000 | Hypereosinophilic |
| Platelets Decreased - cell/mm <sup>3</sup> | 125,000 - 140,000 | 100,000 - 124,000 | 25,000 - 99,000 | < 25,000 |
| PT – increase by factor | 1.0 - 1.10 x | . 1.11 - 1.20 x ULN | 1.21 - 1.25 x ULN | > 1.25 ULN |
| (prothrombin time) | ULN** | | | |
| PTT - increase by factor | 1.0 - 1.2 x ULN | 1.21 - 1.4 x ULN | 1.41 - 1.5 x ULN | > 1.5 x ULN |
| (partial thromboplastin time) | | | | |
| Fibrinogen increase - mg/dL | 400 - 500 | 501 - 600 | > 600 | _ |
| Fibrinogen decrease - mg/dL | 150 - 200 | 125 - 149 | 100-124 | < 100 or associated |
| | | | | with gross bleeding |
| | | | | or disseminated |
| | | | | intravascular |
| | | | | coagulation (DIC) |

The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate. "ULN" is the upper limit of the normal range.

| Urine * | Mild (Grade 1) | Moderate<br>(Grade 2) | Severe (Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Protein | Trace | 1+ | 2+ | Hospitalization or<br>dialysis |
| Glucose | Trace | 1+ | 2+ | Hospitalization for<br>hyperglycemia |
| Blood (microscopic)— red blood cells per high power field (rbc/hpf) | 1 - 10 | 11-50 | > 50 and/or gross<br>blood | Hospitalization or<br>packed red blood<br>cells (PRBC)<br>transfusion |

The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.


# 17.10. Appendix J: Toxicity Grading Scale for Clinical Vital Sign Abnormalities

The following guidance is excerpted from the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (November 27, 2017) as a reference. CTCAE v5.0 and prior versions are available at https://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm.

The grading system can be "useful in defining a particular study's stopping rules (e.g., a certain number of adverse events, as defined in the table, may call for stopping the study.)"

#### Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Publish Date: November 27, 2017

#### Introduction

The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term.

#### SOC

System Organ Class (SOC), the highest level of the MedDRA<sup>1</sup> hierarchy, is identified by anatomical or physiological system, etiology, or purpose (e.g., SOC Investigations for laboratory test results). CTCAE terms are grouped by MedDRA Primary SOCs. Within each SOC, AEs are listed and accompanied by descriptions of severity (Grade).

#### CTCAE Terms

An Adverse Event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may <u>not</u> be considered related to the medical treatment or procedure. An AE is a term that is a unique representation of a specific event used for medical documentation and scientific analyses. Each CTCAE v4.0 term is a MedDRA LLT (Lowest Level Term).

#### Grades

Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:

Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.

Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting ageappropriate instrumental ADL\*.

Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL\*\*.

Grade 4 Life-threatening consequences; urgent intervention indicated.

Grade 5 Death related to AE.

A Semi-colon indicates 'or' within the description of the grade.

A single dash (-) indicates a Grade is not available. Not all Grades are appropriate for all AEs. Therefore, some AEs are listed with fewer than five options for Grade selection.

#### Grade 5

Grade 5 (Death) is not appropriate for some AEs and therefore is not an option.

#### Definitions

A brief Definition is provided to clarify the meaning of each AE term. A single dash (-) indicates a Definition is not available.

#### **Navigational Notes**

A Navigational Note is used to assist the reporter in choosing a correct AE. It may list other AEs that should be considered in addition to <u>or</u> in place of the AE in question. A single dash (-) indicates a Navigational Note has not been defined for the AE term.

#### Activities of Daily Living (ADL)

\*Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

\*\*Self care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

#### These excerpts are from various sections within CTCAE v5.0:

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Fever | 38.0 - 39.0 degrees C (100.4 - | >39.0 - 40.0 degrees C (102.3 - | >40.0 degrees C (>104.0 | >40.0 degrees C (>104.0 | Death |
| | 102.2 degrees F) | 104.0 degrees F) | degrees F) for <=24 hrs | degrees F) for >24 hrs | |
| Definition: A disorder character | zed by elevation of the body's temp | perature above the upper limit of no | ormal. | | |
| Navigational Note: - | | | | | |
| Sinus tachycardia | Asymptomatic, intervention | Symptomatic; non-urgent | Urgent medical intervention | - | - |
| | not indicated | medical intervention indicated | indicated | | |
| Definition: A disorder characteri | zed by a dysrhythmia with a heart r | ate greater than 100 beats per min | ute that originates in the sinus nod | le. | |
| Navigational Note: - | | | | | |
| Sinus bradycardia | Asymptomatic, intervention | Symptomatic, intervention | Symptomatic, intervention | Life-threatening | Death |
| | not indicated | not indicated; change in | indicated | consequences; urgent | |
| | | medication initiated | | intervention indicated | |
| Definition: A disorder characterized by a dysrhythmia with a heart rate less than 60 beats per minute that originates in the sinus node. | | | | | |
| Navigational Note: - | | | | | |

<sup>&</sup>lt;sup>1</sup> CTCAE v5.0 incorporates certain elements of the MedDRA terminology. For further details on MedDRA refer to the MedDRA MSSO Web site (https://www.meddra.org/)

| Hypertension | Adult: Systolic BP 120 - 139 mm Hg or diastolic BP 80 - 89 mm Hg; Pediatric: Systolic/diastolic BP >90th percentile but< 95th percentile; Adolescent: BP ≥120/80 even if < 95th percentile | Adult: Systolic BP 140 - 159 mm Hg or diastolic BP 90 - 99 mm Hg if previously WNL; change in baseline medical intervention indicated; recurrent or persistent (>=24 hrs); symptomatic increase by >20 mm Hg (diastolic) or to >140/90 mm Hg; monotherapy indicated initiated; Pediatric and adolescent: Recurrent or persistent (>=24 hrs) BP >ULN; monotherapy indicated; systolic and /or diastolic BP between the 95th percentile and 5 mmHg above the 99th percentile; Adolescent: Systolic between | Adult: Systolic BP >= 160 mm Hg or diastolic BP >= 100 mm Hg; medical intervention indicated; more than one drug or more intensive therapy than previously used indicated; Pediatric and adolescent: Systolic and/or diastolic > 5 mmHg above the 99th percentile | Adult and Pediatric: Life-<br>threatening consequences<br>(e.g., malignant hypertension,<br>transient or permanent<br>neurologic deficit,<br>hypertensive crisis); urgent<br>intervention indicated | Death |
|---|---|---|---|---|---|
| | | 130-139 or diastolic between | | | |
| | | 80-89 even if < 95th percentile | | | |
| Definition: A disorder charac | cterized by a pathological increase in bl | The state of the s | 1 | | ' |
| Navigational Note: - | , - F | | | | |
| Hypotension | Asymptomatic, intervention | Non-urgent medical | Medical intervention | Life-threatening | Death |
| ** | not indicated | intervention indicated | indicated; hospitalization | consequences and urgent | |
| | | | indicated | intervention indicated | |
| Definition: A disorder charac | terized by a blood pressure that is belo | ow the normal expected for an indiv | idual in a given environment. | | • |
| Navigational Note: - | | - | - | | |
| Hypoxia | - | Decreased oxygen saturation | Decreased oxygen saturation | Life-threatening airway | Death |
| | | with exercise (e.g., pulse | at rest (e.g., pulse oximeter | compromise; urgent | |
| | | oximeter <88%); intermittent | <88% or PaO2 <=55 mm Hg) | intervention indicated (e.g., | |
| | | supplemental oxygen | | tracheotomy or intubation) | |
| Definition: A disorder charac | cterized by a decrease in the level of ox | | 1 | , | ' |
| Navigational Note: - | | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | | | |
| Havigational Note. | T | T | 1 | T. | |


# 17.11. Appendix K: Toxicity Grading Scale for Systemic (General) Adverse Events

The following table is excerpted from the Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. The grading system can be "useful in defining a particular study's stopping rules (e.g., a certain number of adverse events, as defined in the table, may call for stopping the study.)"

The Guidance may be found in its entirety at: https://www.fda.gov/downloads/BiologicsBloodVaccines/ucm091977.

The investigator may find this useful for grading common systemic (general) TEAEs reported after surgery.

| Systemic (General) | Mild (Grade 1) | Moderate(Grade 2) | Severe (Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Nausea/vomiting | No interference<br>with activity or 1 – 2<br>episodes/24 hours | Some interference<br>with activity or > 2<br>episodes/24 hours | Prevents daily<br>activity, requires<br>outpatient IV<br>hydration | ER visit or<br>hospitalization for<br>hypotensive shock |
| Diarrhea | 2 – 3 loose stools or<br>< 400 gms/24 hours | 4-5 stools or<br>400-800 gms/24<br>hours | 6 or more watery<br>stools or<br>> 800gms/24 hours<br>or requires<br>outpatient IV<br>hydration | ER visit or<br>hospitalization |
| Headache | No interference with activity | Repeated use of non-<br>narcotic pain<br>reliever > 24 hours or<br>some interference<br>with activity | Significant; any<br>use of narcotic<br>pain reliever or<br>prevents daily<br>activity | ER visit or<br>hospitalization |
| Fatigue | No interference with activity | Some interference with activity | Significant;<br>prevents daily<br>activity | ER visit or<br>hospitalization |
| Myalgia | No interference with activity | Some interference with activity | Significant;<br>prevents daily<br>activity | ER visit or<br>hospitalization |


# 17.12. Appendix L: Ropivacaine Dosage Recommendations

# **Dosage Recommendations**

| | C | onc. | Volume | Dose | Onset | Duration |
|---|---|---|---|---|---|---|
| | mg/mL | (%) | mL | mg | min | hours |
| SURGICAL ANESTHES | IA | | | | | |
| Lumbar Epidural | 5 | (0.5%) | 15 to 30 | 75 to 150 | 15 to 30 | 2 to 4 |
| Administration | 7.5 | (0.75%) | 15 to 25 | 113 to 188 | 10 to 20 | 3 to 5 |
| Surgery | 10 | (1%) | 15 to 20 | 150 to 200 | 10 to 20 | 4 to 6 |
| Lumbar Epidural | 5 | (0.5%) | 20 to 30 | 100 to 150 | 15 to 25 | 2 to 4 |
| Administration<br>Cesarean Section | 7.5 | (0.75%) | 15 to 20 | 113 to 150 | 10 to 20 | 3 to 5 |
| Thoracic Epidural<br>Administration<br>Surgery | 5<br>7.5 | (0.5%)<br>(0.75%) | 5 to 15<br>5 to 15 | 25 to 75<br>38 to 113 | 10 to 20<br>10 to 20 | n/a*<br>n/a* |
| Major Nerve<br>Block <sup>†</sup> | 5 | (0.5%) | 35 to 50 | 175 to 250 | 15 to 30 | 5 to 8 |
| (e.g., brachial plexus block) | 7.5 | (0.75%) | 10 to 40 | 75 to 300 | 10 to 25 | 6 to 10 |
| Field Block<br>(e.g., minor nerve<br>blocks and infiltration) | 5 | (0.5%) | 1 to 40 | 5 to 200 | 1 to 15 | 2 to 6 |


# 17.13. Appendix M: Knee Injury and Osteoarthritis Outcome Survey (KOOS)

Knee injury and Osteoarthritis Outcome Score (KOOS), English version LK1.0

| | KOO | S KNEE S | URVEY | |
|---|---|---|---|---|
| Today's date: _ | / | / Date of t | oirth:/_ | |
| Name: | | | | |
| <b>INSTRUCTIONS:</b> This survey asks for your view about your knee. This information will help us keep track of how you feel about your knee and how well you are able to perform your usual activities. Answer every question by ticking the appropriate box, only one box for each question. If you are unsure about how to answer a question, please give the best answer you can. | | | | |
| Symptoms These questions should be answered thinking of your knee symptoms during the last week. | | | | |
| S1. Do you have s | welling in you<br>Rarely | r knee?<br>Sometimes | Often | Always |
| S2. Do you feel gr<br>moves? | | licking or any other | type of noise w | |
| Never | Rarely | Sometimes | □ □ | Always |
| S3. Does your known Never | ee catch or han<br>Rarely | g up when moving<br>Sometimes | Often | Always |
| S4. Can you straig | ghten your kne<br>Often | e fully?<br>Sometimes | Rarely | Never |
| S5. Can you bend Always | your knee full<br>Often | y? Sometimes | Rarely | Never |
| Stiffness The following questions concern the amount of joint stiffness you have experienced during the last week in your knee. Stiffness is a sensation of restriction or slowness in the ease with which you move your knee joint. | | | | |
| S6. How severe is | your knee joir<br>Mild | nt stiffness after firs<br>Moderate | st wakening in th<br>Severe | e morning? Extreme |
| S7. How severe is | your knee stif | fness after sitting, l | ying or resting la | ater in the day? Extreme |


| Pain P1. How often do yo Never | ou experience l<br>Monthly | knee pain?<br>Weekly | Daily | Always | |
|---|---|---|---|---|---|
| What amount of I following activities | | ave you experie | enced the last | week during the | • |
| P2. Twisting/pivotin | ng on your knee<br>Mild | e<br>Moderate | Severe | Extreme | |
| P3. Straightening kn | Mild | Moderate | Severe | Extreme | |
| P4. Bending knee fu | illy<br>Mild | Moderate | Severe | Extreme | |
| P5. Walking on flat | surface<br>Mild | Moderate | Severe | Extreme | |
| P6. Going up or dow | vn stairs<br>Mild | Moderate | Severe | Extreme | |
| P7. At night while in None | n bed<br>Mild | Moderate | Severe | Extreme | |
| P8. Sitting or lying None | Mild | Moderate | Severe | Extreme | |
| P9. Standing upright | t<br>Mild | Moderate | Severe | Extreme | |
| Function, daily live. The following questability to move an activities please in last week due to y | stions concer<br>round and to<br>ndicate the d | look after you | irself. For eacl | h of the following | 3 |
| A1. Descending stai | rs<br>Mild | Moderate | Severe | Extreme | |
| A2. Ascending stairs | s<br>Mild | Moderate | Severe | Extreme | |

For each of the following activities please indicate the degree of difficulty you have experienced in the **last week** due to your knee.

| None | sitting<br>Mild | Moderate | Severe | Extreme |
|---|---|---|---|---|
| A4. Standing None | Mild | Moderate | Severe | Extreme |
| A5. Bending to f | loor/pick up an o<br>Mild | object<br>Moderate | Severe | Extreme |
| A6. Walking on | flat surface<br>Mild | Moderate | Severe | Extreme |
| A7. Getting in/or | ut of car<br>Mild | Moderate | Severe | Extreme |
| A8. Going shopp<br>None | oing<br>Mild | Moderate | Severe | Extreme |
| A9. Putting on so | ocks/stockings<br>Mild | Moderate | Severe | Extreme |
| A10. Rising from | n bed<br>Mild | Moderate | Severe | Extreme |
| A11. Taking off | socks/stockings<br>Mild | Moderate | Severe | Extreme |
| A12. Lying in be | ed (turning over,<br>Mild | maintaining knee j<br>Moderate | position)<br>Severe | Extreme |
| A13. Getting in/o | out of bath<br>Mild | Moderate | Severe | Extreme |
| A14. Sitting None | Mild | Moderate | Severe | Extreme |
| A15. Getting on/ | off toilet Mild | Moderate | Severe | Extreme |

For each of the following activities please indicate the degree of difficulty you have experienced in the last week due to your knee. A16. Heavy domestic duties (moving heavy boxes, scrubbing floors, etc) Mild Moderate Extreme Severe A17. Light domestic duties (cooking, dusting, etc) Mild Extreme None Moderate Severe Function, sports and recreational activities The following questions concern your physical function when being active on a higher level. The questions should be answered thinking of what degree of difficulty you have experienced during the last week due to your knee. SP1. Squatting Mild None Moderate Severe Extreme SP2. Running Mild None Moderate Severe Extreme SP3. Jumping Mild None Moderate Severe Extreme SP4. Twisting/pivoting on your injured knee None Mild Moderate Severe Extreme SP5. Kneeling Mild None Moderate Severe Extreme Quality of Life Q1. How often are you aware of your knee problem? Never Monthly Weekly Daily Constantly Q2. Have you modified your life style to avoid potentially damaging activities to your knee? Not at all Mildly Moderately Severely Totally Q3. How much are you troubled with lack of confidence in your knee? Not at all Mildly Moderately Extremely Severely Q4. In general, how much difficulty do you have with your knee?

Thank you very much for completing all the questions in this questionnaire.

Severe

Extreme

Moderate

Mild

None


# **KOOS FAQs**

## **Background information**

#### What is the KOOS?

The Knee injury and Osteoarthritis Outcome Score (KOOS) is a patient-reported outcome measurement instrument, developed to assess the patient's opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury and also consequences of primary osteoarthritis (OA). It holds 42 items in five separately scored subscales: **KOOS Pain, KOOS Symptoms**, Function in daily living (**KOOS ADL**), Function in Sport and Recreation (**KOOS Sport/Rec**), and knee-related Quality of Life (**KOOS QOL**) (<u>Roos and Lohmander 2003</u>).

#### In which populations can the KOOS be used?

KOOS has been used in patients 13-79 years of age.

KOOS is intended to be used for knee injury that can result in posttraumatic osteoarthritis (OA); i.e. knee ligament injury (ACL, posterior cruciate ligament [PCL], medial collateral ligament [MCL]), meniscal tears, knee cartilage lesions, knee OA, and osteochondritis dissecans, etc.

KOOS is meant to be used over short and long time intervals; to assess changes from week to week induced by treatment (examples include: ligament reconstruction (ACL, PCL, MCL), meniscectomy, microfracture, osteochondral autografts, tibial osteotomy, total knee replacement (TKR), exercise (land-based, aquatic-based), intra-articular sodium hyaluronate injection, pharmacologic therapy, and glucosamine supplementation) or over years due to the primary injury, post traumatic OA or primary OA (Roos and Lohmander 2003).

#### How was the KOOS developed?

KOOS was developed by Ewa Roos and co-authors in the 1990s as an instrument to assess the patient's opinion about their knee and associated problems. Items were selected based on: (1) the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), version 3.0; (2) a literature review; (3) an expert panel (patients referred to physical therapy for knee injuries, orthopedic surgeons, and physical therapists from Sweden and the US); and, (4) a pilot study of two questionnaires (one for symptoms of ACL injury, one for symptoms of OA) in individuals with posttraumatic OA.

#### What are the KOOS subscales and what areas of health do they measure?

The KOOS collects data on five knee-specific patient-centered outcomes: (1) **KOOS Pain**; (2) **KOOS Symptoms**: Other symptoms such as swelling, restricted range of motion and mechanical symptoms; (3) **KOOS ADL**: Disability on the level of daily activities; (4) **KOOS Sport/Rec**: Disability on a level physically more demanding than activities of daily living; (5) **KOOS QOL**: Quality of life, mental and social aspects such as awareness and lifestyle changes.

#### In what settings is the KOOS responsive to change?

KOOS' responsiveness has been reported following surgical procedures including ACL reconstruction, meniscectomy, cartilage repair procedures, tibial osteotomy, total knee replacement as well as physical therapy, nutritional and pharmaceutical interventions. Following orthopedic surgery, including total knee replacement, KOOS QOL is usually as responsive, or more responsive, than KOOS Pain and KOOS ADL (Collins and Roos 2012).


#### What is the Minimal Detectable Change of the KOOS in different settings?

The minimal detectable change (MDC) is dependent on the test-retest reliability of an instrument. The more reliable a measure is, the smaller the difference that can be detected longitudinally. The test-retest reliability is, in turn, dependent on factors such as patient characteristics and time between assessments. In studies of patients with knee injury, the MDC ranges for KOOS Pain were 6-6.1, for KOOS Symptoms: 5-8.5, for KOOS ADL: 7-8, for KOOS Sport/Rec: 5.8-12, and for KOOS QOL: 7-7.2 (Collins, Misra et al. 2011).

In one study including patients with knee OA, the MDCs for KOOS Pain were 13.4, for KOOS Symptoms: 15.5, for KOOS ADL: 15.4, for KOOS Sport/Rec: 19.6, and for KOOS QOL: 21.1 (Collins, Misra et al. 2011).

#### What is the Minimal Clinically Important Change in the KOOS in different settings

The minimal clinically important change (MIC) can be defined as the smallest change score needed for the effect to be considered clinically relevant (de Vet, Ostelo et al. 2007). MIC can be calculated in many different ways using anchor-based and distribution-based methods. Recent publications highlight that there is probably no such thing as one MIC for a specific patient-reported outcome measure, such as the KOOS. Instead MIC seems to be dependent on context factors including patient group, intervention, time to follow-up, etc. Therefore, it is more probable that in the future, a range of MICs will be established for an instrument. Research is ongoing to establish the MIC for the KOOS in many different contexts. Until then, a MIC of 8-10 is considered appropriate for the KOOS (Roos and Lohmander 2003). For performing a sample size calculation, usually an SD of 15 can be used. However, the variation within the group to be studied will depend on the characteristics of the group. Usually elderly or more impaired groups have greater within-group variation than younger or healthier groups.

#### What is the Patient Acceptable Symptom State of the KOOS in different settings?

The Patient Acceptable Symptom State (PASS) can be defined as the value beyond which the patients can consider them well. The PASS is an absolute value (not a change value) and can be used as a patient centered and clinically relevant treatment target (the proportion of patients reaching a satisfactory state) (<u>Tubach, Ravaud et al. 2005</u>). Similar to the MIC, research is ongoing within this area to establish PASS for KOOS when used in different contexts.

#### **KOOS** administration

#### Who answers the questionnaire?

The KOOS is self-administered and completed by the patient. No interview or phone formats are available.

#### How long does it take to complete the KOOS?

The KOOS questionnaire takes about 10 minutes to fill out.

#### How is the KOOS administered?

The KOOS is self-explanatory and can be administered in the waiting room prior to a clinical visit or used in a postal mail survey. KOOS has not been validated for interview administration (Collins, Misra et al. 2011).

#### **KOOS Scores**


#### How is the KOOS scored?

The five patient-relevant subscales of KOOS are scored separately: KOOS Pain (9 items); KOOS Symptoms (7 items); KOOS ADL (17 items); KOOS Sport/Rec (5 items); KOOS QOL (4 items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0–100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopaedic assessment scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved. An aggregate total score is not calculated since it is regarded desirable to analyze and interpret the five dimensions separately. Please find more extensive instructions on score calculations in the scoring section of the KOOS User's Guide. For statistical purposes, when used as the primary outcome in an RCT, a single score can be constructed. In this case, the five individual subscale scores should be secondary outcomes. Please see reference (Roos, Engelhart et al. 2011) for more information on this procedure.

#### How are the KOOS scores interpreted?

The score is a percentage score from 0 to 100, with 0 representing extreme problems and 100 representing no problems. This scoring direction, 100 indicating no problems, is common in orthopaedic instruments and generic measures like the SF-36. In measures developed by rheumatologists, like the WOMAC, 100 usually represents the worst possible result.

#### How should the patient be instructed on scoring activities he/she is not able to perform?

It is important to determine whether or not each subscale is relevant at the time point chosen, considering the specific study population. For example, difficulty with Sport/Rec function may not be relevant to assess 2 weeks post-operatively.

The following guideline for study staff is available:

KOOS Pain and KOOS ADL subscales: If a subject avoids an activity (e.g., twisting/pivoting or going up or down stairs) due to doctor's orders or because the subject has chosen to avoid the activity, the subject should be instructed to choose "(4) Extreme" for those items.

KOOS Sport/Rec subscale: The same as above. Also, if a subject does not normally engage in an activity (e.g., running or jumping), the subject should be instructed to leave the item blank.

#### How do I handle missing items?

Missing data: If a mark is placed outside a box, the closest box is chosen. If two boxes are marked, that which indicates the more severe problem is chosen.

As long as at least 50% of the subscale items are answered for each subscale, a mean score can be calculated. If more than 50% of the subscale items are omitted, the response is considered invalid and no subscale score should be calculated. For KOOS Pain, this means that 5 items must be answered; for KOOS Symptoms, 4 items; for KOOS ADL, 9 items; for KOOS Sport/Rec, 3 items; and for KOOS QOL, 2 items in order to calculate a subscale score. Subscale scores are independent and can be reported for any number of the individual subscales, i.e. if a particular subscale is not considered valid (for example, KOOS Sport/Rec 2 weeks after total knee replacement), the results from the other subscales can be reported at this time-point.

NB: The excel Scoring sheet available for download does not automatically take the number of missing items into account.

#### Can a total score be calculated?

An aggregate total score is not calculated since it is regarded desirable to analyze and interpret the five dimensions separately. For statistical purposes, when used as the primary outcome in an RCT, a single score can be constructed. In this case, the five individual subscale scores should be secondary outcomes.


For more information on this procedure, see reference (Roos, Engelhart et al. 2011) or the FAQs section on statistics.

#### How do I present my data?

The results of the five subscales can be plotted as an outcome profile, preferably in a graph with scores from 0-100 on the y-axis and the five subscales on the x-axis (an example is presented in the KOOS User's Guide, under the heading of KOOS Profile). The order of the subscales from left to right should be: KOOS Pain, KOOS Symptoms, KOOS ADL, KOOS Sport/Rec and KOOS QOL. This way profiles can be compared visually across studies. Changing this order makes visual comparison more difficult.

#### How do I use KOOS as the primary outcome in an RCT?

There are two ways to apply the KOOS as the primary outcome in an RCT. Either way, the primary endpoint should be specified *a priori*. You can either (1) choose the single subscale you consider is the most likely to measure the change from the intervention of interest, or you can (2) create a composite score, referred to as KOOS4 or KOOS5, depending on the number of subscales included in this composite score. Please note that this is very different from calculating a total score! Calculating an average score from subscale scores ensures similar weight from all subscales in the composite score. Calculating a total score is never recommended. In either case, all KOOS subscales should be included as secondary endpoints to enable clinical interpretation of the results.

As examples, since exercise is aimed at improving physical function, it may be appropriate to apply the KOOS ADL subscale as the primary endpoint in an older group of OA patients, and the KOOS Sport/Rec subscale as the primary endpoint in a younger group of knee-injured patients in a trial of an exercise intervention. However, in pharmacological trials, the subscale KOOS Pain may be more appropriate as the primary endpoint since pharmacological agents often are supposed to relieve pain. When two different interventions are included (for example a surgical and a non-surgical) or when the intervention is supposed to affect more than one subscale to a similar degree, a composite score may be most appropriate as the primary outcome. Below, an example is given where KOOS4 was applied. You can also read more about "Single Subscale versus Overall score" and "Multiplicity" in the review by Roos et al (Roos, Engelhart et al. 2011).

#### References

Ageberg, E., M. Forssblad, et al. (2010). "Sex differences in patient-reported outcomes after anterior cruciate ligament reconstruction: data from the Swedish knee ligament register." Am J Sports Med 38(7): 1334-1342.

Beaton, D. E., C. Bombardier, et al. (2000). "Guidelines for the process of cross-cultural adaptation of self-report measures." Spine (Phila Pa 1976) 25(24): 3186-3191.

Collins, N. J., D. Misra, et al. (2011). "Measures of knee function: International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form, Knee Injury and Osteoarthritis Outcome Score (KOOS), Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form (KOOS-PS), Knee Outcome Survey Activities of Daily Living Scale (KOS-ADL), Lysholm Knee Scoring Scale, Oxford Knee Score (OKS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Activity Rating Scale (ARS), and Tegner Activity Score (TAS)." Arthritis care & research 63 Suppl 11: S208-228.

Collins, N. J. and E. M. Roos (2012). "Patient-reported outcomes for total hip and knee arthroplasty: commonly used instruments and attributes of a "good" measure." Clinics in geriatric medicine 28(3): 367-394.

de Vet, H. C., R. W. Ostelo, et al. (2007). "Minimally important change determined by a visual method integrating an anchor-based and a distribution-based approach." Quality of life research: an international journal of quality of life aspects of treatment, care and rehabilitation 16(1): 131-142.

Flandry, F., J. P. Hunt, et al. (1991). "Analysis of subjective knee complaints using visual analog scales." Am J Sports Med 19(2): 112-118.

Frobell, R. B., E. M. Roos, et al. (2010). "A randomized trial of treatment for acute anterior cruciate ligament tears." The New England journal of medicine 363(4): 331-342.

Frobell, R. B., E. Svensson, et al. (2008). "Self-reported activity level and knee function in amateur football players: the influence of age, gender, history of knee injury and level of competition." Knee Surg Sports Traumatol Arthrosc 16(7): 713-719. Gudbergsen, H., E. M. Bartels, et al. (2011). "Test-retest of computerized health status questionnaires frequently used in the monitoring of knee osteoarthritis: a randomized crossover trial." BMC musculoskeletal disorders 12: 190.

Lequesne, M. G., C. Mery, et al. (1987). "Indexes of severity for osteoarthritis of the hip and knee. Validation--value in comparison with other assessment tests." Scand J Rheumatol Suppl 65: 85-89.

Östenberg, A., E. M. Roos, et al. (2000). "Physical capacity in Female Soccer Players - Does Age Make a Difference?" Advances in


Physiotherapy 2(1): 39-48.

Paradowski, P. T., S. Bergman, et al. (2006). "Knee complaints vary with age and gender in the adult population. Population-based reference data for the Knee injury and Osteoarthritis Outcome Score (KOOS)." BMC Musculoskelet Disord 7: 38.

Roos, E., L. Engelhart, et al. (2011). "ICRS Recommendation Document: Patient-reported outcome instruments for use in patients with articular cartilage defects." Cartilage 2(2): 122-136.

Roos, E. M., H. P. Roos, et al. (1999). "WOMAC Osteoarthritis Index-additional dimensions for use in subjects with post-traumatic osteoarthritis of the knee. Western Ontario and MacMaster Universities." Osteoarthritis and cartilage 7(2): 216-21.

Roos, E. M. and L. S. Lohmander (2003). "Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis." Health Qual Life Outcomes 1: 64.

Roos, E. M., H. P. Roos, et al. (1998). "Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure." J Orthop Sports Phys Ther 28(2): 88-96.

Roos, E. M. and S. Toksvig-Larsen (2003). "Knee injury and Osteoarthritis Outcome Score (KOOS) - validation and comparison to the WOMAC in total knee replacement." Health Qual Life Outcomes 1(1): 17.

Salavati, M., B. Akhbari, et al. (2011). "Knee injury and Osteoarthritis Outcome Score (KOOS); reliability and validity in competitive athletes after anterior cruciate ligament reconstruction." Osteoarthritis and cartilage / OARS, Osteoarthritis Research Society 19(4): 406-410.

Tanner, S. M., K. N. Dainty, et al. (2007). "Knee-specific quality-of-life instruments: which ones measure symptoms and disabilities most important to patients?" Am J Sports Med 35(9): 1450-1458.

Tubach, F., P. Ravaud, et al. (2005). "Evaluation of clinically relevant states in patient reported outcomes in knee and hip osteoarthritis: the patient acceptable symptom state." Ann Rheum Dis 64(1): 34-37.


# **KOOS Scoring 2012**

A change in how to manage missing items was introduced in 2012. Previously, 2 missing items were allowed in each subscale. From 2012, at least 50% of the items should be responded to. The differences in subscale level are outlined in the following table:

| | Number of items needed<br>for calculation of<br>subscale score (2012<br>rule for missing items) | Number of items needed<br>for calculation of<br>subscale score (1998 rule<br>for missing items) |
|---|---|---|
| Pain | 5 | 7 |
| Symptoms | 4 | 5 |
| ADL | 9 | 15 |
| Sport/Rec | 3 | 3 |
| QOL | 2 | 2 |

## **KOOS Scoring instructions**

Assign the following scores to the boxes:

| None | Mild | Moderate | Severe | Extreme |
|------|------|----------|--------|---------|
| 0 | 1 | 2 | 3 | 4 |

Each subscale score is calculated independently. Calculate the mean score of the individual items of each subscale and divide by 4 (the highest possible score for a single answer option). Traditionally in orthopedics, 100 indicates no problems and 0 indicates extreme problems. The normalized score is transformed to meet this standard.

**Missing data:** If a mark is placed outside a box, the closest box is chosen. If two boxes are marked, that which indicates the more severe problem is chosen.

As long as at least 50% of the subscale items are answered for each subscale, a mean score can be calculated. If more than 50% of the subscale items are omitted, the response is considered invalid and no subscale score should be calculated. For the subscale Pain, this means that 5 items must be answered; for Symptoms, 4 items; for ADL, 9 items; for Sport/Rec, 3 items; and for QOL, 2 items must be answered in order to calculate a subscale score. Subscale scores are independent and can be reported


for any number of the individual subscales, i.e. if a particular subscale is not considered valid (for example, the subscale Sport/Rec 2 weeks after total knee replacement), the results from the other subscale can be reported at this time-point.

## **KOOS Excel Scoring Files**

Excel spreadsheets with formulae to calculate the five subscale scores are available from <a href="www.koos.nu">www.koos.nu</a>. If, for any reason, you prefer to use your own spreadsheets, the Excel formulae are given below. NB: The excel spreadsheet available from <a href="koos.nu">koos.nu</a> does not take the number of missing items into account and will return a total subscale score regardless of missing items.

**Excel:** When the raw data have been entered in the order the items occur in the KOOS questionnaires, these can be copied and pasted directly into an Excel spreadsheet to automatically calculate the five subscore scales. Please note that it has been assumed that the items in the subscale symptoms appear first in the questionnaire.

KOOS Pain: =100-AVERAGE(I2:Q2)/4\*100

KOOS Symptoms: =100-AVERAGE(B2:H2)/4\*100

KOOS ADL: =100-AVERAGE(R2:AH2)/4\*100

KOOS Sport/Rec: =100-AVERAGE(AI2:AM2)/4\*100

KOOS QOL: =100-AVERAGE(AN2:AQ2)/4\*100

#### **KOOS Manual Score Calculation**

The slightly updated version of the formulae (presented above and used from August 2012 in the spreadsheets available from <a href="www.koos.nu">www.koos.nu</a>) does not need any manual imputation: Apply the mean of the observed items within the subscale (e.g. KOOS Pain), divide by 4, and multiply by 100; when this number is then subtracted from 100, you have the KOOS subscale estimate for that particular cross-sectional assessment of the individual patient. For manual calculations, please use the formulae provided below for each subscale:

1. PAIN 
$$100 - \frac{\text{Mean Score (P1-P9)} \times 100}{4} = KOOS Pain$$

2. SYMPTOMS 
$$100 - \frac{\text{Mean Score (S1-S7)} \times 100}{4} = KOOS Symptoms$$

3. ADL 
$$100 - \frac{\text{Mean Score (A1-A17)} \times 100}{4} = KOOS ADL$$

4. SPORT/REC 
$$100 - \frac{\text{Mean Score (SP1-SP5)} \times 100}{4} = KOOS Sport/Rec$$

5. QOL 
$$100 - \frac{\text{Mean Score } (Q1-Q4)\times 100}{4} = KOOS \ QOL$$


#### WOMAC - How to score from the KOOS

Assign scores from 0 to 4 to the boxes as shown above. To get original WOMAC Scores, sum the item scores for each subscale. If you prefer

percentage scores in accordance with the KOOS, use the formula provided below to convert the original WOMAC scores.

Transformed scale = 100 - actual raw score x 100 maximum score

| WOMAC subscores | Original score = sum of Maximum score the following items | |
|---|---|---|
| Pain | P5-P9 | 20 |
| Stiffness | S6-S7 | 8 |
| Function | A1-A17 | 68 |

#### **KOOS** Profile

To visualize differences in the five different KOOS subscores and change between different administrations of the KOOS (e.g. pre-treatment to post-treatment), KOOS Profiles can be plotted. The example from Nilsdotter et al. [17] shows KOOS profiles prior to and at 3 time points following total knee replacement (TKR).



Fig. 1. KOOS profiles prior to and up to 5 years after TKR. Mean KOOS scores (n=80) at the preoperative, 6 months, 12 months and 5 year assessments after TKR.
